A PHASE I/II TRIAL OF ESCALATING DOSE OF YTTRIUM-90-LABELED ANTI-CD20 MONOCLONAL ANTIBODY IN COMBINATION WITH HIGH-DOSE ETOPOSIDE AND CYCLOPHOSPHAMIDE FOLLOWED BY AUTOLOGOUS STEM CELL TRANSPLANTATION FOR PATIENTS WITH POOR RISK/RELAPSED B-CELL NON-HODGKIN'S LYMPHOMA

NCT00562978

Document Date 03/28/2014

#### CITY OF HOPE NATIONAL MEDICAL CENTER 06/20/07 1500 EAST DUARTE ROAD **DUARTE, CA 91010**

#### DEPARTMENT OF HEMATOLOGY / BONE MARROW TRANSPLANTATION

A PHASE I/II TRIAL OF ESCALATING DOSE OF YTTRIUM-90-LABELED ANTI-CD20 TITLE: MONOCLONAL ANTIBODY IN COMBINATION WITH HIGH-DOSE ETOPOSIDE AND

CYCLOPHOSPHAMIDE FOLLOWED BY AUTOLOGOUS STEM CELL TRANSPLANTATION FOR

PATIENTS WITH POOR RISK/RELAPSED B-CELL NON-HODGKIN'S LYMPHOMA

IRB# 98153 CITY OF HOPE PROTOCOL NUMBER/VERSION NUMBER: Version 17 **DATE(S) OF AMENDMENT(S)/REVISION(S):** 

10/29/03, 04/06/04, 06/16/04

05/10/00

Amendment 1 - 01/31/00 -Version 01 Amendment 8 – 02/08/01 -Version 08 2 -05/03/01 -Amendment 05/10/00 -Version 02 Amendment 9 – Version 09 Amendment 3 – 06/05/00 -Version 03 Amendment 10 -08/07/01 -Version 10 Amendment 07/13/00 -Version 04 Amendment 11 -05/30/02 -Version 11 09/08/00 -Amendment 5 – Version 05 Amendment 12 – 10/29/03 -Version 12 04/06/04 -Amendment 6 – 10/25/00 -Version 06 Amendment 13 -Version 13 Amendment 7 - 12/20/00 -Version 07 Amendment 14 – 06/16/04 - Version 14 Amendment 15 - 06/20/07 - Version 15 Amendment 16 - 04/18/12 - Version 16

(title page only change)

Amendment 17 - 03/28/14 -- Version 17

SITE: Lymphoma

Low and Intermediate Grade CD20 (+) HISTOLOGY:

II, III, IV STAGE (IF APPLICABLE):

Chemotherapy/Radioimmunotherapy **MODALITY:** 

Phase I/II TYPE:

PRINCIPAL INVESTIGATOR:

Auayporn Nademanee, M.D. Department of Hematology/Hematopoietic Cell Transplantation 06/16/04

**COLLABORATING INVESTIGATOR:** 

Andrew Raubitschek, M.D. Department of Radioimmunotherapy

**PARTICIPATING CLINICIANS:** 

Stephen J. Forman, M.D. Department of Hematology/Hematopoietic Cell Transplantation 06/16/04

Joycelynne Palmer, Ph.D. Department of Biostatistics 10/29/03

> City of Hope National Medical Center **PARTICIPATING INSTITUTIONS:**

INVESTIGATIONAL NEW DRUG (IND) NUMBER: **BB-IND 8836**  05/10/00, 06/05/00, 09/08/00, 10/29/03, 06/16/04

## TABLE OF CONTENTS

| 1.0 | BACKO | GROUND RATIONALE | 1 |
|---|---|---|---|
| 2.0 | OBJEC | TIVES | 8 |
| 3.0 | STUDY | DESIGN | 8 |
| 4.0 | DRUG | FORMULATION | 9 |
| 5.0 | STAGI | NG CRITERIA | 12 |
| 6.0 | ELIGII | BILITY CRITERIA | 13 |
| 7.0 | EXCLU | JSION CRITERIA | 14 |
| 8.0 | TREAT | TMENT PLAN | 14 |
| 9.0 | STUDY | DESIGN AND RULES FOR DOSE ESCALATION | 18 |
| 10.0 | STUDY | CALENDAR - PREPARATIVE REGIMEN AND PBSCT | 21 |
| 11.0 | CRITE | RIA FOR EVALUATION AND ENDPOINT DEFINITIONS | 22 |
| 12.0 | STATIS | STICAL CONSIDERATIONS | 23 |
| 13.0 | REGIS | TRATION GUIDELINES | 24 |
| 14.0 | RECOI | RDS TO BE KEPT AND DATA SUBMISSION SCHEDULE | 24 |
| 15.0 | GENDI | ER AND MINORITIES | 25 |
| 16.0 | DATA 1 | MANAGEMENT | 25 |
| 17.0 | ETHIC | AL AND REGULATORY CONSIDERATIONS | 25 |
| 18.0 | REFER | RENCES | 26 |
| Apper | ndix I | Common Toxicity Criteria (CTC) | <b>A1</b> |
| Apper | ndix II | <b>Toxicity Module</b> | A38 |
| Apper | ndix III | Infection Module | A39 |
| Apper | ndix IV | Performance Status Scales/Scores | A40 |
| Apper | ndix V | RTOG/EORTC Late Radiation Morbidity Scoring Scheme | A41 |
| Apper | ndix VI | BMT Complex/Multi-Component Events | A44 |

#### 1.0 BACKGROUND RATIONALE

Non-Hodgkin's lymphomas (NHLs) are the sixth most common cause of cancer-related deaths in the United States. The incidence of NHL has increased by 50% over the past 15 years. The incidence of both indolent and aggressive lymphomas increases with age, making these the most commonly diagnosed lymphoid malignancies in patients over 60 years old. Despite the use of aggressive combination chemotherapy regimens, approximately 30-40% of patients with intermediate- and high-grade NHL does not achieve complete remission (CR) or suffers relapse after attaining remission.<sup>2</sup> High-dose chemotherapy or chemo/radiotherapy followed by autologous bone marrow or stem cell transplantation (ASCT) has been shown to induce longterm disease control in about 10-50% of patients with relapsed and refractory intermediate- and high-grade lymphoma.<sup>3</sup> Recently, the benefit of high-dose therapy and ASCT proved to be superior to conventional salvage chemotherapy in a randomized Parma study of 215 patients with chemotherapy-sensitive NHL in relapse. The 5-year event-free survival (EFS) was 46% for the ASCT group as compared to 12% for the salvage therapy without transplantation (p = 0.001). Thus, high-dose therapy and ASCT has become a potential curative modality for patients with recurrent aggressive lymphoma. However, not all patients derive long-term benefits from this treatment and recurrent disease remains the single most common cause of treatment failure posthigh-dose therapy and ASCT. Therefore, new therapeutic approaches are needed.

Patients with low-grade NHL have indolent clinical courses and are not cured by current treatment approaches. Although most patients can achieve a complete remission with standard treatment, the median duration of first CR ranges from 12 to 36 months. Relapsed low-grade lymphoma may still respond to salvage therapy. But the duration of subsequent remissions progressively decreases. High-dose therapy and ASCT has been shown to improve survival and to increase the duration of remission in some patients with relapsed low-grade NHL. However, because of the long natural history and the continued pattern of relapse post-ASCT in some studies, the role of high-dose therapy and ASCT as a potential curative treatment for patients with relapsed low-grade lymphoma has not been clearly established.

Recently, the role of radioimmunotherapy for treatment of NHL has emerged. Radioisotope-labeled monoclonal antibodies provide a mechanism by which radioactivity can be directly targeted to tumors sites while sparing normal tissues. B-cell lymphomas are attractive targets for radioimmunotherapy because of their radiosensitivity, their well-defined surface antigens and the availability of multiple monoclonal antibodies to those antigens.

## 1.1 Results of High-Dose Chemo/Radiotherapy and ASCT for NHL

Several high-dose therapy regimens have been used as preparative regimens for NHL. But so far, none of these regimens have emerged as the best regimen. However, since NHL is radiosensitive and based on experience with acute leukemia, the combination of total body irradiation (TBI) and cyclophosphamide (Cy) has been widely used as a preparative regimen for some patients with lymphoid malignancies. In an attempt to reduce relapse rates, etoposide has been added to the TBI and Cy regimen because of its known activity in lymphoma. The results of phase I and II studies of TBI 12.0 Gy, etoposide 60 mg/kg and Cy 100 mg/kg conducted at City of Hope<sup>6</sup>. Stanford University<sup>7</sup> and Fred Hutchinson Cancer Research Center (FHCRC)<sup>8</sup> demonstrate the activity of this regimen in patients with lymphoid malignancies. The transplantrelated mortality within 100 days was 7-8%, with the common causes of death being venoocclusive disease (VOD), diffuse alveolar hemorrhage and infection. The major transplantrelated morbidities were mucositis and skin toxicities, which were fully reversible. The 5-year EFS and overall survival (OS) were 52% [95% Confidence interval (CI) 42-62%] and 61% (95% CI 50-73%), respectively for 134 patients with NHL who underwent ASCT utilizing this regimen at Stanford. These results have been confirmed in the Southwestern Oncology Group cooperative trial. Despite its effectiveness, the relapse rate of 34-53 % remains considerably high. Thus, new preparative regimens need to be explored.

## 1.2 Radionuclides for Radioimmunotherapy

Iodine-131 (<sup>131</sup>I) has been the gold standard for radioimmunotherapy due to its long track record in treating thyroid carcinomas, its well-defined radiochemistry, its clinical availability, and its potential for both radioimmunoscintigraphy and radioimmunotherapy. <sup>131</sup>I has been employed in the majority of reported clinical trials of radioimmunotherapy. However, there are disadvantages to <sup>131</sup>I, including its long 8-day half life, the risks of radiation exposure to health care providers and the non-specific irradiation to normal organs from gamma components of <sup>131</sup>I.

Yttrium-90 (<sup>90</sup>Y) may be an ideal radionuclide for radioimmunotherapy since it emits beta particles that are more potent than those delivered by <sup>131</sup>I. It is a pure beta emitter, making it a safer reagent for medical personnel to administer. In addition, the short half-life of <sup>90</sup>Y facilitates its use in combination with other agents, i.e. chemotherapy or total body radiation, and allows for high dose rates at localized sites. Unfortunately, <sup>90</sup>Y cannot be used for radioimmunoscintigraphy due to its absence of gamma emissions. Indium-111 (<sup>111</sup>In) has been substituted as an imaging reagent to show tumor localization in patients scheduled for <sup>90</sup>Y therapy, based on its biodistribution which is close to that of <sup>90</sup>Y. <sup>111</sup>In-labeled murine monoclonals have been used successfully in clinical imaging trials for cutaneous T-cell lymphoma, chronic lymphocytic leukemia, melanoma, and colon cancer.

### 1.3 Anti-CD 20

Anti-CD20 (anti-B1) is a murine monoclonal antibody of isotype IgG2a, raised against cryopreserved Burkitt's lymphoma cells. The antibody reacts against the B1 antigen, an epitope of the CD20 developmental cell surface protein. CD20 is a 35 kD cell surface phosphoprotein found on 95% of normal mature B-cells and more than 90% of B-cell non-Hodgkin's lymphomas and B-cell chronic lymphocytic leukemias tested, but not on T-cells, plasma cells, uncommitted

hematopoietic-precursors stem cells, dendritic cells, granulocytes, monocytes, or erythrocytes, or on tumors of T cell, myeloid or erythroid origin. CD20 is not shed and does not modulate from the surface after binding of antibody.

Anti-CD20 has been used extensively as a therapeutic agent for use in bone marrow purging. Clinical use of this antibody in marrow purging has shown it to be selective in eradicating B cell lymphomas as well as normal B-cells, while leaving other lymphocyte population intact. Some subpopulation of B cell precursors is left intact, as evidence by engraftment of the normal B cell compartment.

#### 1.4 IDEC-C2B8

IDEC-C2B8 is a chimeric antibody with a murine variable portion and a human IgG1 kappa constant portion that recognizes the CD20 antigens expressed on normal B-cells and most malignant B-cell lymphomas. IDEC-C2B8 shows specificity for the CD 20 antigen and binds with an apparent affinity of 4.3 x 10<sup>-9</sup>M. IDEC-C2B8 has also been reported to induce apoptosis and to sensitize drug-resistant human B-cell lymphoma cell lines to cytotoxic chemotherapy.

A phase I dose escalation pharmacokinetic trial of IDEC-C2B8 given as a single intravenous infusion using doses ranging from 10 mg/m² to 500 mg/m² in patients with relapsed or refractory low-grade lymphoma was reported by Maloney et al. The median half-life of the free antibody at doses ranging from 100 mg/m² to 500 mg/m² was 4.4 days (range 1.6-10.5 days). In phase II clinical studies, anti-tumor activity has been observed in patients with relapsed or refractory low-grade or follicular B-cell NHL. The majority of adverse events was mild to moderate and included fever, fatigue, chills and nausea which were primarily associated with the initial infusions. No quantifiable human anti-mouse antibodies (HAMA) or human anti-chimeric antibodies (HACA) were observed. Depletion of peripheral B-cells occurred rapidly following the first infusion with recovery beginning 6 months post-treatment. Despite this depletion of B-cells, there was minimal change in serum IgG, IgM, and IgA levels and no increase in the frequency or severity of infectious complications. Anti-tumor activity was observed at various disease sites including peripheral blood, bone marrow, lymph nodes, spleen and abdomen.

A phase III trial to assess the safety and efficacy of IDEC-C2B8 375 mg/m² given once weekly for four doses in 166 patients with relapsed or refractory low-grade or follicular NHL was reported by McLaughlin et al. <sup>10</sup> The overall response rate in 151 evaluable patients was 50% (9CR; 67 PR). The median duration of response has not been reached after a median follow-up of 9+ months. Conversion to negative bcl-2 status occurred in 57% of patients who were positive at baseline and subsequently reevaluated after the fourth infusion. No positive HAMA responses were observed in 67 patients evaluated and the incidence of HACA was less than 1%. Severe neutropenia and thrombocytopenia were observed in less than 2% of patients. IDEC-C2B8 has also been studied in 44 patients with relapsed diffuse large B-cell and mantle cell lymphoma. The overall response rate was 31%, with a 10% CR rate. Thus anti-CD20 monoclonal antibody has become a very effective salvage therapy for CD20+ B-cell low-and intermediate-grade NHL and this treatment has become an important addition to our armamentarium.

IDEC-C2B8 has also been studied in combination with chemotherapy. Czuczman et al<sup>11</sup>

conducted a phase II multi-center study evaluating the safety and anti-tumor activity of IDEC-C2B8 375 mg/m² for six doses in combination with six cycles of CHOP (cyclophosphamide, doxorubicin, vincristine and prednisone) chemotherapy in 40 patients with low-grade NHL. Combination therapy appeared safe and toxicity profile observed was consistent with that seen with CHOP alone. No HAMA or HACA responses were observed. The overall response rate in 35 patients who completed treatment was 100% (21 CR; 14 PR). The median time to disease progression has not been reached with follow-up time of 9-27+ months. Seven of eight patients who were bcl-2 positive at baseline by polymerase chain reaction (PCR) became negative in both peripheral blood and bone marrow following treatment. This combined therapy is being investigated in previously untreated patients with intermediate- and high-grade NHL.

## 1.5 Results of Radiolabeled Antibodies in the Treatment of Non-Hodgkin's Lymphoma

Most recent radioimmunotherapy trials for lymphoma have utilized <sup>131</sup>I-labeled anti-B1 (anti-CD20) antibody. Kaminski et al<sup>12</sup> first reported on a trial utilizing multiple treatments with low dose <sup>131</sup>I-labeled anti-B1 antibody in ten patients who had a CD20 positive B-cell lymphoma in whom primary therapy had failed. Six of the nine treated patients had tumor responses, including patients with bulky or chemotherapy-resistant diseases. Four patients had complete remissions (CR), and two had partial responses. The follow-up time was relatively short, but no disease progression was observed in the four patients who achieved a CR at 8-11 months. Toxicity was minimal with mild or no myelosuppression.

Based on these results, a phase I/II study of <sup>131</sup>I-labeled anti-B1 was conducted in 58 heavily pretreated patients with NHL (28 low-grade, 14 transformed low-grade, 15 intermediate-grade, and 2 high-grade). <sup>13</sup> The median number of prior therapy was 4, 88% had stage III or IV disease, 36% had bulky disease, 51% had an elevated LDH level and 14 had failed BMT. Patients received 1-3 dosimetric doses followed by a therapeutic dose. The dosimetric dose involved the IV administration of 5 mCi of <sup>131</sup>I anti-B1 antibody to determine the rate of whole body clearance so that a whole body radiation dose could be calculated. Each dosimetric dose was preceded by 0, 95, or 475 mg of unlabeled antibody. Therapeutic dose escalation was initiated at 25 cGy and adjusted in 10 cGy increment until the MTD. The MTD was 75 cGy for patients who had not undergone BMT. The overall response rate in these heavily pre-treated patients was 71% with a CR rate of 34%. The median duration of response was 271 days (95% CI; 40-394 days) and the median duration of CR was 566 days. Response was observed in both low-grade and transformed low-grade NHL as well as in patients with bulky disease and patients who had relapsed post-BMT.

Further trials of <sup>131</sup>I-labeled anti-B1 antibody at non-myeloablative doses has been studied in 4 separate clinical trials (phase I and II, single and multi-center) in 113 patients with low-grade NHL including 25 with transformed low-grade NHL. <sup>14</sup> Patients received a single dosimetric dose of 450 mg of unlabeled anti-B1 infusion over one hour followed by 35 mg radiolabeled with 5 mCi <sup>131</sup>I over ½ hour. The therapeutic dose was administered 7 to 14 days after the dosimetric dose and consisted of the same unlabeled and labeled antibody doses. The overall response rate was 77% with a CR rate of 45% and 67% of the complete responders were in continuous remission for > 4 years. Reversible hematologic toxicity was the dose-limiting toxicity. ANC < 100/mm<sup>3</sup> was observed in 2.6% of patients and platelets < 10,000/mm<sup>3</sup> in 5.3%. The nadir

typically occurred at week 5-6 with recovery by week 8-9. The most common non-hematologic toxicities were transient mild to moderate fever, nausea, asthenia, and chills. None of the patients developed HAMA. These results suggest that <sup>131</sup>I-labeled anti-B1 is safe and effective and may induce prolonged CR in heavily pre-treated low-grade and transformed low-grade NHL.

## 1.6 Results of <sup>131</sup>I anti-B1 Monoclonal Antibody with Autologous Bone Marrow Support

Although promising results have been reported with radiolabeled MAb for NHL, these results may be improved by using higher dose or myeloablative radiation dose. The use of radiolabeled MAb at myeloablative radiation dose followed by autologous stem cell rescue has been explored by investigators from The Fred Hutchinson Cancer Research Center. Press et al<sup>15</sup> conducted a trial utilizing higher dose of <sup>131</sup>I-labeled anti-CD20 antibody with autologous bone marrow rescue in 43 patients with B-cell lymphoma in relapse. In this study, sequential biodistribution studies were performed with escalating doses of antibody (0.5, 2.5, and 10 mg/kg) trace-labeled with 5 to 10 mCi of <sup>131</sup>I. Patients whose tumors were estimated to receive greater doses of radiation than liver, lungs, or kidneys (a favorable biodistribution) were eligible for the therapeutic infusion of <sup>131</sup>I-labeled antibody. Of the 43 patients, 24 had a favorable biodistribution, and 19 received therapeutic infusion of 234-777 mCi of <sup>131</sup>I-labeled antibodies (58-1168 mg) followed by autologous marrow infusion. Sixteen patients achieved a CR, two had a partial response and one had a minor response. Nine of the complete responders have remained in continuous CR for 3 to 53 months. Toxicities include myelosuppression, nausea, infection and two episodes of cardiopulmonary toxicity. In this study, cardiopulmonary toxicity was the dose limiting, non-hematopoietic toxicity of high-dose <sup>131</sup>I-labeled antibody.

In an attempt to reduce toxicity to normal tissues and to directly deliver higher dose of radiation to tumor sites. <sup>131</sup>I-labeled-anti-CD20 MAb has been incorporated into high-dose therapy regimen instead of TBI. Press et al<sup>16</sup> reported results of a phase I/II study to define the MTD of an <sup>131</sup>Ilabeled anti-B1 monoclonal antibody which can be given with high-dose etoposide and cyclophosphamide in conjunction with ASCT in 38 (26 low-grade; 12 aggressive) NHL patients. Patients were treated in a cohorts of 4 patients each with doses of <sup>131</sup>I-anti-B1 antibody (2.5 mg/kg, 318-840 mCi) calculated to deliver 20-27 Gy of radiation to dose-limiting, critical normal organs, followed by etoposide (0 or 60 mg/kg), cyclophosphamide (100 mg/kg), and ABMT (15 patients) or ASCT (22 patients). Of the 37 evaluable patients, 33 (89%) were currently alive and 29 (78%) were progression-free after a median follow-up of 1.5 yr. Toxicities included grade 4 myelosuppression in all patients, grade 2-3 nausea in 26 (70%), pulmonary infiltrate in 4 and grade 3 VOD in 2 patients. There were four death; 3 from progressive NHL and 1 from disseminated Varicella. These results suggest that <sup>131</sup>I- anti-B1 antibody can be given at doses delivering  $\geq 25$  Gy to critical normal organs, with pulmonary and gastrointestinal toxicities being dose-limiting. Although additional studies are needed, <sup>131</sup>I-anti-B1 antibody can be safely given in combination with high-dose chemotherapy in an autologous stem cell transplant setting for NHL.

## 1.7 90 Y -Anti-CD20 Radioimmunotherapy for Relapsed NHL

A phase I/II dose escalation study of <sup>90</sup>Y-murine anti-CD20 monoclonal antibody (MAb) in patients with recurrent B-cell lymphoma was performed by Knox et al.<sup>17</sup> The primary objectives

of the study were: (a) to determine the effect of the preinfusion of unlabeled anti-CD20 MAb on the biodistribution of <sup>111</sup>In-anti-CD20 MAb; (b) to determine the maximal tolerated dose of <sup>90</sup>Y-anti-CD20 MAb that does not require bone marrow transplantation; and (c) to evaluate the safety and antitumor effect of <sup>90</sup>Y-anti-CD20 MAb in patients with recurrent B-cell lymphoma. Eighteen patients with relapsed low- or intermediate-grade non-Hodgkin's lymphoma were treated. Biodistribution studies with <sup>111</sup>In- anti-CD20 MAb were performed prior to therapy. Groups of three or four patients were treated at dose levels of approx 13.5, 20, 30, 40, and 50 mCi <sup>90</sup>Y-anti-CD20 MAb. Three patients were retreated at the 40 mCi dose level. The use of unlabeled antibody affected the biodistribution favorably. Nonhematological toxicity was minimal. The only significant toxicity was myelosuppression. The overall response rate following a single dose of <sup>90</sup>Y-anti-CD20 MAb therapy was 72%, with six complete responses and seven partial responses and freedom from progression of 3-29+ mo following treatment. Radioimmunotherapy with less than or equal to 50 mCi <sup>90</sup>Y-anti-CD20 MAb resulted in minimal nonhematological toxicity and durable clinical responses in patients with recurrent B-cell lymphoma. Doses of less than or equal to 40 mCi <sup>90</sup>Y-anti-CD20 MAb were not myeloablative.

Results of a phase I/II study utilizing chimeric antibody Rituximab as the unlabeled clearing antibody and <sup>90</sup>Y conjugated anti-CD20 (IDEC-Y2B8, conjugated to the parent murine monoclonal 2B8) was recently reported. In the study reported by Witzig et al<sup>18</sup>, the first portion of the study compared 100 mg/m<sup>2</sup> with 250 mg/m<sup>2</sup> of Rituximab as the clearing dose and compared dosimetry imaging capabilities. It was determined that 250 mg/m<sup>2</sup> of Rituximab was the optimal dose to be used. In the second portion of the phase I study, the dose of IDEC-Y2B8 was escalated from 0.2 mCi/kg to 0.4 mCi/kg. No bone marrow or stem cell harvest was required. None of the patients treated at 0.2, 0.3 and 0.4 mCi/kg whose baseline platelet count > 150,000/mm<sup>3</sup> developed grade 4 hematologic toxicity, whereas 3 of 6 patients treated at 0.2 or 0.3 mCi/kg with baseline platelet counts between 100,000 to 150,000/mm<sup>3</sup> developed transient grade 4 hematologic toxicity.

The dosimetry from this phase I/II trial of IDEC-Y2B8 was reported by Wiseman et al. <sup>19</sup> Fortytwo patients with low- and intermediate-grade NHL received IDEC-Y2B8 following injection of unlabeled Rituximab (cold antibodies) followed by 2 mg of mouse anti-CD20 antibody labeled with 5 mCi <sup>111</sup>In (IDEC-In2B8). <sup>90</sup>Y 0.2, 0.3, or 0.4 mCi/kg was given 7 days following <sup>111</sup>I. The patients had <sup>111</sup>In dosimetry performed by serial whole body gamma camera imaging, urine collection and blood sampling at 0, 2, 6, 24, 48, 72, 96 and 144 hours. The highest mean calculated <sup>90</sup>Y radiation dose to a normal organ was spleen with 24.16 rads/mCi (0.6-67.0), followed by liver with 17.2 rad/mCi (9.4-39.2) and lungs with 12.9 rads/mCi (4.2-67.7). <sup>90</sup>Y dose of 0.4 mCi/kg was the MTD for bone marrow toxicity (thrombocytopenia and neutropenia). These results suggest that: 1) no organ irradiated beyond safety levels; 2) <sup>111</sup>I can serve as a predictor of <sup>90</sup>Y; 3) Rituximab dose of 250 mg/m² has been established as the "cold" antibody with added benefits of its therapeutic effect; and 4) bone marrow toxicity was the dose-limiting effect with full and predictable recovery.

Outcomes from this trial have been compiled in a submitted publication. <sup>19</sup> The overall response rate (ORR) for the intent-to-treat population (n = 51) was 67% (26% CR, 41% PR); for the low-grade group (n = 34) 82% (27% CR, 56% PR); 43% for intermediate grade (n = 4); and 0% for mantle cell (n = 3). Responses were seen in patients with bulky (> 7 cm) disease (41%) and

splenomegaly (50%). Kaplan-Meier estimate of time-to-progression in responders and duration of response is 12.9+ months and 11.7+ months, respectively. Adverse events were primarily hematologic and correlated with baseline extent of marrow involvement with NHL and baseline platelet count. Only one patient developed an anti-antibody response (HACA/HAMA).

## 1.8 Study Proposal

The high-dose therapy regimen of FTBI 1200 cGy, etoposide 60 mg/kg and Cy 100 mg/kg has been used extensively at City of Hope as a preparative regimen for patients with hematological malignancies. Given the relatively high relapse rate associated with this regimen, the effective anti-lymphoma therapy of IDEC-C2B8, and the safety and feasibility of IDEC-Y2B8 with the ability to directly deliver radiation to tumors sites, we propose to study a new preparative regimen in patients with relapsed NHL which will utilize <sup>90</sup>Y-labeled anti-CD20 antibody (IDEC-Y2B8) instead of TBI in combination with high-dose etoposide and cyclophosphamide. We plan to conduct a phase I/II trial to define the maximum tolerated dose (MTD) of IDEC-Y2B8 that can be given with high-dose etoposide and cyclophosphamide followed by ASCT, and to define the response rate and toxicities associated with this regimen. To avoid liver toxicity, etoposide dose will be started at 40 mg/kg and escalated to 60 mg/kg and the dose of Cy will be fixed at 100 mg/kg.

05/03/01, 06/16/04

The patient will undergo a dosimetry study with IDEC-In2B8 to confirm favorable localization of isotope one week prior to administration of therapeutic dose IDEC-Y2B8. Serial gamma camera images will be obtained at the end of the infusion, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours post-infusion. At each time point, one whole body and 4 spot planar scans will be acquired with the Toshiba dual head camera. In addition, two SPECT images will be obtained at 48 and 72 -96 hour time points. Nuclear Medicine images will be used to estimate the distribution of activity in various organs, especially liver, lungs, kidney, heart and spleen. Blood samples will be drawn prior to IDEC-C2B8 and at approximately 0 hours (immediately prior to IDEC-In2B8), 2 hours, 4 - 6 hours, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours following antibody infusion. These samples will be used to analyze antibody clearance and bone marrow dose estimates. Urine samples will be collected daily for six days to analyze radioisotope clearance.

05/03/01, 08/07/01,

Favorable biodistribution will be defined as tumor dose greater than any normal organ, except spleen and bone marrow, ie. liver, lung, kidney. For patients in CR at time of transplantation, no specific tumor localization is required as long as Ga 67 scan and/or FDG-PET scan is negative. Tumor dose will be calculated from multiple gamma camera images and blood/urine pharmacokinetics. If the patient shows favorable biodistribution, the therapeutic dose will be administered on day -14. Serial gamma camera images will be obtained at the end of the infusion, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours post-infusion. At each time point, one whole body and 4 spot planar scans will be acquired with the Toshiba dual head camera. Nuclear Medicine images will be used to confirm estimates of the distribution of activity in various organs, especially liver, lungs, kidney, heart and spleen. Blood samples will be drawn prior to IDEC-C2B8 and at approximately 0 hours (immediately prior to IDEC-In2B8 / IDEC-Y2B8), 2 hours, 4 - 6 hours, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours following antibody infusion. These samples will be used to analyze antibody clearance and bone

marrow dose estimation. Urine samples will be collected daily for six days to analyze radioisotope clearance. The therapeutic dose will be administered to deliver a target dose of 1000 cGy to the organ projected to receive the highest dose from the imaging study. After the first two dose levels the dose will be increased in increments of 250 cGy until a maximum of 2500 cGy is attained or dose limiting toxicity is encountered.

#### 2.0 OBJECTIVES

05/10/00

10/29/03

- 2.1 To evaluate the safety and efficacy of a new preparative regimen of <sup>90</sup>Y-labeled anti-CD20 MAb (IDEC-Y2B8) in combination with high-dose etoposide and cyclophosphamide followed by ASCT for treatment of patients with relapsed/refractory and poor risk NHL.
- 2.2 To determine the MTD of <sup>90</sup>Y-anti-CD20 MAb which can be given with high-dose etoposide 60 mg/kg and high-dose cyclophosphamide 100 mg/kg followed by ASCT in patients with NHL.
- 2.3 To perform dosimetry study to estimate the radiation dose delivered to the tumor and normal organs.
- 2.4 To evaluate the short-term and long-term complication of this new preparative regimen.

#### 3.0 STUDY DESIGN

This is an open-label phase I-II clinical and efficacy study of a new preparative regimen followed by autologous stem cell support in patients with relapsed and refractory NHL. Patients with low-, and intermediate-grade NHL who have relapsed followed conventional chemotherapy or have failed to achieve remission, and who are candidates for high-dose therapy and ASCT will be eligible for this study. All patients will receive IDEC-Y2B8 in combination with high-dose etoposide and cyclophosphamide followed by ASCT. The dose of Cy will be fixed at 100 mg/kg. There will be two doses escalating schema for etoposide and IDEC-Y2B8. Etoposide will be started at 40 mg/kg (cohort 1) and escalate to 60 mg/kg (cohort 2). The dose of Y2B8 will be the same for cohort 1 and 2, to deliver 1000 cGy to the normal organ receiving the greatest accumulation. If no dose limiting toxicity is observed, while the etoposide dose remains at 60 mg/kg, the dose of Y2B8 will be escalated to 1250 cGy, and then to a maximum of 2500 cGy, or until the MTD has been reached. Therefore, there will be cohorts with 3 patients per cohort as follows (an additional 2 patients per cohort will be accrued if there are eligible patients available prior to the determination of toxicity on the current dose level):

Cohort 1: Y2B8 to deliver 1000 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 40 mg/kg

cyclophosphamide 100 mg/kg

Cohort 2: Y2B8 to deliver 1000 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 3: Y2B8 to deliver 1250 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 4: Y2B8 to deliver 1500 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 5: Y2B8 to deliver 1750 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 6 to 8: Y2B8 to deliver 2000-2500 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

All patients will have peripheral blood stem cell collected with the target CD34+ of  $3.0 \times 10^6$ /kg. Patients will undergo dosimetry studies on day -21 and therapy on day -14. Etoposide will be given on day -4, followed by a day rest and cyclophosphamide on day -2. PBSC will be infused on day +1 when the radiation dose to the reinfused stem cells is estimated to be < 5 cGy.

### 4.0 DRUG FORMULATION

#### 4.1 IDEC-Y2B8

a. Drug Formulation and Procurement

IDEC-2B8-MX-DTPA Two ml glass septum vial containing 2 ml (3.2 mg) IDEC-2B8-MX-DTPA in low metal normal saline at 1.6 mg/ml.

RITUXAN (IDEC-C2B8) Ten ml (100 mg) and/or 50 ml (500 mg) pharmaceutical grade glass vials at a concentration of 10 mg of protein per ml.

<sup>111</sup>In-chloride 5 mCi of Indium-111 chloride supplied in .05M HCl. 40-100 mCi Yttrium-90 chloride supplied in .05M HCl.

#### b. Drug Toxicity

Myelosuppression is the dose limiting toxicity in non marrow supported regimens. With marrow support liver, kidney, and lung are likely to be the dose limiting organs for toxicity. Infusional toxicity of chills and rigors are common with the first administration but rarely with subsequent doses. Decreasing the rate of infusion and the administration of antihistamines can control these toxicities.

c. Drug Storage, Reconstitution and Stability

All antibodies will be stored in the investigational pharmacy at 4°C until the day of use.

05/03/01

10/29/03

Once diluted the unlabeled antibody is to be used within 24 hours if held at 4°C and at room temperature for an additional 12 hours. The radiolabeled solutions should be used within 6 hrs and should be held at 2-8°C until administered.

# 4.2 VP-16 (epipodophyllotoxin, etoposide, 4'-demethyl-9(4,6-o-β) d-ethylideneglycopyranoside).

## a. Drug Formulation and Procurement

VP-16 is supplied by Bristol Laboratories in a 100 mg ampule in 5 cc of a solution containing citric acid, 10 mg; benzyl alcohol, 150 mg; polysorbate 80, purified, 250 mg; polyethylene glycol 300, 3.75 gm; absolute alcohol q s., 5 cc.

## b. Drug Toxicity

Myelosuppression, primarily granulocytopenia, is the dose-limiting toxicity. Gastrointestinal toxicity at high doses includes nausea, emesis and mucositis. Reversible hepatotoxicity may occur at very high doses. The acute side effects of occasional bronchospasm and hypotension are avoided by slow intravenous administration.

### c. Drug Storage, Reconstitution and Stability

The contents of the ampoule are diluted with 50 volumes of NaCl solution for injection, USP, and administered by slow intravenous infusion. Patients will receive the drug through a central venous catheter at a rate of 60 mg/kg/4 hours.

## 4.3 Cyclophosphamide (Neosar, Cytoxan), NSC-26271

## a. Drug Formulation and Procurement

Cyclophosphamide is an alkylating agent dispensed in 100, 200 and 500 mg vials containing a dry powder. Cyclophosphamide will be purchased from Adria Laboratories.

### b. Drug Toxicity

Patients must be well hydrated before and for several hours following administration of cyclophosphamide to reduce the potential for hemorrhagic cystitis. The more common side effects include nausea and vomiting, and alopecia. Acute toxicity includes principally leukopenia, with the nadir occurring 7-14 days after a single IV dose. At high doses, occasional pulmonary toxicity has been reported. Rare cardiac toxicity (congestive heart failure) has occurred in patients previously treated with anthracyclines.

#### c. Drug Storage, Reconstitution and Stability

Cyclophosphamide is reconstituted with either sterile water for injection, USP or bacteriostatic water for injection, USP (Paraben preserved only), using 5 ml for the 100 mg vial, 10 ml for the 200 mg vial or 25 ml for the 500 mg vial. Each ml of reconstituted solution contains 20 mg cyclophosphamide per ml. The drug is diluted in 5% dextrose and water or physiological saline and given by IV infusion.

## 4.4 Mesna (Sodium 2-Mercaptoethane sulfonate)

## a. Drug Formulation and Procurement

Mesna is provided by Bristol Laboratories as a 10% (100 mg/ml) solution in water with 0.25 mg EDTA as excipient in 4 ml ampules.

## b. Drug Storage, Reconstitution and Stability

Mesna solutions have been shown to be stable on extended storage at room temperature in ampules. No change in composition of the ampules was noted at one year's storage in these conditions

On exposure to air Mesna is known to undergo oxidation to disulfide. Since the Mesna concentration of opened ampules may decrease with time, the ampule should be opened just before use and the unused part discarded.

#### c. Administration

Each dose of Mesna will be diluted in 50 cc of 5% dextrose/water or 0.9% normal saline and infused intravenously over 15 minutes.

## 4.5 DTPA (Diethyltriaminepenatacetic acid)

## a. Drug Formulation and Procurement

DTPA will be purchased from Heyl Pharmaceuticals, Berlin, Germany. It is supplied as a 1 gram ampule in 5 mls.

#### b. Drug toxicity

DTPA has been known to cause headaches, fever, chills, flu-like symptoms, nasal stuffiness, nausea, vomiting, abdominal cramping, and diarrhea. Other side effects that are less common include pain at the injection site, dehydration, decreased blood pressure, irregularities of heart rhythm, decreased blood counts, increased calcium, numbness and tingling, sneezing, excessive tearing, kidney damage, and zinc deficiency (which can result in a facial and perianal rash and tongue and mouth sores). In addition, there is always a risk of a very uncommon or previously unknown side effect occurring. Stopping the infusion normally reverses the side effects. Headaches and tingling have been observed at the City of Hope but were reversible. Trace metals will be administered at the end of infusion to replace any depleted heavy metals.

#### c. Drug Storage, Reconstitution and Stability

The DTPA solution will be diluted with 250 mls normal saline and administered over 24 hours. Additional IV fluids will be administered to maintain a minimum of 125 mls/hour of fluid. No other heavy metals should be administered during the 24 hour infusion. Potassium may be administered as needed. DTPA has a long aqueous stability but should

06/05/00

be used within 48 hours of being drawn up by the pharmacy. Patients will receive 250 mgs/m<sup>2</sup> to a maximum of a total dose of 500 mgs.

#### 5.0 STAGING CRITERIA

Staging of disease must be evaluated at least 21 days after the end of the last chemotherapy and within 42 days prior to transplant.

5.1 The Ann Arbor staging criteria will be used. Stage is determined based on extent of disease at the time of diagnosis.

## 5.2 Ann Arbor Classification (AJCC Manual for Staging of Cancer, 4th ed. 1992)

| STAGE I | Involvement of a single lymph node region (1) or a single extralymphatic organ or |
|---|---|
| | site $(1_E)$ . |
| <i>STAGE II</i> | Involvement of two or more lymph node regions on the same side of the diaphragm |
| | (II) or localized involvement of an extralymphatic organ or site and its associated |
| | regional lymph nodes $(11_E)$ . |
| STAGE III | Involvement of lymph node regions on both sides of the diaphragm (111) which may |
| | be accompanied by localized involvement of an associated extralymphatic organ or |
| | site $(111_E)$ or spleen $(111_S)$ or both $(II(1_{SE})$ . |
| STAGE IV | Diffuse or disseminated involvement of one or more extralymphatic organs with or |
| | without associated lymph node involvement, or isolated extralymphatic organ |
| | involvement with distant (non-regional) nodal involvement. |
| A = Asymp | ` ' ' |
| | sweats, weight loss > 10% of body weight |
| D - rever, s | sweats, weight loss / 1070 of body weight |

## 5.3 Definitions of Sensitivity of Disease:

Patients are grouped into one of three groups based on sensitivity of disease:

- 1. Induction failure: patients who did not achieve a CR or PR from induction chemotherapy;
- 2. Resistant Relapse: patients who did not achieve a CR or PR from the most recent standard salvage chemotherapy;
- 3. Sensitive Relapse: patients who did achieve a CR or PR from the most recent standard salvage chemotherapy.

## 5.4 Definitions of Poor Risk Disease

05/10/00

- 1. Age Adjusted International Prognostic Index (IPI) High- (3 risk factors) or High-Intermediate (2 risk factors) based on the following risk factors: stage III-IV, elevated serum lactate dehydrogenase level (LDH) and ECOG performance status 2-4.
- 2. Patients with aggressive NHL including mantle cell lymphoma who required 2 different induction chemotherapy regimens to achieve a partial/complete remission.

| 05/03/01 | | 3. Patients with B-Cell NHL who fail to achieve a complete remission after adequate induction chemotherapy regimen(s). |
|---|---|---|
| 05/10/00 | 6.0 | ELIGIBILITY CRITERIA |
| 05/10/00 | 6.1 | Favorable biodistribution on imaging dose |
| 08/07/01 | 6.2 | $age \ge 18$ and $\le 60$ years |
| 10/29/03 | 6.3 | All patients must have biopsy proven diagnosis of low- and intermediate-grade NHL including follicular small cleaved, follicular mixed, follicular large cell, diffuse small cleaved, diffuse mixed, diffuse large cell, and immunoblastic lymphoma (working formulation B, C, D, E, F, G and H) including mantle cell lymphoma. Transformed low-grade lymphomas are eligible |
| | 6.4 | Demonstrated monoclonal CD20 + B-cell population in lymph nodes and/or bone marrow |
| 05/10/00 | 6.5 | Patients must have relapsed after achieving a complete or partial response to prior therapy, have never responded to prior therapy or have poor risk disease |
| 05/10/00,05/30/02<br>10/29/03 | 6.6 | Patients must have bone marrow aspiration and biopsy within 42 days before salvage chemotherapy or stem cell collection which show $\leq 10\%$ lymphomatous involvement of total cellularity |
| 09/08/00, 05/30/02 | <b>6.</b> 7 | Platelet count should be normal before initiation of chemotherapy for salvage purposes or stem cell mobilization. If the patient collected his/her stem cells at an outside facility, then the platelet count must be normal before the imaging dose of antibody |
| | 6.8 | Normal renal function test with serum creatinine of $\leq 1.5$ mg/dl, or a creatinine clearance of $\geq 60$ ml/min |
| | 6.9 | Adequate pulmonary function as measured by FEV1 $>$ 65% of predicted measured, or a DLCO $\geq$ 50% of predicted measured |
| 04/06/04 | 6.10 | Cardiac Ejection fraction of > 50% by echocardiogram or multiple gated acquisition scan |
| | 6.11 | Adequate liver function tests with a bilirubin of $\leq 1.5~x$ normal and SGOT or SGPT $\leq 2~x$ normal |
| | 6.12 | Negative human immunodeficiency virus antibody |
| 05/03/01 | 6.13 | ECOG performance status 0 or 1; or KPS $\geq$ 80 |
| | 6.14 | No active CNS disease or prior history of CNS disease |
| 07/13/00 | 6.15 | Patients who have received involved field external beam therapy to area excluding lung, heart, liver and kidney are allowed, but will be evaluated on a case by case basis |
| | 6.16 | Patients must have recovered from last therapy and should be at least four weeks from prior radiation or chemotherapy |

6.17 The patient should have a baseline CT scan and Ga 67 scan and/or FDG-PET scan after 08/07/01 the last chemotherapy prior to initiation of treatment 6.18 Normal cytogenetic study on bone marrow (prior to salvage chemotherapy or stem cell 10/29/03 collection). However, cytogenetic study on peripheral blood is acceptable if bone marrow biopsy has already been done and shows no sign of MDS or lymphoma and a repeat bone marrow is deemed unnecessary by attending physician 7.0 **EXCLUSION CRITERIA** 7.1 Presence of human anti-mouse antibody (HAMA) or human anti-chimeric antibody 7.2 Prior radioimmunotherapy Failure to collect adequate number of CD34 + cells  $\geq 3 \times 10^6$  /kg 7.3 7.4 Abnormal cytogenetic study on the bone marrow aspirate sample prior to stem cell collection 7.5 Prior bone marrow transplantation **7.6** Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, 07/13/00 adequately treated noninvasive carcinomas, or other cancer from which the patient has been disease-free for at least five years *7.7* Active evidence of Hepatitis B and C infection; Hepatitis B surface antigen positive *7.8* History of alcohol abuse 02/08/01 *7.9* Patient weighs more than 250 pounds 10/29/03 8.0 TREATMENT PLAN 8.1 Outline of the preparative regimen Dosimetry with 5 mCi IDEC-In2B8 following 250 mg/M<sup>2</sup> Rituxan *Day -21* IDEC-Y2B8 with 5 mCi IDEC-In2B8 following 250 mg/M<sup>2</sup> Rituxan Day -14 Day -7 Bone marrow biopsy and dose estimation 05/30/02 Etoposide 40 mg/kg adjusted ideal body weight (Cohort 1) or 60 mg/kg Day -4 05/30/02, 10/29/03 adjusted ideal body weight for other cohorts Day -2 Cyclophosphamide 100 mg/kg ideal body weight 10/29/03 DTPA infusion Day 0 06/05/00 Day + 1Peripheral Stem Cell reinfusion Start G-CSF 5 µg/kg/d IV Day + 1

## 8.2 Pre-Transplant Therapy

a. Autologous Stem Cell Collection and Cryopreservation

All patients should have bone marrow aspiration and biopsy which show no microscopic evidence of lymphomatous involvement, or  $\leq 10\%$  involvement at the time of stem cell collection. In addition, cytogenetic studies, immunophenotyping, gene rearrangement should be done. Peripheral blood stem cells (PBSCs) will be collected via leukapheresis procedures that have been previously described. Patients will receive PBSCs collected after mobilization by: 1) growth factors, ie. G-CSF 10  $\mu$ g/kg/d or 2) chemotherapy with growth factors. A minimum of CD34+ cells, 3.0 x 10<sup>6</sup>/kg should be collected.

## b. Trimethoprim Sulfa

All patients should receive trimethoprim sulfa (one double-strength tablet PO bid) beginning day -8 through day -2 prior to PBSCT as prophylaxis against PCP. (The choice of trimethoprim sulfa as a prophylactic agent may be altered based on a history of sensitivity to this agent.) Dosing should be discontinued 48 hours prior to PBSC infusion because of potential myelosuppression.

c. CNS Prophylaxis

CNS prophylaxis is recommended for patients with mantle cell lymphoma or diffuse large cell lymphoma who had bone marrow involvement at diagnosis or at time of relapse. For patients with mantle cell lymphoma who have never received high-dose MTX, CNS prophylaxis with intrathecal chemotherapy should be given.

## 8.3 Radioimmunotherapy

- a. Rituxan is to be administered by slow intravenous infusion having been diluted to 1-4 mg/ml in saline. Initial infusion should be through a dedicated line at a rate of 50 mg/hr. If hypersensitivity or infusion-related events do not occur, escalate the infusion rate in 50 mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr. If hypersensitivity or infusion-related events develop, the infusion should be temporarily slowed or interrupted. The infusion can be continued at one-half the previous rate when symptoms abate.
- b. IDEC-In2B8 Administration Two mg of IDEC-In2B8 (5.0 mCi of <sup>111</sup>In) will be administered for the dosimetry portion of the protocol. The imaging dose will be administered over 10 minutes by slow IV injection immediately following the infusion of Rituxan. A .22 micron filter must be on the line between the patient and the infusion port. Flush the line with at least 10 mls of normal saline after the IDEC-In2B8 has been infused.
- c. IDEC-Y2B8 Administration IDEC-Y2B8 (40-100 mCi of <sup>90</sup>Y with 3.2 6.4 mg of antibody) will be administered for the therapy portion of the protocol. The yttrium will be combined with a dose of IDEC-In2B8 (5.0 mCi of <sup>111</sup>In) identical to the dosimetry dose. The combined radiopharmaceuticals will be administered

10/29/03

07/13/00

10/29/03

08/07/01

by controlled infusion pump over 20 minutes. A .22 micron filter must be on the line between the patient and the infusion port. Flush the line with at least 10 mls of normal saline after the IDEC-In/Y2B8 has been infused.

*d.* Bone marrow biopsy.

## 8.4 Chemotherapy

10/25/00, 12/20/00

VP-16 is to be administered as a single infusion on day -4. The dose is 40 or 60 a. mg/kg and is calculated on adjusted ideal body weight to be consistent with standard VP-16 dosing for transplant protocols. The drug is infused undiluted directly into a port of a double or triple lumen indwelling intravenous catheter, with a total infusion time of 4 hours. The drug is to be drawn into one or more plastic syringes and infused with a syringe infusion pump, placed in an evacuated bottle and infused through a pediatric infusion pump, or infused by gravity without a pump. Thus the total dose for a 70 kg patient would be 4,200 mg. At 20 mg/ml, the volume of VP-16 would be 210 ml. The rate of infusion would thus be 210 ml/240 minutes or 0.875 ml/minute. Appropriate anti-emetics and sedatives should be given before the infusion begins. Before, and 2 hours into, the infusion the patient is to receive 25 mg of diphenhydramine, and 100 mg of hydrocortisone to prevent allergic reactions. If necessary, diuretics may be given. The intravenous hydration should be continued before, during and after the VP-16. Since in rare cases metabolic acidosis has been observed after high dose VP-16, additional NaHCO3 may be needed.

10/29/03

b. Cyclophosphamide is administered at a total dose of 100 mg/kg given in one dose on day -2 and is calculated on ideal body weight. Adjustments to the ideal body weight calculation for overweight patients are permitted. For patients who are weigh less than 95% of ideal body weight, cyclophosphamide will be dosed according to actual body weight. The drug should be dissolved in about 250 cc of D5W and infused IV over two hours. Appropriate anti-emetics and sedatives should be given. To prevent hemorrhagic cystitis, all patients should receive hydration with intravenous fluids, according to institutional standards, at the rate of 3.0 l/m2/day beginning four hours prior to cyclophosphamide and continuing until 24 hours after cyclophosphamide. In addition, mesna at 40 mg/kg (based on ideal body weight) will be given immediately before cyclophosphamide (hr 0) and at 3, 6, 9, 12, 15, 18 and 21 hrs later for a total of 8 doses. Each dose of mesna will be given IV over 15 minutes.

06/05/00, 10/29/03, 06/16/04

c. DTPA is to be administered by continuous intravenous infusion through a port of a double or triple lumen indwelling intravenous catheter. The dose should be ≥ 250 mgs/m², but ≤ 500 mgs. The DTPA should be made up in normal saline and infused over 24 hours by infusion pump. No magnesium or other heavy metal should be given during the same time period. Two hours after the end of the DTPA infusion 1 ml of trace metal solution should be infused every eight hours for five days. This should be given by slow intravenous delivery or else as part of standard hyperalimentation. Urine samples will be collected every 12 hours for

72 hours beginning 24 hours prior to DTPA infusion.

## 07/13/00, 05/03/01 8.5 Peripheral Stem Cell Reinfusion

PBSCs will be thawed and infused according to standard guideline at approximately 72 hours after completion of cyclophosphamide.

## 8.6 Growth Factor Therapy

All patients will receive rh-G-CSF, 5 mcg/kg/day IV beginning on day +1, after PBSC infusion and continue daily until ANC >500 for 3 consecutive days.

## 8.7 Supportive Care:

07/13/00

All patients will be housed in private rooms during the period of granulocytopenia. Nonabsorbable antibiotics for gastrointestinal decontamination should be used according to institutional guideline. Trimethoprim-sulfamethoxazole will be administered from day -8 to day -2 and prophylaxis should be re-instituted when white blood cells are > 3000 and continued until 6 months post-transplant. Empiric broad spectrum antibiotics and parenteral nutrition should be used as clinically indicated. Low-dose amphotericin-B (0.1 to 0.2 mg/kg) should be administered on day +1 and continued daily until granulocytopenia resolves. All blood components should be irradiated to 1,500 cGy.

#### a. Access to Vessels

Prior to admission, during pre-transplant evaluation, all patients should have a permanent central catheter placed.

## b. Hyperalimentation

All patients will receive appropriate Hyperalimentation as soon as necessary after admission. The goal will be to prevent even a short duration of negative nitrogen balance.

## c. Platelet Transfusion

- 1. Indication. Platelets are transfused to prevent bleeding and an attempt is made to keep the circulating level greater than 20,000/mm3 at all times. This goal may be changed by the attending physician as clinically indicated.
- 2. Irradiation. All blood products (except the autologous stem cells) are irradiated with 1,500 cGy prior to infusion.

## d. Management of Fever/Infections

Treatment of patients on this protocol is not intended to restrict the freedom of the managing physician to treat suspected or documented infections. In neutropenic patients, however, the following guidelines should be followed.

1. All febrile, neutropenic patients should be treated with IV antibiotic(s), the choice

- of which should be guided by the patient's clinical history, institutional practices and subsequent culture results.
- 2. Patients with documented, invasive fungal infection or with persistent, unexplained fevers while neutropenic and on broad-spectrum antibiotic therapy should receive antifungal therapy with Amphotericin-B.

## 8.8 Criteria for Removal from Protocol Treatment

- a. Progression of disease.
- b. Patients may withdraw from study at any time for any reason.
- 8.9 All reasons for discontinuation of treatment must be documented in the Flow Sheets.
- **8.10** All patients will be followed for survival until death. Secondary malignancy monitoring on this protocol will be done through 5 years post HCT. After such time, secondary malignancy monitoring will be done by the Long Term Follow Up office.

#### 9.0 STUDY DESIGN AND RULES FOR DOSE ESCALATION

This is a phase I/II trial. For the phase I portion of the study, the rules for dose escalation, dose expansion, and termination of escalation are given in section 9.2. Prior to treatment with Y2B8, patients are required to undergo an imaging scan to verify that they have a favorable biodistribution. While waiting to assess toxicities in the initial cohort of 3 to 6 patients, additional patients who are determined to be eligible may be accrued at the unescalated dose level. The rationale for this is twofold. First, patients must be evaluated for distribution as soon as possible in order to have patients ready for timely accrual to the next dose level. If the dose escalation decision is delayed, the investigators want to treat the patients at the unescalated dose level so that their disease does not progress. Second, patients will be accrued to unescalated dose levels to avoid a loss of momentum in patient accrual. Modifications to the standard phase I design involving accrual of cohorts of 3-6 patients per dose level have been incorporated to appropriately handle the varying number of patients accrued to each dose level (see section 9.2). Study design considerations and targeted response rates for the phase II portion of the trial are given in section 9.3. Because the eligibility criteria are the same for both the phase I and the phase II portions of the trial, the patients treated at the dose level defined as the MTD from the phase I portion of the trial will count towards the accrual for the phase II portion of the trial.

#### 9.1 Dose Limiting Toxicity (DLT)

Dose limiting toxicity (DLT) in a given patient is defined as any grade III non-hematologic toxicity not reversible to grade II or less within 96 hours, or any grade IV non-hematologic toxicity. Toxicity will be graded according to the NCI Common Toxicity Criteria (CTC) version 2.0 and toxicity Module (Appendices I and II, http://ctep.info.nih.gov/ctc3/ctc.htm) with the addition of BMT Complex/Multi-Component Events (Appendix VI, http://ctep.info.nih.gov/ctc3/ctc.htm). To be evaluable for toxicity, a patient must receive a complete course of treatment and be observed for 6 weeks after the administration of Y2B8 or have experienced a DLT. All patients who are not evaluable for toxicity will be replaced.

05/03/01

# 9.2 Definition of Maximum Tolerated Dose (MTD) and DLT-Level and Rules for Dose Escalation

This trial differs from the standard phase I design in that additional patients beyond the standard 3 or 6 patients per dose level may be accrued to the current dose level while waiting to assess toxicities in the initial 3 or 6 patients. To this end, a decision rule has been added that incorporates toxicity information from the additional patients accrued to a dose level. As toxicity information on each additional patient accrued to the trial becomes available, the decision to escalate, de-escalate and expand the previous dose level, expand the current cohort or stop the trial will be evaluated. The decision rule (R) will be as follows: Let x = number of DLTs in n patients. Escalate to the next dose level if R = (x + 0.5) / (n + 2) is  $\leq 0.20$ . Stop accrual to a dose level if R > 0.30. Continue accrual to a dose level if R = 0.30. A minimum of three patients must be accrued to a dose level. As soon as 3 patients have been accrued to a dose level and toxicity has been assessed, escalation to the next level is allowed, provided that acceptable toxicity has been observed. If accrual to a dose level must be expanded due to toxicity, a minimum of 6 patients must be accrued to the expanded dose level.

Operationally, the rule is to close a dose level and de-escalate if 2 DLTs are observed among 6 or fewer patients, or if 3 DLTs are observed among any number of patients. The dose will be escalated if 0 DLTs are observed in 3 or more evaluated patients, if 1 DLT is observed in 6 or more evaluated patients, or if 2 DLTs are observed in 11 patients. At most, 11 patients will be accrued to a dose level. However, if a dose is escalated while toxicity follow-up is still outstanding for some patients, the accumulating results from the two dose levels may be pooled for the purpose of justifying the continued accrual to the higher dose.

Table 1 shows values for R based on different combinations of DLTs and numbers of patients. Values indicating continued accrual to the current dose are shown in bold.

Table 1

| | Nu | mber of DLTs | (x) |
|------------------------|------|--------------|------|
| Number of Patients (n) | 0 | 1 | 2 |
| 3 | 0.10 | 0.30 | 0.50 |
| 4 | 0.08 | 0.25 | 0.42 |
| 5 | 0.07 | 0.21 | 0.36 |
| 6 | 0.06 | 0.19 | 0.31 |
| 7 | 0.06 | 0.17 | 0.28 |
| 8 | 0.05 | 0.15 | 0.25 |
| 9 | 0.05 | 0.14 | 0.23 |
| 10 | 0.04 | 0.13 | 0.21 |
| 11 | 0.04 | 0.12 | 0.19 |

This criterion is the posterior mean with a beta (0.5, 1.5) prior, which has a smaller mean, but is no more informative than a flat prior. The criterion is consistent with the conventional rule of expanding a dose level to six patients if 1 out of 3 patients experience DLT and stopping if 2 or

more patients out of 6 treated at the same dose level experience DLT. The proposed criterion rationalizes the conventional design in order to rationally extend if to larger numbers of patients per dose level. The rationalization is that a dose level is opened with a weak prior expectation of a 25% DLT rate, and the dose is escalated or de-escalated as the accumulating data indicate a rate below 20% or above 30%.

The phase I portion of the trial will be closed when 6 patients have been accrued to the highest dose level below the DLT level with at most 1 patient experiencing DLT or when 11 patients have been accrued with at most 2 patients experiencing DLT. This dose level will be defined as the MTD.

To demonstrate an application of the escalation rule, consider the following examples:

Example 1: Three patients are accrued to dose level 1. A fourth patient is accrued to the trial prior to assessment of toxicity for the third patient and is therefore also treated at dose level 1. No DLTs are observed in the first 3 patients such that the fifth patient is accrued to dose level 2 and subsequent to this the fourth patient accrued to dose level 1 experiences a DLT. With 1 DLT in four patients, from Table 1 the value for R is 0.25 therefore accrual to dose level 2 must be halted such that accrual to dose level 1 can be expanded. Six patients will need to be accrued with at most 1 out of 6 patients experiencing DLT in order for accrual to dose level 2 to resume. The patient treated at dose level 2 may be counted among the required 6 patients if no DLT is encountered.

Example 2: Dose level 3 is expanded such that 6 patients are accrued. A seventh patient is accrued to the trial prior to assessment of toxicity for the sixth patient and is therefore also treated at dose level 3. Only one DLT is observed in the first 6 patients such that the eighth patient is accrued to dose level 4 and subsequent to this the seventh patient accrued to dose level 3 experiences a DLT. With 2 DLTs in seven patients, from Table 1 the value for R is 0.28 therefore accrual to dose level 4 must be halted so that accrual to dose level 3 can be expanded. Eleven patients (including the patient treated at dose level 4) will need to be accrued to dose level 3 (or above) with at most 2 patients experiencing DLTs in order for accrual to dose level 4 to resume. Two DLTs among 11 patients corresponds to R = 0.19 which is consistent with 1 DLT among 6 patients. A maximum of 11 patients can be accrued to a single dose level.

## 9.3 Design Considerations for the Phase II Trial

All patients accrued to the dose level established to be the MTD will be included in the assessment of response for the phase II portion of the trial. The primary goal of this portion of the trial is to obtain estimates of the efficacy of IDEC-Y2B8 in combination with high-dose etoposide and cyclophosphamide followed by ASCT for treatment of patients with relapsed and refractory NHL. A minimum of 17 and a maximum of 37 patients will be accrued to this portion of the trial. Justification for the sample size as well as a description of the study design for the phase II portion of the trial is provided in section 12.0.

10/29/03

10/29/03 10/29/03 08/07/01, 10/2 10/29/03 10/29/03

08/07/01

10/29/03 08/07/01, 05/3 05/03/01

05/30/02 05/30/02

08/07/01, 10/2 04/06/04

06/16/04 06/16/04 06/05/00

05/30/02, 10/29/03 10/29/03

10/29/03 10/29/03

#### 10.0 STUDY CALENDAR - PREPARATIVE REGIMEN AND PBSCT

| REQUIRED STUDIES | Pre<br>Study | DAY<br>-21 | DAY<br>-14 | DAY<br>-7 | DAY<br>-4 | DAY<br>-2 | DAY<br>0 | DAY<br>7 | DAY<br>14 | DAY<br>30 | DAY<br>60 | DAY<br>100 | DAY<br>180 | YR<br>1 | YR<br>2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PHYSICAL | | | | | | | | | | | | | | | |
| H & PE | X | | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> |
| Weight and KPS | X | | | X | | | X | | | X | X | X | X | X | X <sup>\$</sup> |
| Tumor Assessment | X | | | | | | | | | X | | | X | X | X <sup>\$</sup> |
| Toxicity Notation | | | | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> | X <sup>\$</sup> |
| LABORATORY | | | | | | | | | | | | | | | |
| CBC/Platelets | X | | | X | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> |
| Differential <sup>¥</sup> | X | | | X | | | | X | X | X | X | X | X | X | X <sup>\$</sup> |
| HAMA/HACA | X | | | | | | | | | | X | X | X" | X | |
| Comp Metabolic Panel + LDH | X | | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> |
| Magnesium | X | | X | X | X | X | X | X | X | X | | | | | |
| PT/PTT | X | | | | | | | | | | | | | | |
| Immunoglobulin Levels | X | | | | | | | | | X | | X | X | X | |
| Peripheral Blood Mononuclear<br>Immunophenotyping | X | | | | | | | | | X | | X | X | X | |
| CMV Titer | X | | | | | | | | | | | | | | |
| Hepatitis Profile | X | | | | | | | | | | | | | | |
| Herpes Simplex | X | | | | | | | | | | | | | | |
| HIV Antibody | X | | | | | | | | | | | | | | |
| BM <sup>%</sup> , # | X | | | Χ^ | | | | | | | | X | | X | X |
| Creatinine Clearance | | | | | | | | | | | | | X | X | |
| X-RAYS AND SCANS | | | | | | | | | | | | | | | |
| Chest X-ray or CT Chest | X | | | X | | | X | | X | X | | X | X | X | X <sup>&amp;</sup> |
| CT scans*, + | X | | | | | | | | | X | | X | X | X | X <sup>&amp;</sup> |
| EKG | X | | | | | | | | | | | | | X | |
| MUGA or ECHO | X | | | | | | | | | | | | X | X | |
| DLCO/FEV1 | X | | | | | | | | | | | | X | X | |
| Ga 67 Scan and/or FDG-PET Scan | $X^{\phi}$ | | | | | | | | | $X^{\Diamond}$ | | | X | X | |
| TREATMENT | | | | | | | | | | | | | | | |
| Stem Collections | X | | | | | | | | | | | | | | |
| IDEC-In2B8 | | X | X | | | | | | | | | | | | |
| IDEC-Y2B8 | | | X | | | | | | | | | | | | |
| Rituxan | | X | X | | | | | | | | | | | | |
| VP-16 | | | | | X | | | | | | | | | | |
| Cyclophosphamide | | | | | | X | | | | | | | | | |
| PBSCT | | | | | | | X <sup>§</sup> | | | | | | | | |
| G-CSF | | | | | | | X§ | | | | | | | | |
| DTPA | | | | | | | X | | | | | | | | |

10/29/03 (delete @.06/20/07) & restaging at Day 100, at 6 months then follow-up evaluation every six months for three years, and then yearly up to 5 yrs post BMT

% bone marrow aspiration and biopsy, cytogenetic study, immunophenotyping and gene rearrangement

05/30/02, 06/20/07 # Follow-up bone marrow is required at day 180, yr 1 up to 5 yrs post BMT.

+ For pts in CR at time of transplant, CT scans to be done between days 30 and 100.

« Day 180 HAMA/HACA acceptable between days 150 and 210

¢ Pre-study PET scan should be done 14 days after stem cell collection to avoid GCSF enhancement effect

¥ ANC is acceptable in lieu of differential

06/16/04 § Day +1

<sup>\$</sup> All late complications such as cataracts formation and occurrence of second malignancies must be documented and reported.

<sup>\*</sup> CT scans of chest, abdomen and pelvis as indicated

#### 11.0 CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS

## **Definitions**

- a. Measurable Disease: Bidimensionally measurable lesions with clearly defined margins by: 1) medical photograph (skin or oral lesion), or plain x-ray with at least one diameter .5 cm or greater (bone lesions are not included) or, 2) CT, MRI or other imaging scan with both diameters greater than the distance between cuts of the imaging study, or 3) palpation with both diameters 2 cm or greater.
- b. Evaluable Disease: Unidimensionally measurable lesions, masses with margins not clearly defined, lesions with both diameters less than 0.5 cm, lesions on scan with either diameter smaller than the distance between cuts, palpable lesions with either diameter less than 2 cm, bone disease.
- c. Non-Evaluable Diseases: Pleural effusions, ascites, disease documented by indirect evidence only (e.g., by lab values).
- d. Objective Status, To Be Recorded at Each Evaluation: If an organ has too many measurable lesions to measure at each evaluation, choose three to be followed before the patient is entered on study. The remaining measurable lesions in that organ will be considered evaluable for the purpose of objective status determination. Unless progression is observed, objective status can only be determined when ALL is measurable and evaluable sites and lesions are assessed.

## 11.1 Complete Response (CR)

Complete disappearance of all measurable evidence of non-evaluable disease. No new lesions. No disease related symptoms. No evidence of non-evaluable disease, including normalization of markers and other abnormal lab values. All measurable, evaluable and non-evaluable lesions and sites must be assessed using the same techniques as baseline. Refers to clinical CR-when restaging surgery is required, a separate pathologic response variable is defined.

## 11.2 Partial Response (PR)

Applies only to patients with at least one measurable lesion. Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. All measurable and evaluable lesions and sites must be assessed using the same techniques as baseline.

#### 11.3 Stable Disease (SD)

Does not qualify for CR, PR or Progression. All measurable and evaluable sites and lesions must be assessed using the same techniques as baseline.

#### 11.4 Progressive Disease (PD)

50% increase or an increase of 10 cm<sup>2</sup> (whichever is smaller) in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same

05/30/02

techniques as baseline, OR clear worsening of any evaluable disease, OR reappearance of any lesion which had disappeared, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). For "scan only" bone disease, increased uptake does not constitute clear worsening. Worsening of existing non-evaluable disease not constitute progression.

#### 11.5 Relapse

Relapse is defined as the re-appearance of any clinical evidence of lymphoma in a patient who has had a CR. Relapse for partial responders are defined as progressive disease relative to disease status during the partial remission.

## 11.6 Duration of Response

This is measured from the documented beginning of response (CR or PR)

## 11.7 Performance Status

Patients will be graded according to the current Performance Status Scales/Scores (Appendix IV).

## 11.8 Time to Progression

From date of registration to date of first observation of progressive disease or death due to any cause.

#### 11.9 Time to Death

From date of registration to date of death due to any cause.

#### 12.0 STATISTICAL CONSIDERATIONS

## 12.1 Study Design and Justification of Sample Size

The definition of dose limiting toxicity is given in section 6.1. The maximum tolerated dose is defined in section 6.2. The number of patients to be treated at each dose level examined in the phase I trial as well as the rules for dose escalation is given in section 6.2.

The phase II portion of the study will follow a two-stage minimax design suggested by Simon (1). It is assumed that a true response rate less than 20% would not warrant further study of this agent. It is also assumed that a response rate of 40% would be considered promising for further studies in these patients. In the first stage, seventeen evaluable patients will be entered. If less than four responses are observed, the accrual will stop with the conclusion that the regimen is not promising for further study. If four or more responses are observed in the first 17 patients, additional 20 patients will be accrued during the second stage of the study. Eleven or more responses out of 37 patients will be considered as evidence warranting further study of the regimen providing other factors, such as toxicity and survival, also appear favorable. If less than 11 responses out of 37 patients are observed, further study of the regimen would not be warranted.

The probability of falsely declaring an agent with a 20% response probability as warranting further

08/07/01

study is 0.10 (alpha) and the probability of correctly declaring an agent with a 40% response probability as warranting further study is 0.90 (power). With 37 patients the true probability of response can be estimated with a maximum standard error equal to 0.08.

The phase I portion study is expected to accrue a minimum of 15-18 evaluable patients and a maximum of 30. The phase II portion of the study will accrue a minimum of 17 patients and a maximum of 37 patients, of which at least six of these patients will have been included in the phase I portion of the study. It should take approximately 24-36 months to complete both the phase I and phase II portions of this trial.

## 12.2 Analysis of Clinical Endpoints

Patients will be considered evaluable for response and evaluable for toxicity as outlined in section 11.0. The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI Common Toxicity Criteria and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course. Baseline information (e.g. the extent of prior therapy) and demographic information will be presented, as well, to describe the patients treated in the phase I portion of the study. All responses will be reported from the phase I portion of the study

Response rates and duration of response will be estimated for the phase II portion of survival. Confidence intervals for the response rate will be established by calculating exact 95% confidence limits for a binomial parameter. The duration of overall and disease-free survival of the patient will be estimated using the product-limit method of Kaplan and Meier.

#### 13.0 REGISTRATION GUIDELINES

Once a signed, written informed consent has been obtained and all pretreatment evaluations have been performed, patients will be entered on study, after review of patient eligibility criteria by the assigned Data Manager from the City of Hope Department of Biostatistics. Patients may be screened for registration by calling the Department of Biostatistics, ext. 62468.

#### 14.0 RECORDS TO BE KEPT AND DATA SUBMISSION SCHEDULE

## 14.1 Confidentiality of Records

The original data collection forms will be stored in secure cabinets in the Department of Biostatistics. All radioimmunotherapy associated data will be kept in the Department of Radioimmunotherapy.

#### 14.2 Patient Consent Form

At the time of registration, signed and dated copies of the patient Informed Consent form with the Human Rights must be available (for patient, chart, and Biostatistics Office).

08/07/01

#### 15.0 GENDER AND MINORITIES

# 15.1 Planned Gender and Minority Inclusion for Transplant Patients with Intermediate Grade Lymphoma at City of Hope

| | American<br>Indian or | Asian or<br>Pacific | Black,<br>not of | Hispanic | White,<br>not of | White,<br>Hispanic | Other or<br>Unknown | Total |
|---|---|---|---|---|---|---|---|---|
| | Alaskan<br>Native | Islander | Hispanic<br>Origin | | Hispanic<br>Origin | or not-<br>Hispanic<br>Unknown | | |
| Female | 0% | 9% | 4% | 16% | 54% | 17% | 0% | 100% |
| Male | 0% | 5% | 2% | 20% | 60% | 12% | 1% | 100% |
| Unknown | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |

# 15.2 Actual Gender and Minority Inclusion for Transplant Patients with Intermediate Grade Lymphoma at City of Hope

| | American | Asian or | Black, | Hispanic | White, | White, | Other or | Total |
|---|---|---|---|---|---|---|---|---|
| | Indian or | Pacific | not of | | not of | Hispanic | Unknown | |
| | Alaskan | Islander | Hispanic | | Hispanic | or not- | | |
| | Native | | Origin | | Origin | Hispanic | | |
| | | | | | | Unknown | | |
| Female | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |
| Male | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |
| Unknown | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |

#### 16.0 DATA MANAGEMENT

Clinical Statistics maintains a patient database at City of Hope Medical Center, Department of Biostatistics to allow storage and retrieval of patient data collected from a wide variety of sources. The investigator will ensure that data collected conform to all established guidelines for coding, collection, key-entry, and verification. All patients are assigned a unique patient number to assure patient confidentiality. Any publications or presentations refer to patient by unique patient number, not name. The licensed medical records department, affiliated with the institution where the patient receives medical care, maintains all original inpatient and outpatient chart documents. Patient research files are kept in a locked room. They are maintained by the COHMC data collection staff. Access is restricted to personnel authorized by the Division of Clinical Research.

#### 17.0 ETHICAL AND REGULATORY CONSIDERATIONS

This study is to be approved by the Institutional Review Board according to City of Hope ethical and regulatory guidelines. All patients will have signed an informed consent for participation in research activities, and will have been given a copy of the Experimental Subject's Bill of Rights.

When results of this study are reported in medical journals or at meetings, identification of those taking part will be withheld. Medical records of patients will be maintained in strictest confidence,

according to current legal requirements. However, they will be made available for review, as required by the Food and Drug Administration (FDA) or other authorized users such as the National Cancer Institute (NCI), under the guidelines established by the Federal Privacy Act, or IDEC Pharmaceuticals Corporation.

#### 18.0 REFERENCES

- 1. Parker SL, Tong T, Bolden S, Wingo PA: Cancer Statistics, 1997 [published erratum appears in CA Cancer J Clin 1997 Mar-Apr;47(2):68]. CA.Cancer J.Clin. 47:5, 1997
- 2. Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CAJ, Miller TP: Comparison of a Standard Regimen (CHOP) with Three Intensive Chemotherapy Regimens for Advanced Non-Hodgkin's Lymphoma [see comments]. N.Engl.J.Med. 328:1002, 1993
- 3. Vose JM, Anderson JR, Kessinger A, Bierman PJ, Coccia P, Reed EC, Gordon B, Armitage JO: High-Dose Chemotherapy and Autologous Hematopoietic Stem-Cell Transplantation for Aggressive Non-Hodgkin's Lymphoma [see comments]. J.Clin.Oncol. 11:1846, 1993
- 4. Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL: Autologous Bone Marrow Transplantation as Compared with Salvage Chemotherapy in Relapses of Chemotherapy-Sensitive Non-Hodgkin's Lymphoma [see comments]. N.Engl.J.Med. 333:1540, 1995
- 5. Bierman PJ, Vose JM, Anderson JR, Bishop MR, Kessinger A, Armitage JO: High-Dose Therapy with Autologous Hematopoietic Rescue for Follicular Low-Grade Non-Hodgkin's Lymphoma. J.Clin.Oncol. 15:445, 1997
- 6. Nademanee A, Schmidt GM, O'Donnell MR, Snyder DS, Parker PM, Stein A, Smith E, Molina A, Wong KK, Stepan DE, Margolin KA, Somlo G, Raschko J, Sniecinski I, Lipsett JA, Dagis A, Niland JC, Forman SJ: Fractionated Total Body Irradiation (FTBI), High-Dose Etoposide (VP-16) and Cyclophosphamide (CY) Followed by Autologous Bone Marrow Transplantation (ABMT): The Results in 110 Patients with Non-Hodgkin's Lymphoma (NHL). Blood 82:143a (559), 1993 (abstr.)
- 7. Horning SJ, Negrin RS, Chao JC, Long GD, Hoppe RT, Blume KG: Fractionated Total-Body Irradiation, Etoposide, and Cyclophosphamide Plus Autografting in Hodgkin's Disease and Non-Hodgkin's Lymphoma. J.Clin.Oncol. 12:2552, 1994
- 8. Weaver CH, Petersen FB, Appelbaum FR, Bensinger WI, Press O, Martin P, Sandmaier B, Deeg HJ, Hansen JA, Brunvand M: High-Dose Fractionated Total-Body Irradiation, Etoposide, and Cyclophosphamide Followed by Autologous Stem-Cell Support in Patients with Malignant Lymphoma. J.Clin.Oncol. 12:2559, 1994
- 9. Maloney DG, Grillo-Lopez AJ, White CA, Bodkin D, Schilder RJ, Neidhart JA, Janakiraman N, Foon KA, Liles TM, Dallaire BK, Wey K, Royston I, Davis T, Levy R: IDEC-C2B8 (Rituximab) Anti-CD20 Monoclonal Antibody Therapy in Patients With Relapsed Low-Grade Non-Hodgkin's Lymphoma. Blood 90:2188, 1997
- McLaughlin P, Grillo-López AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK: Rituximab Chimeric Anti-CD20 Monoclonal Antibody Therapy for Relapsed Indolent Lymphoma: Half of Patients Respond to a Four-Dose Treatment Program. Journal of Clinical Oncology 16:2825, 1998
- 11. Czuczman M, Grillo-López AJ, White CA, Saleh M, Gordon L, LoBuglio AF, Jonas C, Dallaire B, Varns C: IDEC-C2B8/CHOP Chemoimmunotherapy in Patients With Low-

- Grade Lymphoma: Clinical and BCL-2 (PCR) Final Results. Blood 88:453a (1799), 1996 (abstr.)
- 12. Kaminski MS, Zasadny KR, Francis IR, Milik AW, Ross CW, Moon SD, Crawford SM, Burgess JM, Petry NA, Butchko GM: Radioimmunotherapy of B-Cell Lymphoma with [131][Anti-B1 (Anti-CD20) Antibody. N.Engl.J.Med. 329:459, 1993
- 13. Stagg R, Wahl RL, Estes J, Tidmarsh G, Kroll S, Shochat D, Zasadny K, Kaminski MS: Phase I/II Study of Iodine-131 Anti-B1 Antibody for Non-Hodgkin's Lymphoma (NHL): Final Results. Proceedings of ASCO 17:39a (150), 1998 (abstr.)
- 14. Vose J, Saleh M, Lister A, Rohatiner A, Knox S, Radford J, Zelenetz AD, Stagg R, Tidmarsh G, Wahl R, Kaminski MS: Iodine-131 Anti-B1 Antibody for Non-Hodgkin's Lymphoma (NHL): Overall Clinical Trial Experience. Proceedings of ASCO 17:10a (38), 1998 (abstr.)
- 15. Press OW, Eary JF, Appelbaum FR, Martin PJ, Badger CC, Nelp WB, Glenn S, Butchko G, Fisher D, Porter B: Radiolabeled-Antibody Therapy of B-Cell Lymphoma With Autologous Bone Marrow Support [see comments]. N.Engl.J.Med. 329:1219, 1993
- 16. Press O, Eary J, Liu S, Petersdorf S, Bush S, Durack L, Martin P, Maloney D, Matthews D, Fisher D, Gooley T, Appelbaum F, Bernstein I: A Phase I/II Trial of High Dose Iodine-131-Anti-B1 (Anti-CD20) Monoclonal Antibody, Etoposide, Cyclophosphamide, and Autologous Stem Cell Transplantation for Patients With Relapsed B Cell Lymphomas. Proceedings of ASCO 17:3a (9), 1998 (abstr.)
- 17. Knox SJ, Goris ML, Trisler K, Negrin R, Davis T, Liles TM, Grillo-Lopez A, Chinn P, Varns C, Ning S, Fowler S, Deb N, Becker M, Marquez C, Levy R: Yttrium-90-Labeled Anti-CD20 Monoclonal Antibody Therapy of Recurrent B-Cell Lymphoma. Clin.Cancer Res. 2:457, 1996
- 18. Witzig T, Wiseman G, White CA, Solinger A, Gordon L, Raubitschek A, Emmanoulides C, Royston I, Parker E, Chinn P, Grillo-López A: IDEC-Y2B8 <sup>90</sup>Yttrium Anti-CD20 Radioimmunotherapy of Relapsed Non-Hodgkin's Lymphoma (NHL): Interim Results of a Phase I/II Trial. Blood 90:586a (2606), 1997 (abstr.)
- 19. Wiseman GA, Solinger AM, Grillo-López A, Stabin M, Dunn WL, Witzig TE, Spies S, Gordon L, Raubitschek A, Margolin K, Karvelis K, Janakiraman N, Silverman DH, Emmanoulides C, Royston I, Chinn P, Parker E, Carter W, White CA: IDEC-Y2B8 (90 Y Conjugated Anti-CD20) Dosimetry Calculated From 111 In Anti-CD20 in Patients With Low and Intermediate Grade B-Cell Non-Hodgkin's Lymphoma (NHL) Emphasis on Bone Marrow (BM). Blood 90:510a (2273), 1997 (abstr.)
- Witzig TE, White CA, Wiseman GA, Gordon LI, Emmanoulides C, Raubitschek A, Janakiraman N, Gutheil J, Schilder RJ, Spies S, Silverman DH, Parker E, and Grillo-López A: Phase I/II Trial of Yttrium 90 Ibritumomab Tiuxetan (IDEC-Y2B8) Radioimmunotherapy for Treatment of Relapsed or Refractory CD20 Positive B-Cell Mon-Hodgkin's Lymphoma. Submitted 1999.

## Appendix I Common Toxicity Criteria (CTC)

## FINAL 1/30/98

CTC Version 2.0

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| ALLERGY/IMMUNOLOGY | | | | | |
| Allergic reaction/<br>hypersensitivity<br>(including drug<br>fever) | none | transient rash,<br>drug fever <<br>38°C (<100.4°F) | urticaria, drug fever ≥ 38°C (≥100.4°F), and/or asymptomatic bronchospasm | symptomatic<br>bronchospasm,<br>requiring<br>parenteral<br>medication(s),<br>with or without<br>urticaria; allergy-<br>related<br>edema/angioede<br>ma | anaphylaxis |
| DERMATOLOGY/SI | | of other mannestatio | ns of an affergic of n | ypersensitivity reacti | on, is graded in the |
| Allergic rhinitis<br>(including sneezing,<br>nasal stuffiness,<br>postnasal drip) | none | mild, not<br>requiring<br>treatment | moderate,<br>requiring<br>treatment | - | - |
| Autoimmune reaction | none | serologic or other evidence of autoimmune reaction but patient is asymptomatic (e.g., vitiligo), all organ function is normal and no treatment is required | evidence of autoimmune reaction involving a non- essential organ or function (e.g., hypothyroidism), requiring treatment other than immunosuppressi ve drugs | reversible autoimmune reaction involving function of a major organ or other toxicity (e.g., transient colitis or anemia), requiring short- term immunosuppressi ve treatment | autoimmune reaction causing major grade 4 organ dysfunction; progressive and irreversible reaction; long- term administration of high-dose immuno- suppressive therapy required |
| Also consider Hypothy<br>Serum sickness | | Hemoglobin, Hemo | IVSIS. | procent | |
| Urticaria is graded in t manifestations of aller | | | | | |
| Vasculitis | none | mild, not<br>requiring<br>treatment | symptomatic,<br>requiring<br>medication | requiring steroids | ischemic changes<br>or requiring<br>amputation |
| Allergy/Immunology -Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | | AUDITORY | //HEARING | | |
| Conductive hearing lo | | iddle ear/hearing in t | | ARING category. | |
| Earache is graded in th | | | | | |
| External auditory canal Note: Changes associa DERMATOLOGY/SR | | external otitis with erythema or dry desquamation to external ear (pin | external otitis with moist desquamation nae) are graded unde | external otitis<br>with discharge,<br>mastoiditis<br>or Radiation dermatit | necrosis of the canal soft tissue or bone is in the |
| Inner ear/hearing | normal | hearing loss on audiometry only | tinnitus or<br>hearing loss, not<br>requiring hearing<br>aid or treatment | tinnitus or<br>hearing loss,<br>correctable with<br>hearing aid or<br>treatment | severe unilateral<br>or bilateral<br>hearing loss<br>(deafness), not<br>correctable |
| Middle ear/hearing | normal | serous otitis<br>without<br>subjective<br>decrease in<br>hearing | serous otitis or<br>infection<br>requiring medical<br>intervention;<br>subjective<br>decrease in<br>hearing; rupture<br>of tympanic<br>membrane with<br>discharge | otitis with<br>discharge,<br>mastoiditis or<br>conductive<br>hearing loss | necrosis of the<br>canal soft tissue<br>or bone |
| Auditory/Hearing-<br>Other<br>(Specify, | normal | mild | moderate | severe | life-threatening or disabling |
| ) | | DV 00D 700 | | | |
| Dono morrow | named for | | ME MARROW<br>madarataly | garramaler | anlagia an >6 |
| Bone marrow cellularity | normal for age | mildly<br>hypocellular or<br>25% reduction<br>from normal<br>cellularity for age | moderately hypocellular or >25 - \le 50\% reduction from normal cellularity for age or >2 but <4 weeks to recovery of normal bone marrow cellularity | severely hypocellular or >50 - \le 75\% reduction in cellularity for age or 4 - 6 weeks to recovery of normal bone marrow cellularity | aplasia or >6<br>weeks to recovery<br>of normal bone<br>marrow<br>cellularity |
| Normal ranges:<br>children (≤ 18 years)<br>younger adults (19-<br>59) | 90% cellularity average 60-70% cellularity average | | | | |
| older adults (≥ 60 years) Note: Grade Bone mar | 50% cellularity average | nly for changes relate | ed to treatment not d | isease. | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| CD4 count | WNL | < LLN - 500/mm <sup>3</sup> | $200 - < 500/\text{mm}^3$ | $\frac{3}{50 - < 200/\text{mm}^3}$ | < 50/mm <sup>3</sup> |
| Haptoglobin | normal | decreased | - | absent | - |
| Hemoglobin (Hgb) | WNL | < LLN - 10.0 g/dl<br>< LLN - 100 g/L<br>< LLN - 6.2<br>mmol/L | 8.0 - < 10.0 g/dl<br>80 - < 100 g/L<br>4.9 - < 6.2<br>mmol/L | 6.5 - < 8.0 g/dl<br>65 - 80 g/L<br>4.0 - < 4.9<br>mmol/L | < 6.5 g/dl<br>< 65 g/L<br>< 4.0 mmol/L |
| Note: The following cr | riteria may be use | | | | isic process if the |
| protocol so specifies. | J | | | , | • |
| For leukemia studies<br>or bone marrow<br>infiltrative/<br>myelophthisic<br>processes | WNL | 10 - <25%<br>decrease from<br>pretreatment | 25 - <50%<br>decrease from<br>pretreatment | 50 - <75%<br>decrease from<br>pretreatment | ≥75% decrease from pretreatment |
| Hemolysis (e.g.,<br>immune hemolytic<br>anemia, drug-related<br>hemolysis, other) | none | only laboratory<br>evidence of<br>hemolysis [e.g.,<br>direct<br>antiglobulin test<br>(DAT, Coombs')<br>schistocytes] | evidence of red<br>cell destruction<br>and ≥ 2gm<br>decrease in<br>hemoglobin, no<br>transfusion | requiring<br>transfusion<br>and/or medical<br>intervention (e.g.,<br>steroids) | catastrophic<br>consequences of<br>hemolysis (e.g.,<br>renal failure,<br>hypotension,<br>bronchospasm,<br>emergency<br>splenectomy) |
| Also consider Haptogl | | | | | 10 109 /7 |
| Leukocytes (total WBC) | WNL | < LLN - 3.0 x 10 <sup>2</sup><br>/L<br>< LLN -<br>3000/mm <sup>3</sup> | $\geq 2.0 - < 3.0 \times 10^9$ /L $\geq 2000 - < 3000/\text{mm}^3$ | $\geq 1.0 - < 2.0 \times 10^9$ /L $\geq 1000 - < 2000/\text{mm}^3$ | < 1.0 x 10 <sup>9</sup> /L<br>< 1000/mm <sup>3</sup> |
| For BMT studies: | WNL | ≥2.0 - <3.0 X<br>10 <sup>9</sup> /L<br>≥2000 -<br><3000/mm <sup>3</sup> | ≥1.0 - <2.0 x 10 <sup>9</sup><br>/L ≥1000 -<br><2000/mm <sup>3</sup> | $\geq 0.5 - < 1.0 \times 10^9$<br>/L $\geq 500 - < 1000/\text{mm}^3$ | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> |
| Note: The following cr<br>specifies. | riteria using age, | race and sex normal | l values may be used | for pediatric studies | if the protocol so |
| , , | | ≥75 - <100%<br>LLN | ≥50 - <75% LLN | ≥25 - 50% LLN | <25% LLN |
| Lymphopenia | WNL | <lln -="" 1.0="" 10<sup="" x="">9 /L <lln -="" 1000="" mm<sup="">3</lln></lln> | /L<br>≥500 -<br><1000/mm <sup>3</sup> | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> | - |
| Note: The following cr<br>specifies. | riteria using age, | | | | |
| Neutrophils/granuloc ytes | WNL | ≥75-<100%LLN<br>≥1.5 - <2.0 x 10 <sup>9</sup><br>/L | ≥50-<75%LLN<br>≥1.0 - <1.5 x 10 <sup>9</sup><br>/L | ≥25-<50%LLN<br>≥0.5 - <1.0 x 10 <sup>9</sup><br>/L | <0.5 x 10 <sup>9</sup> /L<br><500/mm <sup>3</sup> |
| (ANC/AGC) | | $\geq 1500 - <2000/\text{mm}^3$ | $\geq 1000 - <1500/\text{mm}^3$ | ≥500 -<br><1000/mm <sup>3</sup> | |
| For BMT: | WNL | $\geq 1.0 - < 1.5 \times 10^9$ /L $\geq 1000 - < 1500/\text{mm}^3$ | $\geq 0.5 - < 1.0 \times 10^9$<br>/L<br>$\geq 500 - < 1000/\text{mm}^3$ | $\geq 0.1 - < 0.5 \times 10^9$<br>/L<br>$\geq 100 - < 500/\text{mm}^3$ | <0.1 x 10 <sup>9</sup> /L<br><100/mm <sup>3</sup> |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Note: The following criteria may be used for leukemia studies or bone marrow infiltrative/myelophthisic process if the protocol so specifies. | | | | | |
| For leukemia studies<br>or bone marrow<br>infiltrative/<br>myelophthisic<br>process | WNL | 10 - <25%<br>decrease from<br>baseline | 25 - <50%<br>decrease from<br>baseline | 50 - <75%<br>decrease from<br>baseline | ≥75% decrease from baseline |
| Platelets | WNL | < LLN - <75.0 x<br>10 <sup>9</sup> /L<br>< LLN -<br>75000/mm <sup>3</sup> | ≥50.0 - < 75.0 x<br>10 <sup>9</sup> /L<br>≥50000 - <<br>75000/mm <sup>3</sup> | $\geq 10.0 - < 50.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 10000 - <$<br>$50000 / \text{mm}^3$ | < 10.0 x 10 <sup>9</sup> /L<br>< 10000/mm <sup>3</sup> |
| For BMT: | WNL | ≥50.0 - <75.0 x<br>10 <sup>9</sup> /L<br>≥50000 -<br><75000/mm <sup>3</sup> | $\geq 20.0 - <50.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 20000 - <50000 / \text{mm}^3$ | $\geq 10.0 - <20.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 10000 - <20000/\text{mm}^3$ | <10.0 x 10 <sup>9</sup> /L<br><10000/mm <sup>3</sup> |
| Note: The following cr<br>protocol so specifies. | riteria may be use | | | | nisic process if the |
| For leukemia studies or bone marrow infiltrative/ myelophthisic process | WNL | 10 - <25%<br>decrease from<br>baseline | 25 - <50%<br>decrease from<br>baseline | 50 - <75%<br>decrease from<br>baseline | ≥75% decrease from baseline |
| Transfusion:<br>Platelets | none | - | - | yes | platelet transfusions and other measures required to improve platelet increment; platelet transfusion refractoriness associated with life-threatening bleeding. (e.g., HLA or cross matched platelet transfusions) |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| For BMT: | none | 1 platelet<br>transfusion in 24<br>hours | 2 platelet<br>transfusions in 24<br>hours | ≥3 platelet transfusions in 24 hours | platelet transfusions and other measures required to improve platelet increment; platelet transfusion refractoriness associated with life-threatening bleeding. (e.g., HLA or cross matched platelet transfusions) |
| Also consider Platelet | | | | | |
| Transfusion: pRBCs | none | - | -<br>- | Yes | - |
| For BMT: | none | ≤2 u pRBC<br>(≤15cc/kg) in 24<br>hours elective or<br>planned | 3 u pRBC (>15<br>≤30cc/kg) in 24<br>hours elective or<br>planned | ≥4 u pRBC<br>(>30cc/kg) in 24<br>hours | hemorrhage or<br>hemolysis<br>associated with<br>life-threatening<br>anemia; medical<br>intervention<br>required to<br>improve<br>hemoglobin |
| Also consider Hemog | lobin. | | | | |
| Blood/Bone<br>Marrow-Other<br>(Specify, | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | CARDIOVASCULA | AR (ARRHYTHMIA | <b>A</b> ) | |
| Conduction<br>abnormality/<br>Atrioventricular<br>heart block | none | asymptomatic,<br>not requiring<br>treatment (e.g.,<br>Mobitz type I<br>second-degree<br>AV block,<br>Wenckebach) | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment (e.g., Mobitz type II second-degree AV block, third-degree AV block) | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| Nodal/junctional<br>arrhythmia/dysrhyth<br>mia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| Palpitations Note: Grade palpitation | none ons only in the ab | present sence of a documente | -<br>ed arrhythmia | - | - |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Prolonged QTc<br>interval (QTc > 0.48<br>seconds) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| Sinus bradycardia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| Sinus tachycardia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment of<br>underlying cause | - |
| Supraventricular<br>arrhythmias<br>(SVT/atrial<br>fibrillation/ flutter) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| | | NEUROLOGY categor | | | |
| Vasovagal episode | none | - | present without<br>loss of<br>consciousness | present with loss<br>of consciousness | - |
| Ventricular<br>arrhythmia<br>(PVCs/bigeminy/trig<br>eminy/<br>ventricular<br>tachycardia) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| Cardiovascular/ Arrhythmia-Other (Specify, | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic, and<br>requiring<br>treatment of<br>underlying cause | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) |
| | | CARDIOVASCU | JLAR (GENERAL) | | |
| Acute vascular leak syndrome | absent | - | symptomatic, but<br>not requiring<br>fluid support | respiratory<br>compromise or<br>requiring fluids | life-threatening;<br>requiring pressor<br>support and/or<br>ventilatory<br>support |
| Cardiac-<br>ischemia/infarction | none | non-specific T-<br>wave flattening<br>or changes | asymptomatic,<br>ST- and T- wave<br>changes<br>suggesting<br>ischemia | angina without<br>evidence of<br>infarction | acute myocardial infarction |
| Grade | | | | | | | |
|---|---|---|---|---|---|--|--|
| Toxicity | 0 | 1 | 2 | 3 | 4 | | |
| Cardiac left<br>ventricular function | normal | asymptomatic decline of resting ejection fraction of ≥ 10% but < 20% of baseline value; shortening fraction ≥ 24% but < 30% | asymptomatic but resting ejection fraction below LLN for laboratory or decline of resting ejection fraction ≥ 20% of baseline value; < 24% shortening fraction | CHF responsive to treatment | severe or<br>refractory CHF or<br>requiring<br>intubation | | |
| CNS cerebrovascular | ischemia is grade | ed in the NEUROLO | | | | | |
| Cardiac troponin I (cTnI) | normal | - | - | levels consistent<br>with unstable<br>angina as defined<br>by the<br>manufacturer | levels consistent<br>with myocardial<br>infarction as<br>defined by the<br>manufacturer | | |
| Cardiac troponin T (cTnT) | normal | $\geq 0.03 - < 0.05$ | $\geq 0.05 - < 0.1$ | $\geq 0.1 - < 0.2$ ng/ml | $\geq 0.2 \text{ ng/ml}$ | | |
| Edema | none | ng/ml asymptomatic, not requiring therapy | ng/ml<br>symptomatic,<br>requiring therapy | symptomatic<br>edema limiting<br>function and<br>unresponsive to<br>therapy or<br>requiring drug<br>discontinuation | anasarca (severe<br>generalized<br>edema) | | |
| Hypertension | none | asymptomatic,<br>transient increase<br>by >20 mmHg<br>(diastolic) or to ><br>150/100* if<br>previously WNL;<br>not requiring<br>treatment | recurrent or persistent or symptomatic increase by > 20 mmHg (diastolic) or to > 150/100* if previously WNL; not requiring treatment | requiring therapy<br>or more intensive<br>therapy than<br>previously | hypertensive<br>crisis | | |
| *Note: For pediatric | patients, use age | and sex appropriate | normal values > 95t | h percentile ULN. | | | |
| Hypotension | none | changes, but not<br>requiring therapy<br>(including<br>transient<br>orthostatic<br>hypotension) | requiring brief<br>fluid replacement<br>or other therapy<br>but not<br>hospitalization;<br>no physiologic<br>consequences | requiring therapy<br>and sustained<br>medical attention,<br>but resolves<br>without persisting<br>physiologic<br>consequences | shock (associated<br>with acidemia<br>and impairing<br>vital organ<br>function due to<br>tissue<br>hypoperfusion) | | |
| For pediatric patients | I is graded as Car<br>s, systolic BP 65 i | | its up to 1 year old a | | | | |
| than 1 year of age, us<br>Myocarditis | none | or inree measuremen<br>- | - | CHF responsive to treatment | severe or refractory CHF | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Operative injury of vein/artery | none | primary suture<br>repair for injury,<br>but not requiring<br>transfusion | primary suture<br>repair for injury,<br>requiring<br>transfusion | vascular<br>occlusion<br>requiring surgery<br>or bypass for<br>injury | myocardial<br>infarction;<br>resection of orga<br>(e.g., bowel,<br>limb) |
| Pericardial effusion/<br>pericarditis | none | asymptomatic<br>effusion, not<br>requiring<br>treatment | pericarditis (rub,<br>ECG changes,<br>and/or chest pain) | physiologic<br>consequences<br>resulting from<br>symptoms | tamponade<br>(drainage or<br>pericardial<br>window required |
| Peripheral arterial ischemia | none | - | brief episode of ischemia managed non-surgically and without permanent deficit | requiring surgical intervention | life-threatening of<br>with permanent<br>functional deficit<br>(e.g., amputation |
| Phlebitis | none | - | present | - | - |
| Thrombosis/emb Syncope (fainting) is a | olism is grade | ded in the DERMATOI<br>ad in the CARDIOVASONEUROLOGY category | CULAR (GENERAL<br>7. | ) category. | |
| Thrombosis/embolis m | none | - | deep vein<br>thrombosis, not<br>requiring<br>anticoagulant | deep vein<br>thrombosis,<br>requiring<br>anticoagulant<br>therapy | embolic event<br>including<br>pulmonary<br>embolism |
| Vein/artery operative category. | injury is grade | ed as Operative injury of | f vein/artery in the CA | ARDIOVASCULAR | (GENERAL) |
| Visceral arterial ischemia (non-myocardial) | none | - | brief episode of ischemia managed non-surgically and without permanent deficit | requiring surgical intervention | life-threatening of<br>with permanent<br>functional deficit<br>(e.g., resection of<br>ileum) |
| Cardiovascular/<br>General-Other<br>(Specify, | none | mild | moderate | severe | life-threatening of disabling |
| | | | JLATION | | |
| | | egory for grading the sev | verity of bleeding eve | | 1.1 |
| DIC<br>(disseminated<br>intravascular<br>coagulation)<br>Also grade Platelets.<br>Note: Must have incre | absent | -<br>lit products or D-dimer | in order to grade as F | laboratory findings present with no bleeding | laboratory<br>findings <u>and</u><br>bleeding |
| Fibrinogen | WNL | ≥0.75 - <1.0 x<br>LLN | ≥0.5 - <0.75 x | ≥0.25 - <0.5 x | <0.25 x LLN |
| Note: The following c protocol so specifies. | riteria may be | LLN<br>used for leukemia studi | LLN ies or bone marrow ir | LLN<br>nfiltrative/myelophth | isic process if the |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| For leukemia studies: | WNL | <20% decrease<br>from pretreatment<br>value or LLN | ≥20 - <40%<br>decrease from<br>pretreatment<br>value or LLN | ≥40 - <70%<br>decrease from<br>pretreatment<br>value or LLN | <50 mg% |
| Partial thromboplastin time (PTT) | WNL | > ULN - ≤ 1.5 x<br>ULN | $> 1.5 - \le 2 x$ ULN | >2 x ULN | - |
| Phelbitis is graded in the | he CARDIOVAS | SCULAR (GENERA | L) category. | | |
| Prothrombin time (PT) | WNL | $>$ ULN - $\le 1.5 \text{ x}$ ULN | $> 1.5 - \le 2 x$<br>ULN | >2 x ULN | - |
| Thrombosis/embolism | | CARDIOVASCULA | R (GENERAL) cate | | |
| Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura/TTP or hemolytic uremic syndrome/HUS) | absent | | | laboratory<br>findings present<br>without clinical<br>consequences | laboratory findings and clinical consequences, (e.g., CNS hemorrhage/ bleeding or thrombosis/ embolism or renal failure) requiring therapeutic intervention |
| For BMT: | - | evidence of RBC<br>destruction<br>(schistocytosis)<br>without clinical<br>consequences | evidence of RBC destruction with elevated creatinine (≤3 x ULN) | evidence of RBC<br>destruction with<br>creatinine (>3 x<br>ULN) not<br>requiring dialysis | evidence of RBC<br>destruction with<br>renal failure<br>requiring dialysis<br>and/or<br>encephalopathy |
| Also consider Hemogle<br>Note: Must have micro | | | (e.g. schistocytes h | elmet cells-red cell f | raoments) |
| Coagulation-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | CONSTITUTIONAL SYMPTOMS | | | | |
| Fatigue<br>(lethargy, malaise,<br>asthenia) | none | increased fatigue<br>over baseline, but<br>not altering<br>normal activities | moderate (e.g., decrease in performance status by 1 ECOG level or 20% Karnofsky or <i>Lansky</i> ) or causing difficulty performing some activities | severe (e.g., decrease in performance status by ≥2 ECOG levels or 40% Karnofsky or <i>Lansky</i> ) or loss of ability to perform some activities | bedridden or<br>disabling |
| Note: See Appendix IV | / (http://ctep.info | .nih.gov/ctc3/ctc.htm | n) for performance st | tatus scales. | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Fever (in the absence | none | 38.0 - 39.0°C | 39.1 - 40.0°C | > 40.0°C | > 40.0°C |
| of neutropenia, | | (100.4 - 102.2°F) | (102.3 - 104.0°F | $(>104.0^{\circ}F)$ for $<$ | $(>104.0^{\circ}F)$ for $>$ |
| where neutropenia is | | , | ) | 24hrs | 24hrs |
| defined as AGC < | | | | | |
| $1.0 \times 10^9/L$ ) | | | | | |
| Also consider Allergic | | | | | |
| Note: The temperature | | | | | |
| Hot flashes/flushes are | graded in the El | | | | |
| Rigors, chills | none | mild, requiring | severe and/or | not responsive to | - |
| | | symptomatic | prolonged, | narcotic | |
| | | treatment (e.g., | requiring narcotic | medication | |
| | | blanket) or non- | medication | | |
| | | narcotic | | | |
| G 4: | 1 | medication | <u> </u> | | |
| Sweating | normal | mild and | frequent or | - | - |
| (diaphoresis) Weight gain | < 5% | occasional 5 - <10% | drenching<br>10 - <20% | ≥ 20% | |
| Also consider Ascites, | | | 10 - \2070 | ≥ 20% | - |
| Weight gain - veno- | Eucina, i icurai | CITUSIOII. | | | |
| occlusive disease | | | | | |
| (VOD) | | | | | |
| Note: The following c | riteria is to be us | ed ONLY for weight | gain associated with | Veno-Occlusive Dis | sease |
| | <2% | ≥2 - <5% | ≥5 <b>-</b> <10% | ≥10% or as | ≥10% or fluid |
| | | | | ascities | retention |
| | | | | | resulting in |
| | | | | | pulmonary failure |
| Weight loss | < 5% | 5 - <10% | 10 - < 20% | ≥20% | - |
| Also consider Vomitin | ng, Dehydration, | | | | |
| Constitutional | none | mild | moderate | severe | life-threatening or |
| Symptoms-Other | | | | | disabling |
| (Specify, | | | | | |
| ) | | | | | |
| DERMATOLOGY/SKIN | | | | | |
| Alopecia | normal | mild hair loss | pronounced hair | - | - |
| | | | loss | | |
| Bruising | none | localized or in | generalized | - | - |
| (in absence of grade | | dependent area | | | |
| 3 or 4 | | | | | |
| thrombocytopenia) | | | | | |
| | | 3 or 4 thrombocytope | | | |
| Hemorrhage/bleeding | | thrombocytopenia i | n the HEMORRHAO | JE category, <u>not</u> in the | he |
| DERMATOLOGY/SI | LIN category. | | | | |

| hema or a des hy moist ≥1. diant | vere or quiring IV (and seed on full bornatitis) | skin necrosis or ulceration of full thickness dermis; may include spontaneous bleeding not induced by minor trauma or abrasion life-threatening (e.g., exfoliative or ulcerating dermatitis or requiring enteral |
|---|---|---|
| hema or a des hy moist ≥1. diant | vere or quiring IV (oneralized rash painful to matter) | ulceration of full thickness dermis; may include spontaneous bleeding not induced by minor trauma or abrasion life-threatening (e.g., exfoliative or ulcerating dermatitis or |
| tered, but not severalized requirements requirements | quiring IV ( uids (e.g., orneralized rash painful ornatitis) | (e.g., exfoliative or ulcerating dermatitis or |
| eralized required requirements of the requirem | quiring IV ( uids (e.g., orneralized rash painful ornatitis) | (e.g., exfoliative or ulcerating dermatitis or |
| | 5 | or parenteral<br>nutritional<br>support) |
| - | | - |
| , not pair | in changes with in, interfering ith function | |
| nec<br>nummation or sev<br>bitis pro | ceration or cerosis that is vere or olonged, or quiring surgery | |
| ial or -<br>plete loss of<br>(s) or pain in<br>beds | _ | |
| des | | - |
| eralized -<br>nentation<br>nges | | |
| | idespread and<br>oorly controlled | |
| | plete loss of s) or pain in oeds ful erythema er de eralized - nentation ages ase or in espread, wi ved po ataneously or de | ful erythema erythema with desquamation eralized - enentation ages intense or widespread and ved energy controlled |

| dry desquamation patchy moist desquamation, mostly confined to skin folds and creases; moderate edema Note: Pain associated with radiation dermatitis is graded separately in the PAIN category as Pain due to radiation. Radiation recall none faint erythema or a desquamation, following chemotherapy in the absence of additional radiation therapy that occurs in a previous radiation port) Rash/desquamation none macular or papular eruption or erythema with without associated symptoms symptoms For BMT: none macular or papular eruption or erythema crethens follow surface area Torreation (reaction of dry desquamation) absorbed of additional radiation therapy that occurs in a previous readiation port) Rash/desquamation none macular or papular eruption or erythema with without associated symptoms For BMT: none macular or papular eruption or erythema crethens of body surface area Bracklar or papular eruption or erythema with or eryt | Grade | | | | | |
|---|---|---|---|---|---|---|
| Radiation dermatitis none dry desquamation dry desquamation and desquamation, mostly confined to skin folds; pitting edema Note: Pain associated with radiation dermatitis is graded separately in the PAIN category as Pain due to radiation. Radiation recall none faint erythema or reaction (reaction (reaction following chemotherapy in the absence of additional radiation therapy that occurs in a previous radiation port) Rash/desquamation none Rash/desquamation port) Rash/desquamation none Rash/desquamation none Rash/desquamation or or erythema or papular eruption or or erythema or or ther lesions covering <50% of body surface area without associated For BMT: None macular or papular eruption or erythema or or erythema or papular eruption or erythema or or erythema or or erythema or or erythema or papular eruption or or erythema or or there lesions covering <50% of body surface area without associated sociated area without associated area without associated area without associated or erythema or papular eruption or erythema or or erythema or or erythema or or erythema or or erythema or or erythema or or erythema or abrasion or other lesions covering <50% of body surface area without associated area without associated or evaluation or overing ≈25% of body surface area without associated or evaluation or vesicular in associated area without associated or evaluation or erythema or explema or explanation or erythema or or erythema or abrasion or other lesions covering <50% of body surface area without associated or evaluation or erythema or explanation or erythema or abrasion or other lesions covering <50% of body surface area without associated or evaluation or erythema or explanation or erythema or explanation or ex | Toxicity | 0 | 1 | 2 | 3 | 4 |
| Radiation recall reaction (reaction following chemotherapy in the absence of additional radiation port) Rash/desquamation port Rash/desquamation po | Radiation dermatitis | | dry desquamation | erythema or a<br>patchy moist<br>desquamation,<br>mostly confined<br>to skin folds and<br>creases; moderate<br>edema | desquamation,<br>≥1.5 cm<br>diameter, not<br>confined to skin<br>folds; pitting<br>edema | bleeding not<br>induced by minor<br>trauma or<br>abrasion |
| reaction (reaction following chemotherapy in the absence of additional radiation therapy that occurs in a previous radiation port) Rash/desquamation Rash/ | | | | | | |
| papular eruption or erythema without associated symptoms For BMT: none papular eruption or erythema without associated symptoms papular eruption or erythema with pruritis or other associated symptoms symptoms symptoms covering <50% of body surface or localized desquamation or other lesions covering <50% of body surface area For BMT: none macular or papular eruption or erythema covering <25% of body surface area macular or papular eruption or erythema covering <25% of body surface area without associated some associated accovering ≥25 - eruption, with papular eruption or erythema or eruption or erythema or erythema or erythroderma or ulcerative dermatitis or ulcerative dermatitis or other or vesicular exploration or erythema or vesicular eruption or erythema or vesicular eruption, with | reaction (reaction<br>following<br>chemotherapy in the<br>absence of additional<br>radiation therapy that<br>occurs in a previous<br>radiation port) | | dry desquamation | erythema or a<br>patchy moist<br>desquamation,<br>mostly confined<br>to skin folds and<br>creases; moderate<br>edema | desquamation,<br>≥1.5 cm<br>diameter, not<br>confined to skin<br>folds; pitting<br>edema | ulceration of full<br>thickness dermis;<br>may include<br>bleeding not<br>induced by minor<br>trauma or<br>abrasion |
| papular eruption papular eruption generalized exfoliative or erythema or erythema with erythroderma or dermatitis or covering <25% pruritis or other symptomatic ulcerative of body surface associated macular, papular dermatitis or area without symptoms or vesicular bullous formation associated covering ≥25 - eruption, with | Rash/desquamation | none | papular eruption<br>or erythema<br>without<br>associated | papular eruption or erythema with pruritis or other associated symptoms covering <50% of body surface or localized desquamation or other lesions covering <50% of body surface | generalized<br>erythroderma or<br>macular, papular<br>or vesicular<br>eruption or<br>desquamation<br>covering ≥50% of | exfoliative<br>dermatitis or<br>ulcerative |
| surface or formation, or localized desquamation desquamation or covering ≥50% of other lesions body surface area covering ≥25 - <50% of body surface area | For BMT: | none | papular eruption<br>or erythema<br>covering <25%<br>of body surface<br>area without<br>associated | papular eruption or erythema with pruritis or other associated symptoms covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body | generalized<br>erythroderma or<br>symptomatic<br>macular, papular<br>or vesicular<br>eruption, with<br>bullous<br>formation, or<br>desquamation<br>covering ≥50% of | exfoliative<br>dermatitis or<br>ulcerative |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Urticaria<br>(hives, welts,<br>wheals) | none | requiring no<br>medication | requiring PO or<br>topical treatment<br>or IV medication<br>or steroids for<br><24 hours | requiring IV medication or steroids for ≥24 hours | - |
| Wound- infectious | none | cellulitis | superficial infection | infection<br>requiring IV<br>antibiotics | necrotizing<br>fascitis |
| Wound- non-<br>infectious | none | incisional<br>separation | incisional hernia | fascial disruption without evisceration | fascial disruption with evisceration |
| Dermatology/Skin-<br>Other<br>(Specify, ) | none | mild | moderate | severe | life-threatening or disabling |
| | | ENDO | CRINE | | |
| Cushingoid appearance (e.g., moon face with or without buffalo hump, centripetal obesity, cutaneous striae) Also consider Hypergl | absent | - | present | - | - |
| Feminization of male | absent | - | - | present | - |
| Gynecomastia | none | mild | pronounced or painful | pronounced or<br>painful and<br>requiring surgery | - |
| Hot flashes/flushes | none | mild or no more<br>than 1 per day | moderate and<br>greater than 1 per<br>day | - | - |
| Hypothyroidism | absent | asymptomatic,TS<br>H elevated, no<br>therapy given | symptomatic or<br>thyroid<br>replacement<br>treatment given | patient<br>hospitalized for<br>manifestations of<br>hypothyroidism | myxedema coma |
| Masculinization of female | absent | - | - | present | - |
| SIADH (syndrome<br>of inappropriate<br>antidiuretic<br>hormone) | absent | - | - | present | - |
| Endocrine-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | GASTROIN | NTESTINAL | | |
| Amylase is graded in t | he METABOI | LIC/LABORATORY c | | | |
| Anorexia | none | loss of appetite | oral intake<br>significantly<br>decreased | requiring IV<br>fluids | requiring feeding<br>tube or parenteral<br>nutrition |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Ascites (non-malignant) | none | asymptomatic | symptomatic,<br>requiring<br>diuretics | symptomatic,<br>requiring<br>therapeutic<br>paracentesis | life-threatening<br>physiologic<br>consequences |
| Colitis | none | - | abdominal pain<br>with mucus<br>and/or blood in<br>stool | abdominal pain,<br>fever, change in<br>bowel habits with<br>ileus or peritoneal<br>signs, and<br>radiographic or<br>biopsy<br>documentation | perforation or<br>requiring surgery<br>or toxic<br>megacolon |
| | | g with grade 3 or 4 throm ding, Rectal bleeding/her | | | out grade 3 or 4 |
| Constipation | none | requiring stool<br>softener or<br>dietary<br>modification | requiring laxatives | obstipation<br>requiring manual<br>evacuation or<br>enema | obstruction or toxic megacolon |
| Dehydration | none | dry mucous<br>membranes<br>and/or<br>diminished skin<br>turgor | requiring IV fluid replacement (brief) | requiring IV fluid<br>replacement<br>(sustained) | physiologic<br>consequences<br>requiring<br>intensive care;<br>hemodynamic<br>collapse |
| | | ea, Vomiting, Stomatitis/ | | | |
| Diarrhea Patients without colostomy: | none | increase of < 4<br>stools/day over<br>pre-treatment | increase of 4-6<br>stools/day, or<br>nocturnal stools | increase of ≥7<br>stools/day or<br>incontinence; or<br>need for<br>parenteral<br>support for<br>dehydration | physiologic<br>consequences<br>requiring<br>intensive care; or<br>hemodynamic<br>collapse |
| Patients with a colostomy: | none | mild increase in<br>loose, watery<br>colostomy output<br>compared with<br>pretreatment | moderate increase<br>in loose, watery<br>colostomy output<br>compared with<br>pretreatment, but<br>not interfering<br>with normal<br>activity | severe increase in<br>loose, watery<br>colostomy output<br>compared with<br>pretreatment,<br>interfering with<br>normal activity | physiologic<br>consequences,<br>requiring<br>intensive care; or<br>hemodynamic<br>collapse |
| For BMT | none | >500 - <1000ml<br>of diarrhea/day | >1000 - ≤1500ml<br>of diarrhea/day | >1500ml of diarrhea/day | severe abdominal<br>pain with or<br>without ileus |
| For Pediatric BMT: | 1 // 1 | >5 - 10 ml/kg of diarrhea/day | >10 - 15 ml/kg<br>of diarrhea/day | >15 ml/kg of<br>diarrhea/day | - |
| Also consider Hemor<br>thrombocytopenia, Pa | | g with grade 3 or 4 throm on, Hypotension. | nbocytopenia, Hemoi | rnage/bleeding with | out grade 3 or 4 |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Duodenal ulcer<br>(requires<br>radiographic or<br>endoscopic<br>documentation) | none | - | requiring medical<br>management or<br>non-surgical<br>treatment | uncontrolled by outpatient medical management; requiring hospitalization | perforation or<br>bleeding,<br>requiring<br>emergency<br>surgery |
| Dyspepsia/heartburn | none | mild | moderate | severe | - |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If toxicity is rad pharyngeal related to response to the control of the contr | adiation. | | | | |
| Dysphagia- esophageal related to radiation Also consider Pain due | | | dysphagia, requiring predominantly liquid, pureed or soft diet | dysphagia<br>requiring feeding<br>tube, IV<br>hydration or<br>hyperalimentatio<br>n | complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation |
| Note: Fistula is graded | | | 1 1 . | 1 1 . | 1 . |
| Dysphagia - pharyngeal related to radiation | none | mild dysphagia,<br>but can eat<br>regular diet | dysphagia,<br>requiring<br>predominantly<br>pureed, soft, or<br>liquid diet | dysphagia,<br>requiring feeding<br>tube, IV<br>hydration or<br>hyperalimentatio<br>n | complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation |
| Also consider Pain due<br>Note: Fistula is graded | | | ion. | | |
| Fistula- esophageal | none | - | - | present | requiring surgery |
| Fistula- intestinal | none | | | present | requiring surgery |
| Fistula- pharyngeal | none | - | - | present | requiring surgery |
| Fistula- rectal/anal | none | - | - | present | requiring surgery |
| Flatulence | none | mild | moderate | - | - |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1_ | 2 | 3 | 4 |
| Gastric ulcer<br>(requires<br>radiographic or<br>endoscopic<br>documentation) | none | - | requiring medical<br>management or<br>non-surgical<br>treatment | bleeding without<br>perforation,<br>uncontrolled by<br>outpatient<br>medical<br>management;<br>requiring<br>hospitalization or | perforation or<br>bleeding,<br>requiring<br>emergency<br>surgery |
| | rhage/bleeding | g with grade 3 or 4 thron | mbocytopenia, Hemor | surgery<br>rhage/bleeding with | out grade 3 or 4 |
| thrombocytopenia. Gastritis | none | | requiring medical | uncontrolled by | life-threatening |
| Gasurus | none | | management or<br>non-surgical<br>treatment | out-patient medical management; requiring hospitalization or surgery | bleeding,<br>requiring<br>emergency<br>surgery |
| thrombocytopenia. | | g with grade 3 or 4 thron | nbocytopenia, Hemor | | out grade 3 or 4 |
| | | ORRHAGE category. | | | |
| | | MORRHAGE category a | | | |
| Ileus (or neuroconstipation) | none | - | intermittent, not requiring intervention | requiring non-<br>surgical<br>intervention | requiring surger |
| Mouth dryness | normal | mild | moderate | - | - |
| Esophagitis, Gastritis<br>RENAL/GENITOUR<br>Radiation-related mu | , Stomatitis/phanners<br>AINARY categositis is grade | ed as Mucositis due to ra | eal mucositis), and Tyndiation. | phlitis; or the | · |
| Mucositis due to radiation | none | erythema of the<br>mucosa | patchy<br>pseudomembrano<br>us reaction<br>(patches<br>generally ≤ 1.5<br>cm in diameter<br>and non-<br>contiguous) | confluent<br>pseudomembrano<br>us reaction<br>(contiguous<br>patches generally<br>> 1.5 cm in<br>diameter) | necrosis or deep<br>ulceration; may<br>include bleeding<br>not induced by<br>minor trauma or<br>abrasion |
| Dysphagia related to | on mucositis or<br>radiation is als | of the larynx here.<br>So graded as <u>either</u> Dyspending on the site of tre | hagia- esophageal rel | ated to radiation <u>or</u> I | Dysphagia- |
| Nausea | none | able to eat | oral intake<br>significantly<br>decreased | no significant intake, requiring IV fluids | - |
| Pancreatitis | none | - | - | abdominal pain<br>with pancreatic<br>enzyme elevation | complicated by shock (acute circulatory |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Note: Asymptomatic amylase and Amylase are graded in the METABOLIC/LABORATORY category. | | | | | |
| Pharyngitis is graded in the GASTROINTESTINAL category as Stomatitis/pharyngitis (oral/pharyngeal mucositis). | | | | | |
| Proctitis | none | increased stool<br>frequency,<br>occasional blood-<br>streaked stools, or<br>rectal discomfort<br>(including<br>hemorrhoids), not<br>requiring<br>medication | increased stool<br>frequency,<br>bleeding, mucus<br>discharge, or<br>rectal discomfort<br>requiring<br>medication; anal<br>fissure | increased stool<br>frequency/diarrhe<br>a, requiring<br>parenteral<br>support; rectal<br>bleeding,<br>requiring<br>transfusion; or<br>persistent mucus<br>discharge,<br>necessitating<br>pads | perforation,<br>bleeding or<br>necrosis or other<br>life-threatening<br>complication<br>requiring surgical<br>intervention (e.g.,<br>colostomy) |
| thrombocytopenia, and<br>Note: Fistula is grad<br>Proctitis occurring mo<br>Morbidity Scoring Sch | Also consider Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia, and Pain due to radiation. Note: Fistula is graded separately as Fistula- rectal/anal. Proctitis occurring more than 90 days after the start of radiation therapy is graded in the RTOG/EORTC Late Radiation Morbidity Scoring Scheme. (See Appendix V, http://ctep.info.nih.gov/ctc3/ctc.htm) | | | | |
| Salivary gland | none | slightly thickened | thick, ropy, sticky | - | acute salivary |
| changes | | saliva/may have<br>slightly altered<br>taste (e.g.,<br>metallic);<br>additional fluids<br>may be required | saliva; markedly<br>altered taste;<br>alteration in diet<br>required | | gland necrosis |
| Sense of smell | normal | slightly altered | markedly altered | - | - |
| Stomatitis/pharyngiti<br>s (oral/pharyngeal<br>mucositis) | none | painless ulcers,<br>erythema, or mild<br>soreness in the<br>absence of<br>lesions | painful erythema,<br>edema, or ulcers,<br>but can eat or<br>swallow | painful erythema,<br>edema, or ulcers<br>requiring IV<br>hydration | severe ulceration<br>or requires<br>parenteral or<br>enteral nutritional<br>support or<br>prophylatic<br>intubation |
| For BMT: | none | painless ulcers,<br>erythema, or mild<br>soreness in the<br>absence of<br>lesions | painful erythema,<br>edema or ulcers<br>but can swallow | painful erythema,<br>edema, or ulcers<br>preventing<br>swallowing or<br>requiring<br>hydration or<br>parenteral (or<br>enteral)<br>nutritional<br>support | severe ulceration<br>requiring<br>prophylactic<br>intubation or<br>resulting in<br>documented<br>aspiration<br>pneumonia |
| Note: Radiation-relate | d mucositis is gra | ded as Mucositis due | e to radiation. | , , | |
| Taste disturbance (dysgeusia) | normal | slightly altered | markedly altered | - | _ |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Typhlitis (inflammation of the cecum) | none | - | - | abdominal pain,<br>diarrhea, fever, or<br>radiographic<br>documentation | perforation,<br>bleeding or<br>necrosis or other<br>life-threatening<br>complication<br>requiring surgical<br>intervention (e.g.,<br>colostomy) |
| Also consider Hemorri<br>thrombocytopenia, Hy | | | nbocytopenia, Hemor | rhage/bleeding with | out grade 3 or 4 |
| Vomiting | none | 1 episode in 24<br>hours over<br>pretreatment | 2-5 episodes in<br>24 hours over<br>pretreatment | ≥6 episodes in 24 hours over pretreatment; or need for IV fluids | Requiring parenteral nutrition; or physiologic consequences requiring intensive care; hemodynamic collapse |
| Also consider Dehydra Weight gain is graded | | HITIONIAI CVMDT | OMS antagory | | |
| Weight loss is graded | | | | | |
| Gastrointestinal-<br>Other<br>(Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | НЕМОБ | RRHAGE | | |

Note: Transfusion in this section refers to pRBC infusion.

For <u>any</u> bleeding with grade 3 or 4 platelets (< 50,000), <u>always</u> grade Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia. Also consider platelets, transfusion-pRBCS, and transfusion-platelets in addition to the grade that incorporates the site or type of bleeding.

If the site or type of hemorrhage/bleeding is listed, also use the grading that incorporates the site of bleeding: CNS hemorrhage/bleeding, Hematuria, Hematemesis, Hemoptysis, Hemorrhage/bleeding with surgery, Melena/lower GI bleeding, Petechiae/purpura (Hemorrhage/bleeding into skin), Rectal bleeding/hematochezia, Vaginal bleeding. If the platelet count is  $\geq 50,000$  and the site or type of bleeding is listed, grade the specific site. If the site or type is not listed and the platelet count is  $\geq 50,000$ , grade Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia and specify the site or type in the OTHER category.

| Hemorrhage/ble | none | mild without | requiring | catastrophic |
|----------------|------|--------------|-------------|--------------|
| eding with | | transfusion | transfusion | bleeding, |
| grade 3 or 4 | | | | requiring |
| thrombocytopen | | | | major non- |
| ia | | | | elective |
| | | | | intervention |

Also consider Platelets, Hemoglobin, Transfusion-platelet, Transfusion-pRBCs.

Note: This toxicity must be graded for any bleeding with grade 3 or 4 thrombocytopenia. Also grade the site or type of hemorrhage/bleeding. If the site is not listed, grade as Other in the HEMORRHAGE category.

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 1 | 2 | 3 | 4 | |
| Hemorrhage/ble eding without grade 3 or 4 thrombocytopen ia Also consider Platelets, Note: Bleeding in th | e absence of grade 3 | or 4 thrombocytope | sfusion-pRBCs.<br>enia is graded here or<br>ategory. Also grade a | | |
| CNS<br>hemorrhage/ble<br>eding | none | - | - | bleeding<br>noted on CT<br>or other scan<br>with no<br>clinical<br>consequence<br>s | hemorrhagic<br>stroke or<br>hemorrhagic<br>vascular<br>event<br>(CVA) with<br>neurologic<br>signs and<br>symptoms |
| Epistaxis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hematemesis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hematuria<br>(in the absence<br>of vaginal<br>bleeding) | none | microscopic<br>only | intermittent<br>gross<br>bleeding, no<br>clots | persistent gross bleeding or clots; may require catheterizati on or instrumentat ion, or transfusion | open surgery<br>or necrosis<br>or deep<br>bladder<br>ulceration |
| Hemoptysis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |

| | | | de | | |
|---|---|---|---|---|---|
| Гoxicity | 0 1 | - | 2 | 3 | 4 |
| Hemorrhage/ble eding associated with surgery | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophi<br>bleeding,<br>requiring<br>major non-<br>elective<br>interventio |
| Note: Expected blo Melena/GI | none none | e of surgery is not grant mild without | raded as a toxicity. | requiring | catastrophi |
| bleeding | none | transfusion | - | transfusion | bleeding,<br>requiring<br>major non-<br>elective<br>interventio |
| Petechiae/purpu<br>ra<br>(hemorrhage/bl<br>eeding into skin<br>or mucosa) | none | rare<br>petechiae of<br>skin | petechiae or<br>purpura in<br>dependent<br>areas of skin | generalized petechiae or purpura of skin or petechiae of any mucosal site | - |
| Rectal bleeding/<br>hematochezia | none | mild without<br>transfusion<br>or<br>medication | persistent, requiring medication (e.g., steroid suppositorie s) and/or break from radiation treatment | requiring<br>transfusion | catastrophi<br>bleeding,<br>requiring<br>major non-<br>elective<br>interventio |
| Vaginal<br>bleeding | none | spotting,<br>requiring <<br>2 pads per<br>day | requiring ≥ 2 pads per day, but not requiring transfusion | requiring<br>transfusion | catastrophi<br>bleeding,<br>requiring<br>major non-<br>elective<br>interventio |
| Hemorrhage-<br>Other<br>(Specify site, | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophi<br>bleeding,<br>requiring<br>major non-<br>elective<br>interventio |
| | | НЕРА | TIC | | |
| Alkaline<br>phosphatase | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5.0 x<br>ULN | > 5.0 - 20.0<br>x ULN | > 20.0 x<br>ULN |
| Bilirubin | WNL | > ULN - 1.5<br>x ULN | > 1.5 - 3.0 x<br>ULN | > 3.0 - 10.0<br>x ULN | > 10.0 x<br>ULN |
| Bilirubin- graft ver | | | 1 | 1 . 1. | |
| Note: The following | ig criteria are used<br>normal | only for bilirubin a $\geq 2 - \leq 3$ | ssociated with graf<br>≥3 - <6 | It versus host disease. $\ge 6 - < 15$ | ≥15 mg/10 |

| | | Grad | le | | |
|---|---|---|---|---|---|
| Toxicity | 0 1 | 1 2 | 2 | 3 | 4 |
| GGT | WNL | > ULN - 2.5 | > 2.5 - 5.0 x | > 5.0 - 20.0 | > 20.0 x |
| (γ - Glutamyl | | x ULN | ULN | x ULN | ULN |
| transpeptidase) | | | | | |
| Hepatic | absent | - | - | present | - |
| enlargement | atia anlargament an | ly for changes related | d to VOD or other tr | contract related toxic | aitr |
| Hypoalbumine | WNL | LLN - 3 | $\geq 2 - \langle 3 \text{ g/dl} \rangle$ | <2 g/dl | city. |
| mia | WILL | g/dl | 22 - \3 g/ui | <2 g/u1 | - |
| Liver | normal | - | - | asterixis | encephalopa |
| dysfunction/fail | | | | | thy or coma |
| ure (clinical) | | | | | , |
| | ed viral hepatitis is | graded in the INFEC | TION category. | | |
| Portal vein flow | normal | - | decreased | reversal/retr | - |
| | | | portal vein | ograde | |
| | | | flow | portal vein | |
| CCOT (ACT) | WAII | S LILNE OF | > 2.5. 5.0 | flow | > 20.0 |
| SGOT (AST)<br>(serum glutamic | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5.0 x<br>ULN | > 5.0 - 20.0<br>x ULN | > 20.0 x<br>ULN |
| oxaloacetic | | X ULIN | ULIN | X ULIN | ULIN |
| transaminase) | | | | | |
| SGPT (ALT) | WNL | > ULN - 2.5 | > 2.5 - 5.0 x | > 5.0 - 20.0 | > 20.0 x |
| (serum glutamic | W112 | x ULN | ULN | x ULN | ULN |
| pyruvic | | | | | |
| transaminase) | | | | | |
| Hepatic-Other | none | mild | moderate | severe | life- |
| (Specify, | | | | | threatening |
| ) | | | | | or disabling |
| | INF | ECTION/FEBRIL | E NEUTROPENIA | | |
| Catheter-related | none | mild, no | moderate, | severe, | life- |
| infection | | active | localized | systemic | threatening |
| | | treatment | infection, | infection, | sepsis (e.g., |
| | | | requiring<br>local or oral | requiring IV<br>antibiotic or | septic |
| | | | treatment | antifungal | shock) |
| | | | ucaunem | treatment or | |
| | | | | hospitalizati | |
| | | | | on | |
| Febrile | none | - | - | Present | Life- |
| neutropenia | | | | | threatening |
| (fever of | | | | | sepsis (e.g., |
| unknown origin | | | | | septic |
| without | | | | | shock) |
| clinically or | | | | | |
| microbiological | | | | | |
| ly documented infection) | | | | | |
| (ANC < 1.0 x) | | | | | |
| $10^9/L$ , fever | | | | | |
| ≥38.5°C) | | | | | |
| | nia instead of fever i | may be associated wi | th neutropenia and is | s graded here. | |

| | | Grad | le | | |
|---|---|---|---|---|---|
| Гохісіту | 0 | 1 2 | 2 3 | 3 | |
| Infection (documented clinically or microbiological ly) with grade 3 or 4 neutropenia (ANC < 1.0 x | none | - | - | present | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| | | may be associated with i | | | sence of |
| | | e 3 or 4 neutropenia, grad | le as Febrile neutrope | | 1: 0 |
| Infection with unknown ANC | none | - | - | present | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| | ty criterion is u | sed in the rare case when | | | |
| Infection<br>without<br>neutropenia | none | mild, no<br>active<br>treatment | moderate,<br>localized<br>infection,<br>requiring<br>local or oral<br>treatment | severe, systemic infection, requiring IV antibiotic or antifungal treatment, or hospitalizati on | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| Infection/Febril e Neutropenia- Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| Wound-infectious | s is graded in th | ne DERMATOLOGY/SK | IN category. | | |
| | | LYMPHA | ATICS | | |
| Lymphatics | normal | mild<br>lymphedema | moderate<br>lymphedema<br>requiring<br>compression<br>; lymphocyst | severe lymphedema limiting function; lymphocyst requiring surgery | severe lymphedema limiting function with ulceration |
| Lymphatics-<br>Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | METABOLIC/LA | BORATORY | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Acidosis<br>(metabolic or<br>respiratory) | normal | pH < normal, but ≥7.3 | - | pH < 7.3 | pH < 7.3<br>with life-<br>threatening<br>physiologic<br>consequence<br>s |
| Alkalosis<br>(metabolic or<br>respiratory) | normal | pH ><br>normal, but<br>≤7.5 | - | pH > 7.5 | pH > 7.5<br>with life-<br>threatening<br>physiologic<br>consequence<br>s |
| Amylase | WNL | > ULN - 1.5<br>x ULN | > 1.5 - 2.0 x<br>ULN | > 2.0 - 5.0 x<br>ULN | >5.0 x ULN |
| Bicarbonate | WNL | < LLN - 16<br>mEq/dl | 11 - 15<br>mEq/dl | 8 - 10<br>mEq/dl | < 8 mEq/dl |
| CPK<br>(creatine<br>phosphokinase) | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5 x<br>ULN | > 5 - 10 x<br>ULN | > 10 x ULN |
| Hypercalcemia | WNL | > ULN -<br>11.5 mg/dl<br>> ULN - 2.9<br>mmol/L | >11.5 - 12.5<br>mg/dl<br>> 2.9 - 3.1<br>mmol/L | >12.5 - 13.5<br>mg/dl<br>> 3.1 - 3.4<br>mmol/L | > 13.5 mg/dl<br>> 3.4<br>mmol/L |
| Hypercholester<br>olemia | WNL | > ULN -<br>300 mg/dl<br>> ULN -<br>7.75<br>mmol/L | > 300 - 400<br>mg/dl<br>> 7.75 -<br>10.34<br>mmol/L | > 400 - 500<br>mg/dl<br>>10.34 -<br>12.92<br>mmol/L | > 500 mg/dl<br>> 12.92<br>mmol/L |
| Hyperglycemia | WNL | > ULN -<br>160 mg/dl<br>> ULN - 8.9<br>mmol/L | > 160 - 250<br>mg/dl<br>> 8.9 - 13.9<br>mmol/L | > 250 - 500<br>mg/dl<br>> 13.9 -<br>27.8<br>mmol/L | > 500 mg/dl<br>> 27.8<br>mmol/L or<br>ketoacidosis |
| Hyperkalemia | WNL | > ULN - 5.5<br>mmol/L | > 5.5 - 6.0<br>mmol/L | > 6.0 - 7.0<br>mmol/L | > 7.0<br>mmol/L |
| Hypermagnese<br>mia | WNL | > ULN - 3.0<br>mg/dl<br>> ULN -<br>1.23<br>mmol/L | - | > 3.0 - 8.0<br>mg/dl<br>> 1.23 -<br>3.30<br>mmol/L | > 8.0 mg/dl<br>> 3.30<br>mmol/L |
| Hypernatremia | WNL | > ULN -<br>150 mmol/L | >150 - 155<br>mmol/L | >155 - 160<br>mmol/L | >160<br>mmol/L |
| Hypertriglyceri<br>demia | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5.0 x<br>ULN | > 5.0 - 10 x<br>ULN | > 10 x ULN |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hyperuricemia | WNL | > ULN - \le 10 mg/dl \le 0.59 mmol/L without physiologic consequence | - | > ULN - < 10 mg/dl < 0.59 mmol/L with physiologic consequence | > 10 mg/dl<br>> 0.59<br>mmol/L |
| Also consider Ti | ımor İvsis syndroi | s<br>me, Renal failure, Cr | eatinine Potassium | S | |
| Hypocalcemia | WNL | <lln -="" 8.0<br="">mg/dl<br/><lln -="" 2.0<br="">mmol/L</lln></lln> | 7.0 - < 8.0<br>mg/dl<br>1.75 - < 2.0<br>mmol/L | 6.0 - < 7.0<br>mg/dl<br>1.5 - < 1.75<br>mmol/L | <6.0 mg/dl<br>< 1.5<br>mmol/L |
| Hypoglycemia | WNL | <lln -="" 55<br="">mg/dl<br/><lln -="" 3.0<br="">mmol/L</lln></lln> | 40 - < 55<br>mg/dl<br>2.2 - < 3.0<br>mmol/L | 30 - < 40<br>mg/dl<br>1.7 - < 2.2<br>mmol/L | < 30 mg/dl<br>< 1.7<br>mmol/L |
| Hypokalemia | WNL | <lln -="" 3.0<br="">mmol/L</lln> | - | 2.5 - <3.0<br>mmol/L | <2.5<br>mmol/L |
| Hypomagnesem<br>ia | WNL | <lln -="" 1.2<br="">mg/dl<br/><lln -="" 0.5<br="">mmol/L</lln></lln> | 0.9 - <1.2<br>mg/dl<br>0.4 - < 0.5<br>mmol/L | 0.7 - < 0.9<br>mg/dl<br>0.3 - < 0.4<br>mmol/L | < 0.7 mg/dl<br>< 0.3<br>mmol/L |
| Hyponatremia | WNL | <lln -="" 130<br="">mmol/L</lln> | -<br>- | 120 - <130<br>mmol/L | <120<br>mmol/L |
| Hypophosphate<br>mia | WNL | <lln -2.5<br="">mg/dl<br/><lln -="" 0.8<br="">mmol/L</lln></lln> | $\geq 2.0 - < 2.5$<br>mg/dl<br>$\geq 0.6 - < 0.8$<br>mmol/L | ≥1.0 - <2.0<br>mg/dl<br>≥0.3 - <0.6<br>mmol/L | < 1.0 mg/dl<br><0.3<br>mmol/L |
| Hypothyroidism | is graded in the E | ENDOCRINE categor | | | |
| Lipase | WNL | > ULN - 1.5<br>x ULN | > 1.5 - 2.0 x<br>ULN | > 2.0 - 5.0 x<br>ULN | > 5.0 x ULN |
| Metabolic/Labo<br>ratory-Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | MUSCULO | SKELETAL | | |
| | ded in the PAIN c | ategory. | | | |
| Arthritis | none | mild pain with<br>inflammation,<br>erythema or joint<br>swelling but not<br>interfering with<br>function | moderate pain with inflammation, erythema, or joint swelling interfering with function, but not interfering with activities of daily living | severe pain with<br>inflammation,<br>erythema, or joint<br>swelling and<br>interfering with<br>activities of daily<br>living | disabling |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Muscle weakness<br>(not due to<br>neuropathy) | normal | asymptomatic<br>with weakness on<br>physical exam | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | bedridden or<br>disabling |
| Myalgia is graded in the | | | | | |
| Myositis<br>(inflammation/dama<br>ge of muscle) | none | mild pain, not interfering with function | pain interfering<br>with function, but<br>not interfering<br>with activities of<br>daily living | pain interfering<br>with function and<br>interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| Also consider CPK. | | - (;1 | | | |
| Note: Myositis implies Osteonecrosis (avascular necrosis) | s muscle damag<br>none | asymptomatic<br>and detected by<br>imaging only | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | symptomatic; or disabling |
| Musculoskeletal-<br>Other<br>(Specify, | none | mild | moderate | severe | life-threatening or<br>disabling |
| , | | NEURO | OLOGY | | |
| Aphasia, receptive and | /or expressive, | is graded under Speec | h impairment in the | NEUROLOGY cates | gory. |
| Arachnoiditis/menin gismus/radiculitis | absent | mild pain not interfering with function | moderate pain<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain<br>interfering with<br>activities of daily<br>living | unable to<br>function or<br>perform activities<br>of daily living;<br>bedridden;<br>paraplegia |
| Also consider Headach | | | | 1 | 1 1 1.1 1 |
| Ataxia (incoordination) | normal | asymptomatic but<br>abnormal on<br>physical exam,<br>and not<br>interfering with<br>function | mild symptoms<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | moderate<br>symptoms<br>interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| CNS cerebrovascular ischemia | none | <u>-</u> | - | transient<br>ischemic event or<br>attack (TIA) | permanent event<br>(e.g., cerebral<br>vascular<br>accident) |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Cognitive<br>disturbance/<br>learning problems | none | cognitive disability; not interfering with work/school performance; preservation of intelligence | cognitive disability; interfering with work/school performance; decline of 1 SD (Standard Deviation) or loss of developmental milestones | cognitive disability; resulting in significant impairment of work/school performance; cognitive decline > 2 SD | inability to<br>work/frank<br>mental<br>retardation |
| Confusion | normal | confusion or<br>disorientation or<br>attention deficit<br>of brief duration;<br>resolves<br>spontaneously<br>with no sequelae | confusion or<br>disorientation or<br>attention deficit<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | confusion or<br>delirium<br>interfering with<br>activities of daily<br>living | harmful to others<br>or self; requiring<br>hospitalization |
| Cranial neuropathy is | | EUROLOGY categor | y as Neuropathy-crar | nial. | |
| Delusions | normal | - | - | present | toxic psychosis |
| Depressed level of consciousness | normal | somnolence or<br>sedation not<br>interfering with<br>function | somnolence or<br>sedation<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | obtundation or<br>stupor; difficult<br>to arouse;<br>interfering with<br>activities of daily<br>living | coma |
| Note: Syncope (faintir | ng) is graded in t | he NEUROLOGY ca | itegory. | | |
| Dizziness/lightheade dness | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| Dysphasia, receptive a | nd/or expressive | e, is graded under Spe | | ne NEUROLOGY ca | tegory. |
| Extrapyramidal/<br>involuntary<br>movement/<br>restlessness | none | mild involuntary<br>movements not<br>interfering with<br>function | moderate involuntary movements interfering with function, but not interfering with activities of daily living | severe<br>involuntary<br>movements or<br>torticollis<br>interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| | normal | | - | present | toxic psychosis |
| Hallucinations | поннач | - | <del>-</del> | DIESEIII | 101210 11500 1101212 |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Insomnia Note: This toxicity is g | normal graded when inso | occasional difficulty sleeping not interfering with function mnia is related to tree | difficulty sleeping interfering with function, but not interfering with activities of daily living atment. If pain or oth | frequent difficulty sleeping, interfering with activities of daily living er symptoms interfer | re with sleep do |
| NOT grade as insomni | | | | | |
| Irrit ability (children <3 years of age) | normal | mild; easily<br>consolable | moderate;<br>requiring<br>increased<br>attention | severe;<br>inconsolable | - |
| Leukoencephalopath<br>y associated<br>radiological findings | none | mild increase in SAS (subarachnoid space) and/or mild ventriculomegaly; and/or small (+/- multiple) focal T2 hyperintensities, involving periventricular white matter or < 1/3 of susceptible areas of cerebrum | moderate increase in SAS; and/or moderate ventriculomegaly ; and/or focal T2 hyperintensities extending into centrum ovale; or involving 1/3 to 2/3 of susceptible areas of cerebrum | severe increase in SAS; severe ventriculomegaly; near total white matter T2 hyperintensities or diffuse low attenuation (CT); focal white matter necrosis (cystic) | severe increase in SAS; severe ventriculomegaly; diffuse low attenuation with calcification (CT); diffuse white matter necrosis (MRI) |
| Memory loss | normal | memory loss not interfering with function | memory loss<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | memory loss<br>interfering with<br>activities of daily<br>living | amnesia |
| Mood alteration-<br>anxiety agitation | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | suicidal ideation<br>or danger to self |
| Mood alteration-<br>depression | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | suicidal ideation<br>or danger to self |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Mood alteration-<br>euphoria | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | danger to self |
| Neuropathic pain is gr | | N category. | | | life threatening |
| Neuropathy- cranial | absent | - | present, not<br>interfering with<br>activities of daily<br>living | present,<br>interfering with<br>activities of daily<br>living | life-threatening,<br>disabling |
| Neuropathy- motor | normal | subjective<br>weakness but no<br>objective findings | mild objective<br>weakness<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | objective<br>weakness<br>interfering with<br>activities of daily<br>living | paralysis |
| Neuropathy-sensory | normal | loss of deep<br>tendon reflexes or<br>paresthesia<br>(including<br>tingling) but not<br>interfering with<br>function | objective sensory<br>loss or<br>paresthesia<br>(including<br>tingling),<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | sensory loss or<br>paresthesia<br>interfering with<br>activities of daily<br>living | permanent<br>sensory loss that<br>interferes with<br>function |
| Nystagmus<br>Also consider Vision- | absent<br>double vision. | present | - | - | - |
| Personality/behavior<br>al | normal | change, but not<br>disruptive to<br>patient or family | disruptive to patient or family | disruptive to<br>patient and<br>family; requiring<br>mental health<br>intervention | harmful to others<br>or self; requiring<br>hospitalization |
| Pyramidal tract<br>dysfunction (e.g., ↑<br>tone, hyperreflexia,<br>positive Babinski, ↓<br>fine motor<br>coordination) | normal | asymptomatic<br>with abnormality<br>on physical<br>examination | symptomatic or<br>interfering with<br>function but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden or<br>disabling;<br>paralysis |
| Seizure(s) | none | - | seizure(s) self-<br>limited and<br>consciousness is<br>preserved | seizure(s) in<br>which<br>consciousness is<br>altered | seizures of any<br>type which are<br>prolonged,<br>repetitive, or<br>difficult to<br>control (e.g.,<br>status epilepticus,<br>intractable<br>epilepsy) |

| | | Gı | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Speech impairment<br>(e.g., dysphasia or<br>aphasia) | normal | - | awareness of<br>receptive or<br>expressive<br>dysphasia, not<br>impairing ability<br>to communicate | receptive or<br>expressive<br>dysphasia,<br>impairing ability<br>to communicate | inability to communicate |
| Syncope (fainting) | absent | - | - | present | -<br>1 · |
| Also consider CARD | none | mild and brief or intermittent but not interfering with function | moderate tremor interfering with function, but not interfering with activities of daily living | severe tremor<br>interfering with<br>activities of daily<br>living | - |
| Vertigo | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| Neurology-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | OCULAI | R/VISUAL | | |
| Cataract | none | asymptomatic | symptomatic,<br>partial visual loss | symptomatic, visual loss requiring treatment or interfering with function | - |
| Conjunctivitis | none | abnormal ophthalmologic changes, but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Dry eye | normal | mild, not<br>requiring<br>treatment | moderate or requiring artificial tears | - | - |
| Glaucoma | none | increase in<br>intraocular<br>pressure but no<br>visual loss | increase in intraocular pressure with retinal changes | visual<br>impairment | unilateral or<br>bilateral loss of<br>vision (blindness) |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Keratitis<br>(corneal<br>inflammation/<br>corneal ulceration) | none | abnormal ophthalmologic changes but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | unilateral or<br>bilateral loss of<br>vision (blindness) |
| Tearing (watery eyes) | none | mild: not<br>interfering with<br>function | moderate:<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | - |
| Vision- blurred vision | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- double<br>vision (diplopia) | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- flashing<br>lights/floaters | normal | mild, not<br>interfering with<br>function | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- night<br>blindness<br>(nyctalopia) | normal | abnormal electro-<br>retinography but<br>asymptomatic | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and<br>interfering with<br>activities of daily<br>living | - |
| Vision- photophobia | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Ocular/Visual-Other (Specify, | normal | mild | moderate | severe | unilateral or<br>bilateral loss of<br>vision (blindness) |

| | | G | rade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Abdominal pain or cramping | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Arthralgia<br>(joint pain) | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Arthritis (joint pain w | ith clinical sig | ns of inflammation) is g | graded in the MUSCU | JLOSKELETAL cat | egory. |
| Bone pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Chest pain<br>(non-cardiac and<br>non-pleuritic) | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Dysmenorrhea | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Dyspareunia | none | mild pain not interfering with function | moderate pain interfering with sexual activity | severe pain<br>preventing sexual<br>activity | - |
| | he RENAL/GI | ENITOURINARY cate | | | |
| Earache (otalgia) | none | mild pain not interfering with function | moderate pain:<br>pain or analgesics<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |

| | | G | rade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Headache | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Hepatic pain | none | mild pain not interfering with function | moderate pain:<br>pain or analgesics<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Myalgia<br>(muscle pain) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Neuropathic pain<br>(e.g., jaw pain,<br>neurologic pain,<br>phantom limb pain,<br>post-infectious<br>neuralgia, or painful<br>neuropathies) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pain due to radiation | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pelvic pain | none | mild pain not interfering with function | moderate pain:<br>pain or analgesics<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pleuritic pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Rectal or perirectal pain (proctalgia) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Tumor pain (onset or exacerbation of tumor pain due to treatment) Tumor flair is graded | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pain-Other | none | mild | moderate | severe | disabling |
| (Specify, | попс | mid | moderate | Severe | uisaoiiiig |
| | | PULM | ONARY | | |
| Adult Respiratory<br>Distress Syndrome<br>(ARDS) | absent | - | - | - | present |
| Apnea | none | - | - | present | requiring intubation |
| Carbon monoxide diffusion capacity (DL <sub>CO</sub> ) | ≥ 90% of pretreatment or normal value | ≥75 - <90% of pretreatment or normal value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of pretreatment or normal value | < 25% of<br>pretreatment or<br>normal value |
| Cough | absent | mild, relieved by<br>non-prescription<br>medication | requiring narcotic antitussive | severe cough or<br>coughing spasms,<br>poorly controlled<br>or unresponsive<br>to treatment | - |
| Dyspnea (shortness of breath) | normal | - | dyspnea on exertion | dyspnea at<br>normal level of<br>activity | dyspnea at rest or<br>requiring<br>ventilator support |
| FEV <sub>1</sub> | ≥ 90% of pretreatment or normal value | ≥75 - <90% of pretreatment or normal value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of pretreatment or normal value | < 25% of<br>pretreatment or<br>normal value |
| Hiccoughs (hiccups, singultus) | none | mild, not<br>requiring<br>treatment | moderate,<br>requiring<br>treatment | severe,<br>prolonged, and<br>refractory to<br>treatment | - |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hypoxia | normal | - | decreased O <sub>2</sub> saturation with exercise | decreased O <sub>2</sub> saturation at rest, requiring supplemental oxygen | decreased O <sub>2</sub> saturation, requiring pressure support (CPAP) or assisted ventilation |
| Pleural effusion<br>(non-malignant) | none | asymptomatic<br>and not requiring<br>treatment | symptomatic,<br>requiring<br>diuretics | symptomatic, requiring O <sub>2</sub> or therapeutic | life-threatening<br>(e.g., requiring<br>intubation) |
| Dlauritia nain ia arada | d in the DAIN est | 20071 | | thoracentesis | |
| Pleuritic pain is graded<br>Pneumonitis/pulmon<br>ary infiltrates | none | radiographic changes but asymptomatic or symptoms not requiring steroids | radiographic<br>changes and<br>requiring steroids<br>or diuretics | radiographic<br>changes and<br>requiring oxygen | radiographic<br>changes and<br>requiring assisted<br>ventilation |
| Pneumothorax | none | no intervention | chest tube | sclerosis or | life-threatening |
| | | required | required | surgery required | |
| Pulmonary embolism | | | | | category. |
| Pulmonary fibrosis | none | radiographic<br>changes, but<br>asymptomatic or<br>symptoms not<br>requiring steroids | requiring steroids<br>or diuretics | requiring oxygen | requiring assisted ventilation |
| Note: Radiation-relate | d pulmonary fibro | | RTOG/EORTC Late | Radiation Morbidity | Scoring Scheme- |
| Lung. (See Appendix | | | | | s coming s chieffing |
| Voice changes/stridor/laryn x (e.g., hoarseness, loss of voice, laryngitis) | normal | mild or<br>intermittent<br>hoarseness | persistent<br>hoarseness, but<br>able to vocalize;<br>may have mild to<br>moderate edema | whispered<br>speech, not able<br>to vocalize; may<br>have marked<br>edema | marked<br>dyspnea/stridor<br>requiring<br>tracheostomy or<br>intubation |
| Radiation-related | hemoptysis from TINAL category. | Radiation-related h | raded as Grade 4 Mu | y.<br>acositis due to radiati<br>horacic cavity is grad | |
| Pulmonary-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| , | | RENAL/CENI | ITOURINARY | | |
| Bladder spasms | absent | mild symptoms,<br>not requiring<br>intervention | symptoms<br>requiring<br>antispasmotic | severe symptoms<br>requiring narcotic | - |
| Creatinine Note: Adjust to age-ap | WNL | > ULN - 1.5 x<br>ULN | > 1.5 - 3.0 x<br>ULN | > 3.0 - 6.0 x<br>ULN | > 6.0 x ULN |
| Dysuria | none | mild symptoms | symptoms | symptoms not | |
| (painful urination) | 110110 | requiring no intervention | relieved with<br>therapy | relieved despite<br>therapy | |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Fistula or GU fistula<br>(e.g., vaginal,<br>vesicovaginal) | none | - | - | requiring intervention | requiring surgery |
| Hemoglobinuria | - | present | - | - | - |
| Hematuria (in the abse | ence of vaginal b | | the HEMORRHAGI | | |
| Incontinence | none | with coughing, sneezing, etc. | spontaneous,<br>some control | no control (in the absence of fistula) | - |
| Operative injury to bladder and/or ureter | none | - | injury of bladder<br>with primary<br>repair | sepsis, fistula, or<br>obstruction<br>requiring<br>secondary<br>surgery; loss of<br>one kidney;<br>injury requiring<br>anastomosis or<br>re-implantation | septic obstruction<br>of both kidneys<br>or vesicovaginal<br>fistula requiring<br>diversion |
| Proteinuria | normal or < 0.15 g/24 hours | 1+ or 0.15 - 1.0<br>g/24 hours | 2+ to 3+ or 1.0 -<br>3.5 g/24 hours | 4+ or > 3.5 g/24 hours | nephrotic<br>syndrome |
| Note: If there is an inc | | een absolute value an | d uristix reading, use | e the absolute value for | or grading. |
| Renal failure | none | - | - | requiring dialysis,<br>but reversible | requiring dialysis and irreversible |
| Ureteral obstruction | none | unilateral, not requiring surgery | - | bilateral, not<br>requiring surgery | stent,<br>nephrostomy<br>tube, or surgery |
| Urinary electrolyte<br>wasting (e.g.,<br>Fanconi's syndrome,<br>renal tubular<br>acidosis)<br>Also consider Acidosi | none | asymptomatic,<br>not requiring<br>treatment | mild, reversible<br>and manageable<br>with oral<br>replacement | reversible but<br>requiring IV<br>replacement | irreversible,<br>requiring<br>continued<br>replacement |
| Urinary | normal | increase in | increase > 2 x | hourly or more | |
| frequency/urgency | поппа | frequency or<br>nocturia up to 2 x<br>normal | normal but < hourly | with urgency, or requiring catheter | - |
| Urinary retention | normal | hesitancy or<br>dribbling, but no<br>significant<br>residual urine;<br>retention<br>occurring during<br>the immediate<br>postoperative<br>period | hesitancy requiring medication or occasional in/out catheterization (<4 x per week), or operative bladder atony requiring indwelling catheter beyond immediate postoperative period but for < 6 weeks | requiring frequent in/out catheterization (≥ 4 x per week) or urological intervention (e.g., TURP, suprapubic tube, urethrotomy) | bladder rupture |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Urine color change<br>(not related to other<br>dietary or<br>physiologic cause<br>e.g., bilirubin,<br>concentrated urine,<br>hematuria) | normal | asymptomatic,<br>change in urine<br>color | - | - | - |
| Vaginal bleeding is gra | aded in the HEM | ORRHAGE categor | V. | | |
| Vaginitis<br>(not due to infection) | none | mild, not<br>requiring<br>treatment | moderate,<br>relieved with<br>treatment | severe, not<br>relieved with<br>treatment, or<br>ulceration not<br>requiring surgery | ulceration<br>requiring surgery |
| Renal/Genitourinary-<br>Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | SECONDARY | MALIGNANCY | | |
| Secondary Malignancy-Other (Specify type,) excludes metastastic tumors | none | - | - | - | present |
| | <b>C</b> 1 | EVITAT /DEPDANI | UCTIVE FUNCTIO | N | |
| Dyspareunia is graded | | | JCIIVE FUNCTIO | 71 | |
| Dysmenorrhea is grade | ed in the PAIN ca | ategory. | | | |
| Erectile impotence | normal | mild (erections<br>impaired but<br>satisfactory) | moderate<br>(erections<br>impaired,<br>unsatisfactory for<br>intercourse) | no erections | - |
| Female sterility | normal | - | - | sterile | - |
| Femininization of male | | | | | |
| Irregular menses<br>(change from<br>baseline) | normal | occasionally irregular or lengthened interval, but continuing menstrual cycles | very irregular, but<br>continuing<br>menstrual cycles | persistent<br>amenorrhea | - |
| Libido | normal | decrease in interest | severe loss of interest | - | - |
| Male infertility | - | - | Oligospermia<br>(low sperm<br>count) | Azoospermia<br>(no sperm) | - |
| Masculinization of fen | nale is graded in | the ENDOCRINE ca | tegory. | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Vaginal dryness | normal | mild | requiring | - | - |
| | | | treatment and/or | | |
| | | | interfering with | | |
| | | | sexual function, | | |
| C 1/D 1 .: | | '1 1 | dyspareunia | | 1: 11: |
| Sexual/Reproductive | none | mild | moderate | severe | disabling |
| Function-Other (Specify, | | | | | |
| (specify, | | | | | |
| , | | | | | |
| | | | ded in previous cate | | |
| Acute vascular leak sy | | | | | |
| ARDS (Adult Respira | | | | | |
| Autoimmune reactions | | | | | |
| DIC (disseminated int | | | | | |
| Fanconi's syndrome is | | | | | |
| Renal tubular acidosis Stevens-Johnson synd | | | | | |
| SIADH (syndrome of | | | | | у. |
| Thrombotic microangi | | | | | gymdrom/HIIC) ig |
| graded in the COAGU | | | openie purpura/111 ( | of hemorytic dreinic | syndrom/1103) is |
| Tumor flare | none | mild pain not | moderate pain; | severe pain; pain | Disabling |
| | | interfering with | pain or analgesics | or analgesics | |
| | | function | interfering with | interfering with | |
| | | | function, but not | function and | |
| | | | interfering with | interfering with | |
| | | | activities of daily | activities of daily | |
| A1: 1 II | .1 | | living | living | |
| Also consider Hyperca<br>Note: Tumor flare is | | o constallation of a | mantona and sice sie | direct relation to ini | itiation of the areas |
| | | | mptoms and signs in ). The symptoms/sign | | |
| visible tumor, hy | | | ther electrolyte distu | | n, inframmation of |
| Tumor lysis | absent | - | - | present | - |
| syndrome | | | | | |
| Also consider Hyperka | alemia, Creatinin | e | . 1 1 | 1 1 1 2 | |
| Urinary electrolyte wa RENAL/GENITOUR | | | tubular acidosis) is | graded under the | |
| Syndromes-Other | | | 1 4 . | | 1:0 4 |
| 25 | none | mild | moderate | severe | life-threatening or |
| (Specify, | none | mild | moderate | severe | life-threatening or disabling |

## Appendix II Toxicity Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| Toxicity: | Date of Treatment | : | Course Number: |
|---|---|---|---|
| Date of onset: | | | Grade at onset: |
| Date of first change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Did toxicity resolve? | Yes | No | |
| If so, date of resolution of toxicity: | | | |
| Date of last observation (if prior to | | | |
| recovery): | | | |
| Reason(s) observations stopped (if | | | |
| prior to recovery): | | | |
| Was patient retreated? | Yes | No | |
| If yes, was treatment delayed for | Yes | No | |
| recovery? | | | |
| Date of next treatment? | | | |
| Dose reduced for next treatment? | Yes | No | |
| Additional Comments: | | | |
| If module is being activated for new | toxicity, not currer | ntly in CTC, please | e provide definitions for |
| toxicity grading: | • • | , 1 | |
| Grade 0 = | | | |
| Grade 1 = | | | |
| Grade 2 = | | | |
| Grade 3 = | | | |
| Grade 4 = | | | |

## Appendix III Infection Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| | | • | definitions to grade the following (CHOOSE O | • | ection. |
|---|---|---|---|---|---|
| | BACTERIAL | <b>FUNGAL</b> | PROTOZOAL | VIRAL | UNKNOWN |
| 3. | Specify site of infe<br>BLOOD CULTUR<br>BONE INFECTIO<br>CATHETER (intra<br>CATHETER (intra<br>CENTRAL NERV<br>EAR INFECTION<br>EYE INFECTION<br>GASTROINTEST<br>ORAL INFECTIO<br>PNEUMONIA<br>SKIN INFECTION<br>UPPER RESPIRA<br>URINARY TRAC<br>VAGINAL INFEC | RE POSITIVE N avenous) avenous), tunnel OUS SYSTEM INAL INFECTION TORY INFECT | INFECTION<br>ON | LL THAT APPLY): | |
| | INFECTION, not of | otherwise specifi | ed (Specify site, | ) | |
| 4.<br>5. | Specify organism,<br>Prophylactic antibit<br>Yes<br>If prophylaxis was | if known:<br>lotic, antifungal,<br>No<br>given prior to in | or antiviral therapy adr | ministration below: | |
| | Antifungal prophy | laxis | | | |
| | Other prophylaxis | | | | |

## Appendix IV Performance Status Scales/Scores

| ECOG or Zubrod Scale | | Karnofsky Score |
|---|---|---|
| 0 | Asymptomatic and fully active | 100% |
| 1 | Symptomatic; fully ambulatory; restricted in physically strenuous activity | 80-90% |
| 2 | Symptomatic; ambulatory; capable of self-care; more than 50% of waking hours are spent out of bed | 60-70% |
| 3 | Symptomatic; limited self-care; spends more than 50% of time in bed, but not bedridden | 40-50% |
| 4 | Completely disabled; no self-care; bedridden | 20-30% |

Appendix V
RTOG/EORTC Late Radiation Morbidity Scoring Scheme
Use for toxicities occurring greater than 90 days after radiation therapy.

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Bladder-<br>Late RT Morbidity<br>Scoring | No change<br>from baseline | Slight epithelial<br>atrophy/minor<br>telangiectasia<br>(microscopic<br>hematuria) | Moderate<br>frequency/<br>generalized<br>telangiectasia/<br>intermittent<br>macroscopic<br>hematuria | Severe frequency and dysuria/severe generalized telangiectasia (often with petechiae); frequent hematuria; reduction in bladder capacity (< 150 cc) | Necrosis/contract<br>ed bladder<br>(capacity < 100<br>cc)/severe<br>hemorrhagic<br>cystitis |
| Bone-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic;<br>no growth<br>retardation;<br>reduced bone<br>density | Moderate pain or<br>tenderness;<br>growth<br>retardation;<br>irregular bone<br>sclerosis | Severe pain or<br>tenderness;<br>complete arrest of<br>bone growth;<br>dense bone<br>sclerosis | Necrosis/<br>spontaneous<br>fracture |
| Brain-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild headache;<br>slight lethargy | Moderate<br>headache; great<br>lethargy | Severe<br>headaches; severe<br>CNS dysfunction<br>(partial loss of<br>power or<br>dyskinesia) | Seizures or paralysis; coma |
| Esophagus-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild fibrosis;<br>slight difficulty in<br>swallowing<br>solids; no pain on<br>swallowing | Unable to take<br>solid food<br>normally;<br>swallowing semi-<br>solid food;<br>dilatation may be<br>indicated | Severe fibrosis;<br>able to swallow<br>only liquids; may<br>have pain on<br>swallowing;<br>dilation required | Necrosis/<br>perforation;<br>fistula |
| Heart-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic or<br>mild symptoms;<br>transient T wave<br>inversion and ST<br>changes; sinus<br>tachycardia > 110<br>(at rest) | Moderate angina<br>on effort; mild<br>pericarditis;<br>normal heart size;<br>persistent<br>abnormal T wave<br>and ST changes;<br>low QRS | Severe angina; pericardial effusion; constrictive pericarditis; moderate heart failure; cardiac enlargement; EKG abnormalities | Tamponade/sever<br>e heart<br>failure/severe<br>constrictive<br>pericarditis |
| Joint-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild joint<br>stiffness; slight<br>limitation of<br>movement | Moderate<br>stiffness;<br>intermittent or<br>moderate joint<br>pain; moderate | Severe joint<br>stiffness; pain<br>with severe<br>limitation of<br>movement | Necrosis/complet<br>e fixation |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | | | limitation of movement | | |
| Kidney-<br>Late RT Morbidity<br>Scoring | No change from baseline | Transient albuminuria; no hypertension; mild impairment of renal function; urea 25 - 35 mg%; creatinine 1.5 - 2.0 mg%; creatinine clearance > 75% | Persistent moderate albuminuria (2+); mild hypertension; no related anemia; moderate impairment of renal function; urea > 36 - 60 mg%; creatinine clearance > 50 - 74% | Severe albuminuria; severe hypertension; persistent anemia (< 10 g%); severe renal failure; urea > 60 mg%; creatinine > 4 mg%; creatinine clearance < 50% | Malignant hypertension; uremic coma/urea > 100% |
| Larynx-<br>Late RT Morbidity<br>Scoring | No change from baseline | Hoarseness;<br>slight arytenoid<br>edema | Moderate arytenoid edema; chondritis | Severe edema;<br>severe chondritis | Necrosis |
| Liver-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild lassitude;<br>nausea;<br>dyspepsia;<br>slightly abnormal<br>liver function | Moderate<br>symptoms; some<br>abnormal liver<br>function tests;<br>serum albumin<br>normal | Disabling hepatic insufficiency; liver function tests grossly abnormal; low albumin; edema or ascites | Necrosis/hepatic<br>coma or<br>encephalopathy |
| Lung-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic or<br>mild symptoms<br>(dry cough);<br>slight<br>radiographic<br>appearances | Moderate<br>symptomatic<br>fibrosis or<br>pneumonitis<br>(severe cough);<br>low grade fever;<br>patchy<br>radiographic<br>appearances | Severe<br>symptomatic<br>fibrosis or<br>pneumonitis;<br>dense<br>radiographic<br>changes | Severe<br>respiratory<br>insufficiency/<br>continuous<br>O2/assisted<br>ventilation |
| Mucous membrane-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight atrophy<br>and dryness | Moderate atrophy and telangiectasia; little mucus | Marked atrophy<br>with complete<br>dryness; severe<br>telangiectasia | Ulceration |
| Salivary glands-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight dryness of<br>mouth; good<br>response on<br>stimulation | Moderate dryness<br>of mouth; poor<br>response on<br>stimulation | Complete dryness<br>of mouth; no<br>response on<br>stimulation | Fibrosis |
| Skin-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight atrophy;<br>pigmentation<br>change; some<br>hair loss | Patchy atrophy;<br>moderate<br>telangiectasia;<br>total hair loss | Marked atrophy;<br>gross<br>telangiectasia | Ulceration |
| Small/Large<br>intestine-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild diarrhea;<br>mild cramping;<br>bowel movement<br>5 x daily slight<br>rectal discharge | Moderate diarrhea and colic; bowel movement > 5 x daily; excessive | Obstruction or bleeding, requiring surgery | Necrosis/<br>perforation fistula |
| Grade | | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| Toxicity | 0 | 1 | 2 | 3 | 4 | | | | |
| | | or bleeding | rectal mucus or intermittent bleeding | | | | | | |
| Spinal cord-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild Lhermitte's syndrome | Severe<br>Lhermitte's<br>syndrome | Objective<br>neurological<br>findings at or<br>below cord level<br>treatment | Mono-, para-,<br>quadriplegia | | | | |
| Subcutaneous tissue-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight induration<br>(fibrosis) and loss<br>of subcutaneous<br>fat | Moderate fibrosis<br>but<br>asymptomatic;<br>slight field<br>contracture; <<br>10% linear<br>reduction | Severe induration<br>and loss of<br>subcutaneous<br>tissue; field<br>contracture ><br>10% linear<br>measurement | Necrosis | | | | |
| Eye-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic cataract; minor corneal ulceration or keratitis | Symptomatic cataract; moderate corneal ulceration; minor retinopathy or glaucoma | Severe keratitis;<br>severe<br>retinopathy or<br>detachment;<br>severe glaucoma | Panophthalmitis;<br>blindness | | | | |
| Radiation-Other (Specify, | None | Mild | Moderate | Severe | Life-threatening or disabling | | | | |

## Appendix VI BMT Complex/Multi-Component Events

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | | | Events in bone marrow to | | |
| The grading sc | ale must use the | CTC criteria for | r grading the specific con | nponent events (to | oxicities). |
| Failure to engraft | absent | mild | moderate | severe | life-threatening |
| Also consider Hemo | globin (Hgb), N | Neutrophils/grant | alocytes (ANC/AGC), Pla | atelets | |
| Graft versus host | absent | mild | moderate | severe | life-threatening |
| disease | | | | | - |
| Also consider Fatigu | ue, Rash/desqua | mation, Diarrhea | a, Bilirubin-GVHD | | |
| Stem cell infusion | absent | mild | moderate | severe | life-threatening |
| complications | | | | | |
| | | | hythmia, Hypertension, I | | |
| | | | Nausea, Vomiting, Hemor | | |
| | | | ade 3 or 4 thrombocytope | | |
| | | | emia, Hypernatremia, Hyp | | ssed level of |
| consciousness, Seizi | ures, Abdomina | l pain, Headache | e, Creatinine, Hemoglobir | nuria | |
| Veno-Occlusive | absent | mild | moderate | severe | life-threatening |
| Disease (VOD) | | | | | |
| Also consider Weig | ht gain-VOD, B | ilirubin, Depress | sed level of consciousness | s, Hepatic pain, R | enal failure, Hepatic |
| enlargement. | | | | | |

#### CITY OF HOPE NATIONAL MEDICAL CENTER 06/20/07 1500 EAST DUARTE ROAD **DUARTE, CA 91010**

#### DEPARTMENT OF HEMATOLOGY / BONE MARROW TRANSPLANTATION

A PHASE I/II TRIAL OF ESCALATING DOSE OF YTTRIUM-90-LABELED ANTI-CD20 TITLE: MONOCLONAL ANTIBODY IN COMBINATION WITH HIGH-DOSE ETOPOSIDE AND

CYCLOPHOSPHAMIDE FOLLOWED BY AUTOLOGOUS STEM CELL TRANSPLANTATION FOR

PATIENTS WITH POOR RISK/RELAPSED B-CELL NON-HODGKIN'S LYMPHOMA

IRB# 98153 CITY OF HOPE PROTOCOL NUMBER/VERSION NUMBER: Version 17 **DATE(S) OF AMENDMENT(S)/REVISION(S):** 

10/29/03, 04/06/04, 06/16/04

05/10/00

Amendment 1 - 01/31/00 -Version 01 Amendment 8 – 02/08/01 -Version 08 2 -05/03/01 -Amendment 05/10/00 -Version 02 Amendment 9 – Version 09 Amendment 3 – 06/05/00 -Version 03 Amendment 10 -08/07/01 -Version 10 Amendment 07/13/00 -Version 04 Amendment 11 -05/30/02 -Version 11 09/08/00 -Amendment 5 -Version 05 Amendment 12 – 10/29/03 -Version 12 04/06/04 -Amendment 6 – 10/25/00 -Version 06 Amendment 13 -Version 13 Amendment 7 - 12/20/00 -Version 07 Amendment 14 – 06/16/04 – Version 14 Amendment 15 - 06/20/07 - Version 15 Amendment 16 - 04/18/12 - Version 16

(title page only change)

Amendment 17 - 03/28/14 -- Version 17

SITE: Lymphoma

Low and Intermediate Grade CD20 (+) HISTOLOGY:

II, III, IV STAGE (IF APPLICABLE):

Chemotherapy/Radioimmunotherapy **MODALITY:** 

Phase I/II TYPE:

PRINCIPAL INVESTIGATOR:

Auayporn Nademanee, M.D. Department of Hematology/Hematopoietic Cell Transplantation 06/16/04

**COLLABORATING INVESTIGATOR:** 

Andrew Raubitschek, M.D. Department of Radioimmunotherapy

**PARTICIPATING CLINICIANS:** 

Stephen J. Forman, M.D. Department of Hematology/Hematopoietic Cell Transplantation 06/16/04

Joycelynne Palmer, Ph.D. Department of Biostatistics 10/29/03

> City of Hope National Medical Center **PARTICIPATING INSTITUTIONS:**

INVESTIGATIONAL NEW DRUG (IND) NUMBER: **BB-IND 8836**  05/10/00, 06/05/00, 09/08/00, 10/29/03, 06/16/04

## TABLE OF CONTENTS

| 1.0 | BACKO | GROUND RATIONALE | 1 |
|---|---|---|---|
| 2.0 | OBJEC | TIVES | 8 |
| 3.0 | STUDY | DESIGN | 8 |
| 4.0 | DRUG | FORMULATION | 9 |
| 5.0 | STAGI | NG CRITERIA | 12 |
| 6.0 | ELIGII | BILITY CRITERIA | 13 |
| 7.0 | EXCLU | JSION CRITERIA | 14 |
| 8.0 | TREAT | TMENT PLAN | 14 |
| 9.0 | STUDY | DESIGN AND RULES FOR DOSE ESCALATION | 18 |
| 10.0 | STUDY | CALENDAR - PREPARATIVE REGIMEN AND PBSCT | 21 |
| 11.0 | CRITE | RIA FOR EVALUATION AND ENDPOINT DEFINITIONS | 22 |
| 12.0 | STATIS | STICAL CONSIDERATIONS | 23 |
| 13.0 | REGIS | TRATION GUIDELINES | 24 |
| 14.0 | RECOI | RDS TO BE KEPT AND DATA SUBMISSION SCHEDULE | 24 |
| 15.0 | GENDI | ER AND MINORITIES | 25 |
| 16.0 | DATA 1 | MANAGEMENT | 25 |
| 17.0 | ETHIC | AL AND REGULATORY CONSIDERATIONS | 25 |
| 18.0 | REFER | RENCES | 26 |
| Apper | ndix I | Common Toxicity Criteria (CTC) | <b>A1</b> |
| Apper | ndix II | <b>Toxicity Module</b> | A38 |
| Apper | ndix III | Infection Module | A39 |
| Apper | ndix IV | Performance Status Scales/Scores | A40 |
| Apper | ndix V | RTOG/EORTC Late Radiation Morbidity Scoring Scheme | A41 |
| Apper | ndix VI | BMT Complex/Multi-Component Events | A44 |

#### 1.0 BACKGROUND RATIONALE

Non-Hodgkin's lymphomas (NHLs) are the sixth most common cause of cancer-related deaths in the United States. The incidence of NHL has increased by 50% over the past 15 years. The incidence of both indolent and aggressive lymphomas increases with age, making these the most commonly diagnosed lymphoid malignancies in patients over 60 years old. Despite the use of aggressive combination chemotherapy regimens, approximately 30-40% of patients with intermediate- and high-grade NHL does not achieve complete remission (CR) or suffers relapse after attaining remission.<sup>2</sup> High-dose chemotherapy or chemo/radiotherapy followed by autologous bone marrow or stem cell transplantation (ASCT) has been shown to induce longterm disease control in about 10-50% of patients with relapsed and refractory intermediate- and high-grade lymphoma.<sup>3</sup> Recently, the benefit of high-dose therapy and ASCT proved to be superior to conventional salvage chemotherapy in a randomized Parma study of 215 patients with chemotherapy-sensitive NHL in relapse. The 5-year event-free survival (EFS) was 46% for the ASCT group as compared to 12% for the salvage therapy without transplantation (p = 0.001). Thus, high-dose therapy and ASCT has become a potential curative modality for patients with recurrent aggressive lymphoma. However, not all patients derive long-term benefits from this treatment and recurrent disease remains the single most common cause of treatment failure posthigh-dose therapy and ASCT. Therefore, new therapeutic approaches are needed.

Patients with low-grade NHL have indolent clinical courses and are not cured by current treatment approaches. Although most patients can achieve a complete remission with standard treatment, the median duration of first CR ranges from 12 to 36 months. Relapsed low-grade lymphoma may still respond to salvage therapy. But the duration of subsequent remissions progressively decreases. High-dose therapy and ASCT has been shown to improve survival and to increase the duration of remission in some patients with relapsed low-grade NHL. However, because of the long natural history and the continued pattern of relapse post-ASCT in some studies, the role of high-dose therapy and ASCT as a potential curative treatment for patients with relapsed low-grade lymphoma has not been clearly established.

Recently, the role of radioimmunotherapy for treatment of NHL has emerged. Radioisotope-labeled monoclonal antibodies provide a mechanism by which radioactivity can be directly targeted to tumors sites while sparing normal tissues. B-cell lymphomas are attractive targets for radioimmunotherapy because of their radiosensitivity, their well-defined surface antigens and the availability of multiple monoclonal antibodies to those antigens.

## 1.1 Results of High-Dose Chemo/Radiotherapy and ASCT for NHL

Several high-dose therapy regimens have been used as preparative regimens for NHL. But so far, none of these regimens have emerged as the best regimen. However, since NHL is radiosensitive and based on experience with acute leukemia, the combination of total body irradiation (TBI) and cyclophosphamide (Cy) has been widely used as a preparative regimen for some patients with lymphoid malignancies. In an attempt to reduce relapse rates, etoposide has been added to the TBI and Cy regimen because of its known activity in lymphoma. The results of phase I and II studies of TBI 12.0 Gy, etoposide 60 mg/kg and Cy 100 mg/kg conducted at City of Hope<sup>6</sup>. Stanford University<sup>7</sup> and Fred Hutchinson Cancer Research Center (FHCRC)<sup>8</sup> demonstrate the activity of this regimen in patients with lymphoid malignancies. The transplantrelated mortality within 100 days was 7-8%, with the common causes of death being venoocclusive disease (VOD), diffuse alveolar hemorrhage and infection. The major transplantrelated morbidities were mucositis and skin toxicities, which were fully reversible. The 5-year EFS and overall survival (OS) were 52% [95% Confidence interval (CI) 42-62%] and 61% (95% CI 50-73%), respectively for 134 patients with NHL who underwent ASCT utilizing this regimen at Stanford. These results have been confirmed in the Southwestern Oncology Group cooperative trial. Despite its effectiveness, the relapse rate of 34-53 % remains considerably high. Thus, new preparative regimens need to be explored.

## 1.2 Radionuclides for Radioimmunotherapy

Iodine-131 (<sup>131</sup>I) has been the gold standard for radioimmunotherapy due to its long track record in treating thyroid carcinomas, its well-defined radiochemistry, its clinical availability, and its potential for both radioimmunoscintigraphy and radioimmunotherapy. <sup>131</sup>I has been employed in the majority of reported clinical trials of radioimmunotherapy. However, there are disadvantages to <sup>131</sup>I, including its long 8-day half life, the risks of radiation exposure to health care providers and the non-specific irradiation to normal organs from gamma components of <sup>131</sup>I.

Yttrium-90 (<sup>90</sup>Y) may be an ideal radionuclide for radioimmunotherapy since it emits beta particles that are more potent than those delivered by <sup>131</sup>I. It is a pure beta emitter, making it a safer reagent for medical personnel to administer. In addition, the short half-life of <sup>90</sup>Y facilitates its use in combination with other agents, i.e. chemotherapy or total body radiation, and allows for high dose rates at localized sites. Unfortunately, <sup>90</sup>Y cannot be used for radioimmunoscintigraphy due to its absence of gamma emissions. Indium-111 (<sup>111</sup>In) has been substituted as an imaging reagent to show tumor localization in patients scheduled for <sup>90</sup>Y therapy, based on its biodistribution which is close to that of <sup>90</sup>Y. <sup>111</sup>In-labeled murine monoclonals have been used successfully in clinical imaging trials for cutaneous T-cell lymphoma, chronic lymphocytic leukemia, melanoma, and colon cancer.

### 1.3 Anti-CD 20

Anti-CD20 (anti-B1) is a murine monoclonal antibody of isotype IgG2a, raised against cryopreserved Burkitt's lymphoma cells. The antibody reacts against the B1 antigen, an epitope of the CD20 developmental cell surface protein. CD20 is a 35 kD cell surface phosphoprotein found on 95% of normal mature B-cells and more than 90% of B-cell non-Hodgkin's lymphomas and B-cell chronic lymphocytic leukemias tested, but not on T-cells, plasma cells, uncommitted

hematopoietic-precursors stem cells, dendritic cells, granulocytes, monocytes, or erythrocytes, or on tumors of T cell, myeloid or erythroid origin. CD20 is not shed and does not modulate from the surface after binding of antibody.

Anti-CD20 has been used extensively as a therapeutic agent for use in bone marrow purging. Clinical use of this antibody in marrow purging has shown it to be selective in eradicating B cell lymphomas as well as normal B-cells, while leaving other lymphocyte population intact. Some subpopulation of B cell precursors is left intact, as evidence by engraftment of the normal B cell compartment.

#### 1.4 IDEC-C2B8

IDEC-C2B8 is a chimeric antibody with a murine variable portion and a human IgG1 kappa constant portion that recognizes the CD20 antigens expressed on normal B-cells and most malignant B-cell lymphomas. IDEC-C2B8 shows specificity for the CD 20 antigen and binds with an apparent affinity of 4.3 x 10<sup>-9</sup>M. IDEC-C2B8 has also been reported to induce apoptosis and to sensitize drug-resistant human B-cell lymphoma cell lines to cytotoxic chemotherapy.

A phase I dose escalation pharmacokinetic trial of IDEC-C2B8 given as a single intravenous infusion using doses ranging from 10 mg/m² to 500 mg/m² in patients with relapsed or refractory low-grade lymphoma was reported by Maloney et al. The median half-life of the free antibody at doses ranging from 100 mg/m² to 500 mg/m² was 4.4 days (range 1.6-10.5 days). In phase II clinical studies, anti-tumor activity has been observed in patients with relapsed or refractory low-grade or follicular B-cell NHL. The majority of adverse events was mild to moderate and included fever, fatigue, chills and nausea which were primarily associated with the initial infusions. No quantifiable human anti-mouse antibodies (HAMA) or human anti-chimeric antibodies (HACA) were observed. Depletion of peripheral B-cells occurred rapidly following the first infusion with recovery beginning 6 months post-treatment. Despite this depletion of B-cells, there was minimal change in serum IgG, IgM, and IgA levels and no increase in the frequency or severity of infectious complications. Anti-tumor activity was observed at various disease sites including peripheral blood, bone marrow, lymph nodes, spleen and abdomen.

A phase III trial to assess the safety and efficacy of IDEC-C2B8 375 mg/m² given once weekly for four doses in 166 patients with relapsed or refractory low-grade or follicular NHL was reported by McLaughlin et al. <sup>10</sup> The overall response rate in 151 evaluable patients was 50% (9CR; 67 PR). The median duration of response has not been reached after a median follow-up of 9+ months. Conversion to negative bcl-2 status occurred in 57% of patients who were positive at baseline and subsequently reevaluated after the fourth infusion. No positive HAMA responses were observed in 67 patients evaluated and the incidence of HACA was less than 1%. Severe neutropenia and thrombocytopenia were observed in less than 2% of patients. IDEC-C2B8 has also been studied in 44 patients with relapsed diffuse large B-cell and mantle cell lymphoma. The overall response rate was 31%, with a 10% CR rate. Thus anti-CD20 monoclonal antibody has become a very effective salvage therapy for CD20+ B-cell low-and intermediate-grade NHL and this treatment has become an important addition to our armamentarium.

IDEC-C2B8 has also been studied in combination with chemotherapy. Czuczman et al<sup>11</sup>

conducted a phase II multi-center study evaluating the safety and anti-tumor activity of IDEC-C2B8 375 mg/m² for six doses in combination with six cycles of CHOP (cyclophosphamide, doxorubicin, vincristine and prednisone) chemotherapy in 40 patients with low-grade NHL. Combination therapy appeared safe and toxicity profile observed was consistent with that seen with CHOP alone. No HAMA or HACA responses were observed. The overall response rate in 35 patients who completed treatment was 100% (21 CR; 14 PR). The median time to disease progression has not been reached with follow-up time of 9-27+ months. Seven of eight patients who were bcl-2 positive at baseline by polymerase chain reaction (PCR) became negative in both peripheral blood and bone marrow following treatment. This combined therapy is being investigated in previously untreated patients with intermediate- and high-grade NHL.

## 1.5 Results of Radiolabeled Antibodies in the Treatment of Non-Hodgkin's Lymphoma

Most recent radioimmunotherapy trials for lymphoma have utilized <sup>131</sup>I-labeled anti-B1 (anti-CD20) antibody. Kaminski et al<sup>12</sup> first reported on a trial utilizing multiple treatments with low dose <sup>131</sup>I-labeled anti-B1 antibody in ten patients who had a CD20 positive B-cell lymphoma in whom primary therapy had failed. Six of the nine treated patients had tumor responses, including patients with bulky or chemotherapy-resistant diseases. Four patients had complete remissions (CR), and two had partial responses. The follow-up time was relatively short, but no disease progression was observed in the four patients who achieved a CR at 8-11 months. Toxicity was minimal with mild or no myelosuppression.

Based on these results, a phase I/II study of <sup>131</sup>I-labeled anti-B1 was conducted in 58 heavily pretreated patients with NHL (28 low-grade, 14 transformed low-grade, 15 intermediate-grade, and 2 high-grade). <sup>13</sup> The median number of prior therapy was 4, 88% had stage III or IV disease, 36% had bulky disease, 51% had an elevated LDH level and 14 had failed BMT. Patients received 1-3 dosimetric doses followed by a therapeutic dose. The dosimetric dose involved the IV administration of 5 mCi of <sup>131</sup>I anti-B1 antibody to determine the rate of whole body clearance so that a whole body radiation dose could be calculated. Each dosimetric dose was preceded by 0, 95, or 475 mg of unlabeled antibody. Therapeutic dose escalation was initiated at 25 cGy and adjusted in 10 cGy increment until the MTD. The MTD was 75 cGy for patients who had not undergone BMT. The overall response rate in these heavily pre-treated patients was 71% with a CR rate of 34%. The median duration of response was 271 days (95% CI; 40-394 days) and the median duration of CR was 566 days. Response was observed in both low-grade and transformed low-grade NHL as well as in patients with bulky disease and patients who had relapsed post-BMT.

Further trials of <sup>131</sup>I-labeled anti-B1 antibody at non-myeloablative doses has been studied in 4 separate clinical trials (phase I and II, single and multi-center) in 113 patients with low-grade NHL including 25 with transformed low-grade NHL. <sup>14</sup> Patients received a single dosimetric dose of 450 mg of unlabeled anti-B1 infusion over one hour followed by 35 mg radiolabeled with 5 mCi <sup>131</sup>I over ½ hour. The therapeutic dose was administered 7 to 14 days after the dosimetric dose and consisted of the same unlabeled and labeled antibody doses. The overall response rate was 77% with a CR rate of 45% and 67% of the complete responders were in continuous remission for > 4 years. Reversible hematologic toxicity was the dose-limiting toxicity. ANC < 100/mm<sup>3</sup> was observed in 2.6% of patients and platelets < 10,000/mm<sup>3</sup> in 5.3%. The nadir

typically occurred at week 5-6 with recovery by week 8-9. The most common non-hematologic toxicities were transient mild to moderate fever, nausea, asthenia, and chills. None of the patients developed HAMA. These results suggest that <sup>131</sup>I-labeled anti-B1 is safe and effective and may induce prolonged CR in heavily pre-treated low-grade and transformed low-grade NHL.

## 1.6 Results of <sup>131</sup>I anti-B1 Monoclonal Antibody with Autologous Bone Marrow Support

Although promising results have been reported with radiolabeled MAb for NHL, these results may be improved by using higher dose or myeloablative radiation dose. The use of radiolabeled MAb at myeloablative radiation dose followed by autologous stem cell rescue has been explored by investigators from The Fred Hutchinson Cancer Research Center. Press et al<sup>15</sup> conducted a trial utilizing higher dose of <sup>131</sup>I-labeled anti-CD20 antibody with autologous bone marrow rescue in 43 patients with B-cell lymphoma in relapse. In this study, sequential biodistribution studies were performed with escalating doses of antibody (0.5, 2.5, and 10 mg/kg) trace-labeled with 5 to 10 mCi of <sup>131</sup>I. Patients whose tumors were estimated to receive greater doses of radiation than liver, lungs, or kidneys (a favorable biodistribution) were eligible for the therapeutic infusion of <sup>131</sup>I-labeled antibody. Of the 43 patients, 24 had a favorable biodistribution, and 19 received therapeutic infusion of 234-777 mCi of <sup>131</sup>I-labeled antibodies (58-1168 mg) followed by autologous marrow infusion. Sixteen patients achieved a CR, two had a partial response and one had a minor response. Nine of the complete responders have remained in continuous CR for 3 to 53 months. Toxicities include myelosuppression, nausea, infection and two episodes of cardiopulmonary toxicity. In this study, cardiopulmonary toxicity was the dose limiting, non-hematopoietic toxicity of high-dose <sup>131</sup>I-labeled antibody.

In an attempt to reduce toxicity to normal tissues and to directly deliver higher dose of radiation to tumor sites. <sup>131</sup>I-labeled-anti-CD20 MAb has been incorporated into high-dose therapy regimen instead of TBI. Press et al<sup>16</sup> reported results of a phase I/II study to define the MTD of an <sup>131</sup>Ilabeled anti-B1 monoclonal antibody which can be given with high-dose etoposide and cyclophosphamide in conjunction with ASCT in 38 (26 low-grade; 12 aggressive) NHL patients. Patients were treated in a cohorts of 4 patients each with doses of <sup>131</sup>I-anti-B1 antibody (2.5 mg/kg, 318-840 mCi) calculated to deliver 20-27 Gy of radiation to dose-limiting, critical normal organs, followed by etoposide (0 or 60 mg/kg), cyclophosphamide (100 mg/kg), and ABMT (15 patients) or ASCT (22 patients). Of the 37 evaluable patients, 33 (89%) were currently alive and 29 (78%) were progression-free after a median follow-up of 1.5 yr. Toxicities included grade 4 myelosuppression in all patients, grade 2-3 nausea in 26 (70%), pulmonary infiltrate in 4 and grade 3 VOD in 2 patients. There were four death; 3 from progressive NHL and 1 from disseminated Varicella. These results suggest that <sup>131</sup>I- anti-B1 antibody can be given at doses delivering ≥ 25 Gy to critical normal organs, with pulmonary and gastrointestinal toxicities being dose-limiting. Although additional studies are needed, <sup>131</sup>I-anti-B1 antibody can be safely given in combination with high-dose chemotherapy in an autologous stem cell transplant setting for NHL.

## 1.7 90 Y -Anti-CD20 Radioimmunotherapy for Relapsed NHL

A phase I/II dose escalation study of  $^{90}$ Y-murine anti-CD20 monoclonal antibody (MAb) in patients with recurrent B-cell lymphoma was performed by Knox et al.  $^{17}$  The primary objectives

of the study were: (a) to determine the effect of the preinfusion of unlabeled anti-CD20 MAb on the biodistribution of <sup>111</sup>In-anti-CD20 MAb; (b) to determine the maximal tolerated dose of <sup>90</sup>Y-anti-CD20 MAb that does not require bone marrow transplantation; and (c) to evaluate the safety and antitumor effect of <sup>90</sup>Y-anti-CD20 MAb in patients with recurrent B-cell lymphoma. Eighteen patients with relapsed low- or intermediate-grade non-Hodgkin's lymphoma were treated. Biodistribution studies with <sup>111</sup>In- anti-CD20 MAb were performed prior to therapy. Groups of three or four patients were treated at dose levels of approx 13.5, 20, 30, 40, and 50 mCi <sup>90</sup>Y-anti-CD20 MAb. Three patients were retreated at the 40 mCi dose level. The use of unlabeled antibody affected the biodistribution favorably. Nonhematological toxicity was minimal. The only significant toxicity was myelosuppression. The overall response rate following a single dose of <sup>90</sup>Y-anti-CD20 MAb therapy was 72%, with six complete responses and seven partial responses and freedom from progression of 3-29+ mo following treatment. Radioimmunotherapy with less than or equal to 50 mCi <sup>90</sup>Y-anti-CD20 MAb resulted in minimal nonhematological toxicity and durable clinical responses in patients with recurrent B-cell lymphoma. Doses of less than or equal to 40 mCi <sup>90</sup>Y-anti-CD20 MAb were not myeloablative.

Results of a phase I/II study utilizing chimeric antibody Rituximab as the unlabeled clearing antibody and <sup>90</sup>Y conjugated anti-CD20 (IDEC-Y2B8, conjugated to the parent murine monoclonal 2B8) was recently reported. In the study reported by Witzig et al<sup>18</sup>, the first portion of the study compared 100 mg/m<sup>2</sup> with 250 mg/m<sup>2</sup> of Rituximab as the clearing dose and compared dosimetry imaging capabilities. It was determined that 250 mg/m<sup>2</sup> of Rituximab was the optimal dose to be used. In the second portion of the phase I study, the dose of IDEC-Y2B8 was escalated from 0.2 mCi/kg to 0.4 mCi/kg. No bone marrow or stem cell harvest was required. None of the patients treated at 0.2, 0.3 and 0.4 mCi/kg whose baseline platelet count > 150,000/mm<sup>3</sup> developed grade 4 hematologic toxicity, whereas 3 of 6 patients treated at 0.2 or 0.3 mCi/kg with baseline platelet counts between 100,000 to 150,000/mm<sup>3</sup> developed transient grade 4 hematologic toxicity.

The dosimetry from this phase I/II trial of IDEC-Y2B8 was reported by Wiseman et al. <sup>19</sup> Fortytwo patients with low- and intermediate-grade NHL received IDEC-Y2B8 following injection of unlabeled Rituximab (cold antibodies) followed by 2 mg of mouse anti-CD20 antibody labeled with 5 mCi <sup>111</sup>In (IDEC-In2B8). <sup>90</sup>Y 0.2, 0.3, or 0.4 mCi/kg was given 7 days following <sup>111</sup>I. The patients had <sup>111</sup>In dosimetry performed by serial whole body gamma camera imaging, urine collection and blood sampling at 0, 2, 6, 24, 48, 72, 96 and 144 hours. The highest mean calculated <sup>90</sup>Y radiation dose to a normal organ was spleen with 24.16 rads/mCi (0.6-67.0), followed by liver with 17.2 rad/mCi (9.4-39.2) and lungs with 12.9 rads/mCi (4.2-67.7). <sup>90</sup>Y dose of 0.4 mCi/kg was the MTD for bone marrow toxicity (thrombocytopenia and neutropenia). These results suggest that: 1) no organ irradiated beyond safety levels; 2) <sup>111</sup>I can serve as a predictor of <sup>90</sup>Y; 3) Rituximab dose of 250 mg/m² has been established as the "cold" antibody with added benefits of its therapeutic effect; and 4) bone marrow toxicity was the dose-limiting effect with full and predictable recovery.

Outcomes from this trial have been compiled in a submitted publication. <sup>19</sup> The overall response rate (ORR) for the intent-to-treat population (n = 51) was 67% (26% CR, 41% PR); for the low-grade group (n = 34) 82% (27% CR, 56% PR); 43% for intermediate grade (n = 4); and 0% for mantle cell (n = 3). Responses were seen in patients with bulky (> 7 cm) disease (41%) and

splenomegaly (50%). Kaplan-Meier estimate of time-to-progression in responders and duration of response is 12.9+ months and 11.7+ months, respectively. Adverse events were primarily hematologic and correlated with baseline extent of marrow involvement with NHL and baseline platelet count. Only one patient developed an anti-antibody response (HACA/HAMA).

## 1.8 Study Proposal

The high-dose therapy regimen of FTBI 1200 cGy, etoposide 60 mg/kg and Cy 100 mg/kg has been used extensively at City of Hope as a preparative regimen for patients with hematological malignancies. Given the relatively high relapse rate associated with this regimen, the effective anti-lymphoma therapy of IDEC-C2B8, and the safety and feasibility of IDEC-Y2B8 with the ability to directly deliver radiation to tumors sites, we propose to study a new preparative regimen in patients with relapsed NHL which will utilize <sup>90</sup>Y-labeled anti-CD20 antibody (IDEC-Y2B8) instead of TBI in combination with high-dose etoposide and cyclophosphamide. We plan to conduct a phase I/II trial to define the maximum tolerated dose (MTD) of IDEC-Y2B8 that can be given with high-dose etoposide and cyclophosphamide followed by ASCT, and to define the response rate and toxicities associated with this regimen. To avoid liver toxicity, etoposide dose will be started at 40 mg/kg and escalated to 60 mg/kg and the dose of Cy will be fixed at 100 mg/kg.

05/03/01, 06/16/04

The patient will undergo a dosimetry study with IDEC-In2B8 to confirm favorable localization of isotope one week prior to administration of therapeutic dose IDEC-Y2B8. Serial gamma camera images will be obtained at the end of the infusion, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours post-infusion. At each time point, one whole body and 4 spot planar scans will be acquired with the Toshiba dual head camera. In addition, two SPECT images will be obtained at 48 and 72 -96 hour time points. Nuclear Medicine images will be used to estimate the distribution of activity in various organs, especially liver, lungs, kidney, heart and spleen. Blood samples will be drawn prior to IDEC-C2B8 and at approximately 0 hours (immediately prior to IDEC-In2B8), 2 hours, 4 - 6 hours, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours following antibody infusion. These samples will be used to analyze antibody clearance and bone marrow dose estimates. Urine samples will be collected daily for six days to analyze radioisotope clearance.

05/03/01, 08/07/01,

Favorable biodistribution will be defined as tumor dose greater than any normal organ, except spleen and bone marrow, ie. liver, lung, kidney. For patients in CR at time of transplantation, no specific tumor localization is required as long as Ga 67 scan and/or FDG-PET scan is negative. Tumor dose will be calculated from multiple gamma camera images and blood/urine pharmacokinetics. If the patient shows favorable biodistribution, the therapeutic dose will be administered on day -14. Serial gamma camera images will be obtained at the end of the infusion, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours post-infusion. At each time point, one whole body and 4 spot planar scans will be acquired with the Toshiba dual head camera. Nuclear Medicine images will be used to confirm estimates of the distribution of activity in various organs, especially liver, lungs, kidney, heart and spleen. Blood samples will be drawn prior to IDEC-C2B8 and at approximately 0 hours (immediately prior to IDEC-In2B8 / IDEC-Y2B8), 2 hours, 4 - 6 hours, 24 hours, 48 hours, 72 - 96 hours, 120 hours and 144 hours following antibody infusion. These samples will be used to analyze antibody clearance and bone

marrow dose estimation. Urine samples will be collected daily for six days to analyze radioisotope clearance. The therapeutic dose will be administered to deliver a target dose of 1000 cGy to the organ projected to receive the highest dose from the imaging study. After the first two dose levels the dose will be increased in increments of 250 cGy until a maximum of 2500 cGy is attained or dose limiting toxicity is encountered.

#### 2.0 OBJECTIVES

05/10/00

10/29/03

- 2.1 To evaluate the safety and efficacy of a new preparative regimen of <sup>90</sup>Y-labeled anti-CD20 MAb (IDEC-Y2B8) in combination with high-dose etoposide and cyclophosphamide followed by ASCT for treatment of patients with relapsed/refractory and poor risk NHL.
- 2.2 To determine the MTD of <sup>90</sup>Y-anti-CD20 MAb which can be given with high-dose etoposide 60 mg/kg and high-dose cyclophosphamide 100 mg/kg followed by ASCT in patients with NHL.
- 2.3 To perform dosimetry study to estimate the radiation dose delivered to the tumor and normal organs.
- 2.4 To evaluate the short-term and long-term complication of this new preparative regimen.

#### 3.0 STUDY DESIGN

This is an open-label phase I-II clinical and efficacy study of a new preparative regimen followed by autologous stem cell support in patients with relapsed and refractory NHL. Patients with low-, and intermediate-grade NHL who have relapsed followed conventional chemotherapy or have failed to achieve remission, and who are candidates for high-dose therapy and ASCT will be eligible for this study. All patients will receive IDEC-Y2B8 in combination with high-dose etoposide and cyclophosphamide followed by ASCT. The dose of Cy will be fixed at 100 mg/kg. There will be two doses escalating schema for etoposide and IDEC-Y2B8. Etoposide will be started at 40 mg/kg (cohort 1) and escalate to 60 mg/kg (cohort 2). The dose of Y2B8 will be the same for cohort 1 and 2, to deliver 1000 cGy to the normal organ receiving the greatest accumulation. If no dose limiting toxicity is observed, while the etoposide dose remains at 60 mg/kg, the dose of Y2B8 will be escalated to 1250 cGy, and then to a maximum of 2500 cGy, or until the MTD has been reached. Therefore, there will be cohorts with 3 patients per cohort as follows (an additional 2 patients per cohort will be accrued if there are eligible patients available prior to the determination of toxicity on the current dose level):

Cohort 1: Y2B8 to deliver 1000 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 40 mg/kg

cyclophosphamide 100 mg/kg

Cohort 2: Y2B8 to deliver 1000 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 3: Y2B8 to deliver 1250 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 4: Y2B8 to deliver 1500 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 5: Y2B8 to deliver 1750 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

Cohort 6 to 8: Y2B8 to deliver 2000-2500 cGy to highest normal

organ excluding spleen and bone marrow

etoposide 60 mg/kg

cyclophosphamide 100 mg/kg

All patients will have peripheral blood stem cell collected with the target CD34+ of  $3.0 \times 10^6$ /kg. Patients will undergo dosimetry studies on day -21 and therapy on day -14. Etoposide will be given on day -4, followed by a day rest and cyclophosphamide on day -2. PBSC will be infused on day +1 when the radiation dose to the reinfused stem cells is estimated to be < 5 cGy.

### 4.0 DRUG FORMULATION

#### 4.1 IDEC-Y2B8

a. Drug Formulation and Procurement

IDEC-2B8-MX-DTPA Two ml glass septum vial containing 2 ml (3.2 mg) IDEC-2B8-MX-DTPA in low metal normal saline at 1.6 mg/ml.

RITUXAN (IDEC-C2B8) Ten ml (100 mg) and/or 50 ml (500 mg) pharmaceutical grade glass vials at a concentration of 10 mg of protein per ml.

<sup>111</sup>In-chloride 5 mCi of Indium-111 chloride supplied in .05M HCl. 40-100 mCi Yttrium-90 chloride supplied in .05M HCl.

#### b. Drug Toxicity

Myelosuppression is the dose limiting toxicity in non marrow supported regimens. With marrow support liver, kidney, and lung are likely to be the dose limiting organs for toxicity. Infusional toxicity of chills and rigors are common with the first administration but rarely with subsequent doses. Decreasing the rate of infusion and the administration of antihistamines can control these toxicities.

c. Drug Storage, Reconstitution and Stability

All antibodies will be stored in the investigational pharmacy at 4°C until the day of use.

05/03/01

10/29/03

Once diluted the unlabeled antibody is to be used within 24 hours if held at 4°C and at room temperature for an additional 12 hours. The radiolabeled solutions should be used within 6 hrs and should be held at 2-8°C until administered.

# 4.2 VP-16 (epipodophyllotoxin, etoposide, 4'-demethyl-9(4,6-o-β) d-ethylideneglycopyranoside).

## a. Drug Formulation and Procurement

VP-16 is supplied by Bristol Laboratories in a 100 mg ampule in 5 cc of a solution containing citric acid, 10 mg; benzyl alcohol, 150 mg; polysorbate 80, purified, 250 mg; polyethylene glycol 300, 3.75 gm; absolute alcohol q s., 5 cc.

## b. Drug Toxicity

Myelosuppression, primarily granulocytopenia, is the dose-limiting toxicity. Gastrointestinal toxicity at high doses includes nausea, emesis and mucositis. Reversible hepatotoxicity may occur at very high doses. The acute side effects of occasional bronchospasm and hypotension are avoided by slow intravenous administration.

### c. Drug Storage, Reconstitution and Stability

The contents of the ampoule are diluted with 50 volumes of NaCl solution for injection, USP, and administered by slow intravenous infusion. Patients will receive the drug through a central venous catheter at a rate of 60 mg/kg/4 hours.

## 4.3 Cyclophosphamide (Neosar, Cytoxan), NSC-26271

## a. Drug Formulation and Procurement

Cyclophosphamide is an alkylating agent dispensed in 100, 200 and 500 mg vials containing a dry powder. Cyclophosphamide will be purchased from Adria Laboratories.

### b. Drug Toxicity

Patients must be well hydrated before and for several hours following administration of cyclophosphamide to reduce the potential for hemorrhagic cystitis. The more common side effects include nausea and vomiting, and alopecia. Acute toxicity includes principally leukopenia, with the nadir occurring 7-14 days after a single IV dose. At high doses, occasional pulmonary toxicity has been reported. Rare cardiac toxicity (congestive heart failure) has occurred in patients previously treated with anthracyclines.

#### c. Drug Storage, Reconstitution and Stability

Cyclophosphamide is reconstituted with either sterile water for injection, USP or bacteriostatic water for injection, USP (Paraben preserved only), using 5 ml for the 100 mg vial, 10 ml for the 200 mg vial or 25 ml for the 500 mg vial. Each ml of reconstituted solution contains 20 mg cyclophosphamide per ml. The drug is diluted in 5% dextrose and water or physiological saline and given by IV infusion.

## 4.4 Mesna (Sodium 2-Mercaptoethane sulfonate)

## a. Drug Formulation and Procurement

Mesna is provided by Bristol Laboratories as a 10% (100 mg/ml) solution in water with 0.25 mg EDTA as excipient in 4 ml ampules.

## b. Drug Storage, Reconstitution and Stability

Mesna solutions have been shown to be stable on extended storage at room temperature in ampules. No change in composition of the ampules was noted at one year's storage in these conditions

On exposure to air Mesna is known to undergo oxidation to disulfide. Since the Mesna concentration of opened ampules may decrease with time, the ampule should be opened just before use and the unused part discarded.

#### c. Administration

Each dose of Mesna will be diluted in 50 cc of 5% dextrose/water or 0.9% normal saline and infused intravenously over 15 minutes.

## 4.5 DTPA (Diethyltriaminepenatacetic acid)

## a. Drug Formulation and Procurement

DTPA will be purchased from Heyl Pharmaceuticals, Berlin, Germany. It is supplied as a 1 gram ampule in 5 mls.

#### b. Drug toxicity

DTPA has been known to cause headaches, fever, chills, flu-like symptoms, nasal stuffiness, nausea, vomiting, abdominal cramping, and diarrhea. Other side effects that are less common include pain at the injection site, dehydration, decreased blood pressure, irregularities of heart rhythm, decreased blood counts, increased calcium, numbness and tingling, sneezing, excessive tearing, kidney damage, and zinc deficiency (which can result in a facial and perianal rash and tongue and mouth sores). In addition, there is always a risk of a very uncommon or previously unknown side effect occurring. Stopping the infusion normally reverses the side effects. Headaches and tingling have been observed at the City of Hope but were reversible. Trace metals will be administered at the end of infusion to replace any depleted heavy metals.

#### c. Drug Storage, Reconstitution and Stability

The DTPA solution will be diluted with 250 mls normal saline and administered over 24 hours. Additional IV fluids will be administered to maintain a minimum of 125 mls/hour of fluid. No other heavy metals should be administered during the 24 hour infusion. Potassium may be administered as needed. DTPA has a long aqueous stability but should

06/05/00

be used within 48 hours of being drawn up by the pharmacy. Patients will receive 250 mgs/m<sup>2</sup> to a maximum of a total dose of 500 mgs.

#### 5.0 STAGING CRITERIA

Staging of disease must be evaluated at least 21 days after the end of the last chemotherapy and within 42 days prior to transplant.

5.1 The Ann Arbor staging criteria will be used. Stage is determined based on extent of disease at the time of diagnosis.

## 5.2 Ann Arbor Classification (AJCC Manual for Staging of Cancer, 4th ed. 1992)

| STAGE I | Involvement of a single lymph node region (1) or a single extralymphatic organ or |
|---|---|
| | site $(1_E)$ . |
| <i>STAGE II</i> | Involvement of two or more lymph node regions on the same side of the diaphragm |
| | (II) or localized involvement of an extralymphatic organ or site and its associated |
| | regional lymph nodes $(11_E)$ . |
| STAGE III | Involvement of lymph node regions on both sides of the diaphragm (111) which may |
| | be accompanied by localized involvement of an associated extralymphatic organ or |
| | site $(111_E)$ or spleen $(111_S)$ or both $(II(1_{SE})$ . |
| STAGE IV | Diffuse or disseminated involvement of one or more extralymphatic organs with or |
| | without associated lymph node involvement, or isolated extralymphatic organ |
| | involvement with distant (non-regional) nodal involvement. |
| A = Asymp | ` ' ' |
| | sweats, weight loss > 10% of body weight |
| D - rever, s | sweats, weight loss / 1070 of body weight |

## 5.3 Definitions of Sensitivity of Disease:

Patients are grouped into one of three groups based on sensitivity of disease:

- 1. Induction failure: patients who did not achieve a CR or PR from induction chemotherapy;
- 2. Resistant Relapse: patients who did not achieve a CR or PR from the most recent standard salvage chemotherapy;
- 3. Sensitive Relapse: patients who did achieve a CR or PR from the most recent standard salvage chemotherapy.

## 5.4 Definitions of Poor Risk Disease

05/10/00

- 1. Age Adjusted International Prognostic Index (IPI) High- (3 risk factors) or High-Intermediate (2 risk factors) based on the following risk factors: stage III-IV, elevated serum lactate dehydrogenase level (LDH) and ECOG performance status 2-4.
- 2. Patients with aggressive NHL including mantle cell lymphoma who required 2 different induction chemotherapy regimens to achieve a partial/complete remission.

| 05/03/01 | | 3. Patients with B-Cell NHL who fail to achieve a complete remission after adequate induction chemotherapy regimen(s). |
|---|---|---|
| 05/10/00 | 6.0 | ELIGIBILITY CRITERIA |
| 05/10/00 | 6.1 | Favorable biodistribution on imaging dose |
| 08/07/01 | 6.2 | age $\geq 18$ and $\leq 60$ years |
| 10/29/03 | 6.3 | All patients must have biopsy proven diagnosis of low- and intermediate-grade NHL including follicular small cleaved, follicular mixed, follicular large cell, diffuse small cleaved, diffuse mixed, diffuse large cell, and immunoblastic lymphoma (working formulation B, C, D, E, F, G and H) including mantle cell lymphoma. Transformed low-grade lymphomas are eligible |
| | 6.4 | Demonstrated monoclonal CD20 + B-cell population in lymph nodes and/or bone marrow |
| 05/10/00 | 6.5 | Patients must have relapsed after achieving a complete or partial response to prior therapy, have never responded to prior therapy or have poor risk disease |
| 05/10/00,05/30/02<br>10/29/03 | 6.6 | Patients must have bone marrow aspiration and biopsy within 42 days before salvage chemotherapy or stem cell collection which show $\leq 10\%$ lymphomatous involvement of total cellularity |
| 09/08/00, 05/30/02 | <b>6.</b> 7 | Platelet count should be normal before initiation of chemotherapy for salvage purposes or stem cell mobilization. If the patient collected his/her stem cells at an outside facility, then the platelet count must be normal before the imaging dose of antibody |
| | 6.8 | Normal renal function test with serum creatinine of $\leq 1.5$ mg/dl, or a creatinine clearance of $\geq 60$ ml/min |
| | 6.9 | Adequate pulmonary function as measured by FEV1 $>$ 65% of predicted measured, or a DLCO $\geq$ 50% of predicted measured |
| 04/06/04 | 6.10 | Cardiac Ejection fraction of > 50% by echocardiogram or multiple gated acquisition scan |
| | 6.11 | Adequate liver function tests with a bilirubin of $\leq 1.5~x$ normal and SGOT or SGPT $\leq 2~x$ normal |
| | 6.12 | Negative human immunodeficiency virus antibody |
| 05/03/01 | 6.13 | ECOG performance status 0 or 1; or KPS $\geq$ 80 |
| | 6.14 | No active CNS disease or prior history of CNS disease |
| 07/13/00 | 6.15 | Patients who have received involved field external beam therapy to area excluding lung, heart, liver and kidney are allowed, but will be evaluated on a case by case basis |
| | 6.16 | Patients must have recovered from last therapy and should be at least four weeks from prior radiation or chemotherapy |

| 08/07/01 | <b>6.17</b> | - | hould have a baseline CT scan and Ga 67 scan and/or FDG-PET scan after otherapy prior to initiation of treatment |
|---|---|---|---|
| 10/29/03 | 6.18 | collection). I biopsy has all | genetic study on bone marrow (prior to salvage chemotherapy or stem cell<br>However, cytogenetic study on peripheral blood is acceptable if bone marrow<br>ready been done and shows no sign of MDS or lymphoma and a repeat bone<br>emed unnecessary by attending physician |
| | 7.0 | EXCLUSIO | N CRITERIA |
| | 7.1 | Presence of h | numan anti-mouse antibody (HAMA) or human anti-chimeric antibody |
| | 7.2 | Prior radioim | munotherapy |
| | 7.3 | Failure to col | lect adequate number of CD34 + cells $\geq 3x10^6$ /kg |
| | 7.4 | Abnormal cy collection | togenetic study on the bone marrow aspirate sample prior to stem cell |
| | 7.5 | Prior bone ma | arrow transplantation |
| 07/13/00 | 7.6 | adequately tre | ancy except for adequately treated basal cell or squamous cell skin cancer, eated noninvasive carcinomas, or other cancer from which the patient has free for at least five years |
| | 7.7 | Active evider | nce of Hepatitis B and C infection; Hepatitis B surface antigen positive |
| 02/08/01 | <b>7.8</b> | History of alc | cohol abuse |
| 10/29/03 | 7.9 | Patient weigh | ns more than 250 pounds |
| | 8.0 | TREATME | NT PLAN |
| | <i>8.1</i> | Outline of th | e preparative regimen |
| | | <i>Day -21</i> | Dosimetry with 5 mCi IDEC-In2B8 following 250 mg/M <sup>2</sup> Rituxan |
| | | <i>Day -14</i> | IDEC-Y2B8 with 5 mCi IDEC-In2B8 following 250 mg/M <sup>2</sup> Rituxan |
| 05/30/02 | | <i>Day -7</i> | Bone marrow biopsy and dose estimation |
| 05/30/02, 10/29/03 | | Day -4 | Etoposide 40 mg/kg adjusted ideal body weight (Cohort 1) or 60 mg/kg adjusted ideal body weight for other cohorts |
| 10/29/03 | | <i>Day -2</i> | Cyclophosphamide 100 mg/kg ideal body weight |
| 06/05/00 | | Day 0 | DTPA infusion |
| | | <i>Day</i> +1 | Peripheral Stem Cell reinfusion |
| | | Dav + 1 | Start G-CSF 5 ug/kg/d IV |

## 8.2 Pre-Transplant Therapy

a. Autologous Stem Cell Collection and Cryopreservation

All patients should have bone marrow aspiration and biopsy which show no microscopic evidence of lymphomatous involvement, or  $\leq 10\%$  involvement at the time of stem cell collection. In addition, cytogenetic studies, immunophenotyping, gene rearrangement should be done. Peripheral blood stem cells (PBSCs) will be collected via leukapheresis procedures that have been previously described. Patients will receive PBSCs collected after mobilization by: 1) growth factors, ie. G-CSF 10  $\mu$ g/kg/d or 2) chemotherapy with growth factors. A minimum of CD34+ cells, 3.0 x 10<sup>6</sup>/kg should be collected.

## b. Trimethoprim Sulfa

All patients should receive trimethoprim sulfa (one double-strength tablet PO bid) beginning day -8 through day -2 prior to PBSCT as prophylaxis against PCP. (The choice of trimethoprim sulfa as a prophylactic agent may be altered based on a history of sensitivity to this agent.) Dosing should be discontinued 48 hours prior to PBSC infusion because of potential myelosuppression.

c. CNS Prophylaxis

CNS prophylaxis is recommended for patients with mantle cell lymphoma or diffuse large cell lymphoma who had bone marrow involvement at diagnosis or at time of relapse. For patients with mantle cell lymphoma who have never received high-dose MTX, CNS prophylaxis with intrathecal chemotherapy should be given.

## 8.3 Radioimmunotherapy

- a. Rituxan is to be administered by slow intravenous infusion having been diluted to 1-4 mg/ml in saline. Initial infusion should be through a dedicated line at a rate of 50 mg/hr. If hypersensitivity or infusion-related events do not occur, escalate the infusion rate in 50 mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr. If hypersensitivity or infusion-related events develop, the infusion should be temporarily slowed or interrupted. The infusion can be continued at one-half the previous rate when symptoms abate.
- b. IDEC-In2B8 Administration Two mg of IDEC-In2B8 (5.0 mCi of <sup>111</sup>In) will be administered for the dosimetry portion of the protocol. The imaging dose will be administered over 10 minutes by slow IV injection immediately following the infusion of Rituxan. A .22 micron filter must be on the line between the patient and the infusion port. Flush the line with at least 10 mls of normal saline after the IDEC-In2B8 has been infused.
- c. IDEC-Y2B8 Administration IDEC-Y2B8 (40-100 mCi of <sup>90</sup>Y with 3.2 6.4 mg of antibody) will be administered for the therapy portion of the protocol. The yttrium will be combined with a dose of IDEC-In2B8 (5.0 mCi of <sup>111</sup>In) identical to the dosimetry dose. The combined radiopharmaceuticals will be administered

10/29/03

07/13/00

10/29/03

08/07/01

by controlled infusion pump over 20 minutes. A .22 micron filter must be on the line between the patient and the infusion port. Flush the line with at least 10 mls of normal saline after the IDEC-In/Y2B8 has been infused.

*d.* Bone marrow biopsy.

## 8.4 Chemotherapy

10/25/00, 12/20/00

VP-16 is to be administered as a single infusion on day -4. The dose is 40 or 60 a. mg/kg and is calculated on adjusted ideal body weight to be consistent with standard VP-16 dosing for transplant protocols. The drug is infused undiluted directly into a port of a double or triple lumen indwelling intravenous catheter, with a total infusion time of 4 hours. The drug is to be drawn into one or more plastic syringes and infused with a syringe infusion pump, placed in an evacuated bottle and infused through a pediatric infusion pump, or infused by gravity without a pump. Thus the total dose for a 70 kg patient would be 4,200 mg. At 20 mg/ml, the volume of VP-16 would be 210 ml. The rate of infusion would thus be 210 ml/240 minutes or 0.875 ml/minute. Appropriate anti-emetics and sedatives should be given before the infusion begins. Before, and 2 hours into, the infusion the patient is to receive 25 mg of diphenhydramine, and 100 mg of hydrocortisone to prevent allergic reactions. If necessary, diuretics may be given. The intravenous hydration should be continued before, during and after the VP-16. Since in rare cases metabolic acidosis has been observed after high dose VP-16, additional NaHCO3 may be needed.

10/29/03

b. Cyclophosphamide is administered at a total dose of 100 mg/kg given in one dose on day -2 and is calculated on ideal body weight. Adjustments to the ideal body weight calculation for overweight patients are permitted. For patients who are weigh less than 95% of ideal body weight, cyclophosphamide will be dosed according to actual body weight. The drug should be dissolved in about 250 cc of D5W and infused IV over two hours. Appropriate anti-emetics and sedatives should be given. To prevent hemorrhagic cystitis, all patients should receive hydration with intravenous fluids, according to institutional standards, at the rate of 3.0 l/m2/day beginning four hours prior to cyclophosphamide and continuing until 24 hours after cyclophosphamide. In addition, mesna at 40 mg/kg (based on ideal body weight) will be given immediately before cyclophosphamide (hr 0) and at 3, 6, 9, 12, 15, 18 and 21 hrs later for a total of 8 doses. Each dose of mesna will be given IV over 15 minutes.

06/05/00, 10/29/03, 06/16/04

c. DTPA is to be administered by continuous intravenous infusion through a port of a double or triple lumen indwelling intravenous catheter. The dose should be ≥ 250 mgs/m², but ≤ 500 mgs. The DTPA should be made up in normal saline and infused over 24 hours by infusion pump. No magnesium or other heavy metal should be given during the same time period. Two hours after the end of the DTPA infusion 1 ml of trace metal solution should be infused every eight hours for five days. This should be given by slow intravenous delivery or else as part of standard hyperalimentation. Urine samples will be collected every 12 hours for

72 hours beginning 24 hours prior to DTPA infusion.

## 07/13/00, 05/03/01 8.5 Peripheral Stem Cell Reinfusion

PBSCs will be thawed and infused according to standard guideline at approximately 72 hours after completion of cyclophosphamide.

## 8.6 Growth Factor Therapy

All patients will receive rh-G-CSF, 5 mcg/kg/day IV beginning on day +1, after PBSC infusion and continue daily until ANC >500 for 3 consecutive days.

## 8.7 Supportive Care:

07/13/00

All patients will be housed in private rooms during the period of granulocytopenia. Nonabsorbable antibiotics for gastrointestinal decontamination should be used according to institutional guideline. Trimethoprim-sulfamethoxazole will be administered from day -8 to day -2 and prophylaxis should be re-instituted when white blood cells are > 3000 and continued until 6 months post-transplant. Empiric broad spectrum antibiotics and parenteral nutrition should be used as clinically indicated. Low-dose amphotericin-B (0.1 to 0.2 mg/kg) should be administered on day +1 and continued daily until granulocytopenia resolves. All blood components should be irradiated to 1,500 cGy.

#### a. Access to Vessels

Prior to admission, during pre-transplant evaluation, all patients should have a permanent central catheter placed.

## b. Hyperalimentation

All patients will receive appropriate Hyperalimentation as soon as necessary after admission. The goal will be to prevent even a short duration of negative nitrogen balance.

## c. Platelet Transfusion

- 1. Indication. Platelets are transfused to prevent bleeding and an attempt is made to keep the circulating level greater than 20,000/mm3 at all times. This goal may be changed by the attending physician as clinically indicated.
- 2. Irradiation. All blood products (except the autologous stem cells) are irradiated with 1,500 cGy prior to infusion.

## d. Management of Fever/Infections

Treatment of patients on this protocol is not intended to restrict the freedom of the managing physician to treat suspected or documented infections. In neutropenic patients, however, the following guidelines should be followed.

1. All febrile, neutropenic patients should be treated with IV antibiotic(s), the choice

- of which should be guided by the patient's clinical history, institutional practices and subsequent culture results.
- 2. Patients with documented, invasive fungal infection or with persistent, unexplained fevers while neutropenic and on broad-spectrum antibiotic therapy should receive antifungal therapy with Amphotericin-B.

## 8.8 Criteria for Removal from Protocol Treatment

- a. Progression of disease.
- b. Patients may withdraw from study at any time for any reason.
- 8.9 All reasons for discontinuation of treatment must be documented in the Flow Sheets.
- **8.10** All patients will be followed for survival until death. Secondary malignancy monitoring on this protocol will be done through 5 years post HCT. After such time, secondary malignancy monitoring will be done by the Long Term Follow Up office.

#### 9.0 STUDY DESIGN AND RULES FOR DOSE ESCALATION

This is a phase I/II trial. For the phase I portion of the study, the rules for dose escalation, dose expansion, and termination of escalation are given in section 9.2. Prior to treatment with Y2B8, patients are required to undergo an imaging scan to verify that they have a favorable biodistribution. While waiting to assess toxicities in the initial cohort of 3 to 6 patients, additional patients who are determined to be eligible may be accrued at the unescalated dose level. The rationale for this is twofold. First, patients must be evaluated for distribution as soon as possible in order to have patients ready for timely accrual to the next dose level. If the dose escalation decision is delayed, the investigators want to treat the patients at the unescalated dose level so that their disease does not progress. Second, patients will be accrued to unescalated dose levels to avoid a loss of momentum in patient accrual. Modifications to the standard phase I design involving accrual of cohorts of 3-6 patients per dose level have been incorporated to appropriately handle the varying number of patients accrued to each dose level (see section 9.2). Study design considerations and targeted response rates for the phase II portion of the trial are given in section 9.3. Because the eligibility criteria are the same for both the phase I and the phase II portions of the trial, the patients treated at the dose level defined as the MTD from the phase I portion of the trial will count towards the accrual for the phase II portion of the trial.

#### 9.1 Dose Limiting Toxicity (DLT)

Dose limiting toxicity (DLT) in a given patient is defined as any grade III non-hematologic toxicity not reversible to grade II or less within 96 hours, or any grade IV non-hematologic toxicity. Toxicity will be graded according to the NCI Common Toxicity Criteria (CTC) version 2.0 and toxicity Module (Appendices I and II, http://ctep.info.nih.gov/ctc3/ctc.htm) with the addition of BMT Complex/Multi-Component Events (Appendix VI, http://ctep.info.nih.gov/ctc3/ctc.htm). To be evaluable for toxicity, a patient must receive a complete course of treatment and be observed for 6 weeks after the administration of Y2B8 or have experienced a DLT. All patients who are not evaluable for toxicity will be replaced.

05/03/01

# 9.2 Definition of Maximum Tolerated Dose (MTD) and DLT-Level and Rules for Dose Escalation

This trial differs from the standard phase I design in that additional patients beyond the standard 3 or 6 patients per dose level may be accrued to the current dose level while waiting to assess toxicities in the initial 3 or 6 patients. To this end, a decision rule has been added that incorporates toxicity information from the additional patients accrued to a dose level. As toxicity information on each additional patient accrued to the trial becomes available, the decision to escalate, de-escalate and expand the previous dose level, expand the current cohort or stop the trial will be evaluated. The decision rule (R) will be as follows: Let x = number of DLTs in n patients. Escalate to the next dose level if R = (x + 0.5) / (n + 2) is  $\leq 0.20$ . Stop accrual to a dose level if R > 0.30. Continue accrual to a dose level if R = 0.30. A minimum of three patients must be accrued to a dose level. As soon as 3 patients have been accrued to a dose level and toxicity has been assessed, escalation to the next level is allowed, provided that acceptable toxicity has been observed. If accrual to a dose level must be expanded due to toxicity, a minimum of 6 patients must be accrued to the expanded dose level.

Operationally, the rule is to close a dose level and de-escalate if 2 DLTs are observed among 6 or fewer patients, or if 3 DLTs are observed among any number of patients. The dose will be escalated if 0 DLTs are observed in 3 or more evaluated patients, if 1 DLT is observed in 6 or more evaluated patients, or if 2 DLTs are observed in 11 patients. At most, 11 patients will be accrued to a dose level. However, if a dose is escalated while toxicity follow-up is still outstanding for some patients, the accumulating results from the two dose levels may be pooled for the purpose of justifying the continued accrual to the higher dose.

Table 1 shows values for R based on different combinations of DLTs and numbers of patients. Values indicating continued accrual to the current dose are shown in bold.

Table 1

| | Nu | mber of DLTs | (x) |
|------------------------|------|--------------|------|
| Number of Patients (n) | 0 | 1 | 2 |
| 3 | 0.10 | 0.30 | 0.50 |
| 4 | 0.08 | 0.25 | 0.42 |
| 5 | 0.07 | 0.21 | 0.36 |
| 6 | 0.06 | 0.19 | 0.31 |
| 7 | 0.06 | 0.17 | 0.28 |
| 8 | 0.05 | 0.15 | 0.25 |
| 9 | 0.05 | 0.14 | 0.23 |
| 10 | 0.04 | 0.13 | 0.21 |
| 11 | 0.04 | 0.12 | 0.19 |

This criterion is the posterior mean with a beta (0.5, 1.5) prior, which has a smaller mean, but is no more informative than a flat prior. The criterion is consistent with the conventional rule of expanding a dose level to six patients if 1 out of 3 patients experience DLT and stopping if 2 or

more patients out of 6 treated at the same dose level experience DLT. The proposed criterion rationalizes the conventional design in order to rationally extend if to larger numbers of patients per dose level. The rationalization is that a dose level is opened with a weak prior expectation of a 25% DLT rate, and the dose is escalated or de-escalated as the accumulating data indicate a rate below 20% or above 30%.

The phase I portion of the trial will be closed when 6 patients have been accrued to the highest dose level below the DLT level with at most 1 patient experiencing DLT or when 11 patients have been accrued with at most 2 patients experiencing DLT. This dose level will be defined as the MTD.

To demonstrate an application of the escalation rule, consider the following examples:

Example 1: Three patients are accrued to dose level 1. A fourth patient is accrued to the trial prior to assessment of toxicity for the third patient and is therefore also treated at dose level 1. No DLTs are observed in the first 3 patients such that the fifth patient is accrued to dose level 2 and subsequent to this the fourth patient accrued to dose level 1 experiences a DLT. With 1 DLT in four patients, from Table 1 the value for R is 0.25 therefore accrual to dose level 2 must be halted such that accrual to dose level 1 can be expanded. Six patients will need to be accrued with at most 1 out of 6 patients experiencing DLT in order for accrual to dose level 2 to resume. The patient treated at dose level 2 may be counted among the required 6 patients if no DLT is encountered.

Example 2: Dose level 3 is expanded such that 6 patients are accrued. A seventh patient is accrued to the trial prior to assessment of toxicity for the sixth patient and is therefore also treated at dose level 3. Only one DLT is observed in the first 6 patients such that the eighth patient is accrued to dose level 4 and subsequent to this the seventh patient accrued to dose level 3 experiences a DLT. With 2 DLTs in seven patients, from Table 1 the value for R is 0.28 therefore accrual to dose level 4 must be halted so that accrual to dose level 3 can be expanded. Eleven patients (including the patient treated at dose level 4) will need to be accrued to dose level 3 (or above) with at most 2 patients experiencing DLTs in order for accrual to dose level 4 to resume. Two DLTs among 11 patients corresponds to R = 0.19 which is consistent with 1 DLT among 6 patients. A maximum of 11 patients can be accrued to a single dose level.

## 9.3 Design Considerations for the Phase II Trial

All patients accrued to the dose level established to be the MTD will be included in the assessment of response for the phase II portion of the trial. The primary goal of this portion of the trial is to obtain estimates of the efficacy of IDEC-Y2B8 in combination with high-dose etoposide and cyclophosphamide followed by ASCT for treatment of patients with relapsed and refractory NHL. A minimum of 17 and a maximum of 37 patients will be accrued to this portion of the trial. Justification for the sample size as well as a description of the study design for the phase II portion of the trial is provided in section 12.0.

10/29/03

10/29/03 10/29/03 08/07/01, 10/2 10/29/03 10/29/03

08/07/01

10/29/03 08/07/01, 05/3 05/03/01

05/30/02 05/30/02

08/07/01, 10/2 04/06/04

06/16/04 06/16/04 06/05/00

05/30/02, 10/29/03 10/29/03

10/29/03 10/29/03

#### 10.0 STUDY CALENDAR - PREPARATIVE REGIMEN AND PBSCT

| REQUIRED STUDIES | Pre<br>Study | DAY<br>-21 | DAY<br>-14 | DAY<br>-7 | DAY<br>-4 | DAY<br>-2 | DAY<br>0 | DAY<br>7 | DAY<br>14 | DAY<br>30 | DAY<br>60 | DAY<br>100 | DAY<br>180 | YR<br>1 | YR<br>2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PHYSICAL | | | | | | | | | | | | | | | |
| H & PE | X | | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> |
| Weight and KPS | X | | | X | | | X | | | X | X | X | X | X | X <sup>\$</sup> |
| Tumor Assessment | X | | | | | | | | | X | | | X | X | X <sup>\$</sup> |
| Toxicity Notation | | | | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> | X <sup>\$</sup> |
| LABORATORY | | | | | | | | | | | | | | | |
| CBC/Platelets | X | | | X | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> |
| Differential <sup>¥</sup> | X | | | X | | | | X | X | X | X | X | X | X | X <sup>\$</sup> |
| HAMA/HACA | X | | | | | | | | | | X | X | X" | X | |
| Comp Metabolic Panel + LDH | X | | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>\$</sup> |
| Magnesium | X | | X | X | X | X | X | X | X | X | | | | | |
| PT/PTT | X | | | | | | | | | | | | | | |
| Immunoglobulin Levels | X | | | | | | | | | X | | X | X | X | |
| Peripheral Blood Mononuclear<br>Immunophenotyping | X | | | | | | | | | X | | X | X | X | |
| CMV Titer | X | | | | | | | | | | | | | | |
| Hepatitis Profile | X | | | | | | | | | | | | | | |
| Herpes Simplex | X | | | | | | | | | | | | | | |
| HIV Antibody | X | | | | | | | | | | | | | | |
| BM <sup>%</sup> , # | X | | | Χ^ | | | | | | | | X | | X | X |
| Creatinine Clearance | | | | | | | | | | | | | X | X | |
| X-RAYS AND SCANS | | | | | | | | | | | | | | | |
| Chest X-ray or CT Chest | X | | | X | | | X | | X | X | | X | X | X | X <sup>&amp;</sup> |
| CT scans*, + | X | | | | | | | | | X | | X | X | X | X <sup>&amp;</sup> |
| EKG | X | | | | | | | | | | | | | X | |
| MUGA or ECHO | X | | | | | | | | | | | | X | X | |
| DLCO/FEV1 | X | | | | | | | | | | | | X | X | |
| Ga 67 Scan and/or FDG-PET Scan | $X^{\phi}$ | | | | | | | | | $X^{\Diamond}$ | | | X | X | |
| TREATMENT | | | | | | | | | | | | | | | |
| Stem Collections | X | | | | | | | | | | | | | | |
| IDEC-In2B8 | | X | X | | | | | | | | | | | | |
| IDEC-Y2B8 | | | X | | | | | | | | | | | | |
| Rituxan | | X | X | | | | | | | | | | | | |
| VP-16 | | | | | X | | | | | | | | | | |
| Cyclophosphamide | | | | | | X | | | | | | | | | |
| PBSCT | | | | | | | X§ | | | | | | | | |
| G-CSF | | | | | | | X§ | | | | | | | | |
| DTPA | | | | | | | X | | | | | | | | |

10/29/03 (delete @.06/20/07) & restaging at Day 100, at 6 months then follow-up evaluation every six months for three years, and then yearly up to 5 yrs post BMT

% bone marrow aspiration and biopsy, cytogenetic study, immunophenotyping and gene rearrangement

05/30/02, 06/20/07 # Follow-up bone marrow is required at day 180, yr 1 up to 5 yrs post BMT.

+ For pts in CR at time of transplant, CT scans to be done between days 30 and 100.

« Day 180 HAMA/HACA acceptable between days 150 and 210

¢ Pre-study PET scan should be done 14 days after stem cell collection to avoid GCSF enhancement effect

¥ ANC is acceptable in lieu of differential

06/16/04 § Day +1

<sup>\$</sup> All late complications such as cataracts formation and occurrence of second malignancies must be documented and reported.

<sup>\*</sup> CT scans of chest, abdomen and pelvis as indicated

#### 11.0 CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS

## **Definitions**

- a. Measurable Disease: Bidimensionally measurable lesions with clearly defined margins by: 1) medical photograph (skin or oral lesion), or plain x-ray with at least one diameter .5 cm or greater (bone lesions are not included) or, 2) CT, MRI or other imaging scan with both diameters greater than the distance between cuts of the imaging study, or 3) palpation with both diameters 2 cm or greater.
- b. Evaluable Disease: Unidimensionally measurable lesions, masses with margins not clearly defined, lesions with both diameters less than 0.5 cm, lesions on scan with either diameter smaller than the distance between cuts, palpable lesions with either diameter less than 2 cm, bone disease.
- c. Non-Evaluable Diseases: Pleural effusions, ascites, disease documented by indirect evidence only (e.g., by lab values).
- d. Objective Status, To Be Recorded at Each Evaluation: If an organ has too many measurable lesions to measure at each evaluation, choose three to be followed before the patient is entered on study. The remaining measurable lesions in that organ will be considered evaluable for the purpose of objective status determination. Unless progression is observed, objective status can only be determined when ALL is measurable and evaluable sites and lesions are assessed.

## 11.1 Complete Response (CR)

Complete disappearance of all measurable evidence of non-evaluable disease. No new lesions. No disease related symptoms. No evidence of non-evaluable disease, including normalization of markers and other abnormal lab values. All measurable, evaluable and non-evaluable lesions and sites must be assessed using the same techniques as baseline. Refers to clinical CR-when restaging surgery is required, a separate pathologic response variable is defined.

## 11.2 Partial Response (PR)

Applies only to patients with at least one measurable lesion. Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. All measurable and evaluable lesions and sites must be assessed using the same techniques as baseline.

#### 11.3 Stable Disease (SD)

Does not qualify for CR, PR or Progression. All measurable and evaluable sites and lesions must be assessed using the same techniques as baseline.

#### 11.4 Progressive Disease (PD)

50% increase or an increase of 10 cm<sup>2</sup> (whichever is smaller) in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same

05/30/02

techniques as baseline, OR clear worsening of any evaluable disease, OR reappearance of any lesion which had disappeared, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). For "scan only" bone disease, increased uptake does not constitute clear worsening. Worsening of existing non-evaluable disease not constitute progression.

#### 11.5 Relapse

Relapse is defined as the re-appearance of any clinical evidence of lymphoma in a patient who has had a CR. Relapse for partial responders are defined as progressive disease relative to disease status during the partial remission.

## 11.6 Duration of Response

This is measured from the documented beginning of response (CR or PR)

## 11.7 Performance Status

Patients will be graded according to the current Performance Status Scales/Scores (Appendix IV).

## 11.8 Time to Progression

From date of registration to date of first observation of progressive disease or death due to any cause.

#### 11.9 Time to Death

From date of registration to date of death due to any cause.

#### 12.0 STATISTICAL CONSIDERATIONS

## 12.1 Study Design and Justification of Sample Size

The definition of dose limiting toxicity is given in section 6.1. The maximum tolerated dose is defined in section 6.2. The number of patients to be treated at each dose level examined in the phase I trial as well as the rules for dose escalation is given in section 6.2.

The phase II portion of the study will follow a two-stage minimax design suggested by Simon (1). It is assumed that a true response rate less than 20% would not warrant further study of this agent. It is also assumed that a response rate of 40% would be considered promising for further studies in these patients. In the first stage, seventeen evaluable patients will be entered. If less than four responses are observed, the accrual will stop with the conclusion that the regimen is not promising for further study. If four or more responses are observed in the first 17 patients, additional 20 patients will be accrued during the second stage of the study. Eleven or more responses out of 37 patients will be considered as evidence warranting further study of the regimen providing other factors, such as toxicity and survival, also appear favorable. If less than 11 responses out of 37 patients are observed, further study of the regimen would not be warranted.

The probability of falsely declaring an agent with a 20% response probability as warranting further

08/07/01

study is 0.10 (alpha) and the probability of correctly declaring an agent with a 40% response probability as warranting further study is 0.90 (power). With 37 patients the true probability of response can be estimated with a maximum standard error equal to 0.08.

The phase I portion study is expected to accrue a minimum of 15-18 evaluable patients and a maximum of 30. The phase II portion of the study will accrue a minimum of 17 patients and a maximum of 37 patients, of which at least six of these patients will have been included in the phase I portion of the study. It should take approximately 24-36 months to complete both the phase I and phase II portions of this trial.

## 12.2 Analysis of Clinical Endpoints

Patients will be considered evaluable for response and evaluable for toxicity as outlined in section 11.0. The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI Common Toxicity Criteria and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course. Baseline information (e.g. the extent of prior therapy) and demographic information will be presented, as well, to describe the patients treated in the phase I portion of the study. All responses will be reported from the phase I portion of the study

Response rates and duration of response will be estimated for the phase II portion of survival. Confidence intervals for the response rate will be established by calculating exact 95% confidence limits for a binomial parameter. The duration of overall and disease-free survival of the patient will be estimated using the product-limit method of Kaplan and Meier.

#### 13.0 REGISTRATION GUIDELINES

Once a signed, written informed consent has been obtained and all pretreatment evaluations have been performed, patients will be entered on study, after review of patient eligibility criteria by the assigned Data Manager from the City of Hope Department of Biostatistics. Patients may be screened for registration by calling the Department of Biostatistics, ext. 62468.

#### 14.0 RECORDS TO BE KEPT AND DATA SUBMISSION SCHEDULE

## 14.1 Confidentiality of Records

The original data collection forms will be stored in secure cabinets in the Department of Biostatistics. All radioimmunotherapy associated data will be kept in the Department of Radioimmunotherapy.

#### 14.2 Patient Consent Form

At the time of registration, signed and dated copies of the patient Informed Consent form with the Human Rights must be available (for patient, chart, and Biostatistics Office).

08/07/01

#### 15.0 GENDER AND MINORITIES

# 15.1 Planned Gender and Minority Inclusion for Transplant Patients with Intermediate Grade Lymphoma at City of Hope

| | American<br>Indian or | Asian or<br>Pacific | Black,<br>not of | Hispanic | White,<br>not of | White,<br>Hispanic | Other or<br>Unknown | Total |
|---|---|---|---|---|---|---|---|---|
| | Alaskan<br>Native | Islander | Hispanic<br>Origin | | Hispanic<br>Origin | or not-<br>Hispanic<br>Unknown | | |
| Female | 0% | 9% | 4% | 16% | 54% | 17% | 0% | 100% |
| Male | 0% | 5% | 2% | 20% | 60% | 12% | 1% | 100% |
| Unknown | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |

# 15.2 Actual Gender and Minority Inclusion for Transplant Patients with Intermediate Grade Lymphoma at City of Hope

| | American | Asian or | Black, | Hispanic | White, | White, | Other or | Total |
|---|---|---|---|---|---|---|---|---|
| | Indian or | Pacific | not of | | not of | Hispanic | Unknown | |
| | Alaskan | Islander | Hispanic | | Hispanic | or not- | | |
| | Native | | Origin | | Origin | Hispanic | | |
| | | | | | | Unknown | | |
| Female | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |
| Male | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |
| Unknown | 0% | 0% | 0% | 0% | 0% | 0% | 0% | 0% |

#### 16.0 DATA MANAGEMENT

Clinical Statistics maintains a patient database at City of Hope Medical Center, Department of Biostatistics to allow storage and retrieval of patient data collected from a wide variety of sources. The investigator will ensure that data collected conform to all established guidelines for coding, collection, key-entry, and verification. All patients are assigned a unique patient number to assure patient confidentiality. Any publications or presentations refer to patient by unique patient number, not name. The licensed medical records department, affiliated with the institution where the patient receives medical care, maintains all original inpatient and outpatient chart documents. Patient research files are kept in a locked room. They are maintained by the COHMC data collection staff. Access is restricted to personnel authorized by the Division of Clinical Research.

#### 17.0 ETHICAL AND REGULATORY CONSIDERATIONS

This study is to be approved by the Institutional Review Board according to City of Hope ethical and regulatory guidelines. All patients will have signed an informed consent for participation in research activities, and will have been given a copy of the Experimental Subject's Bill of Rights.

When results of this study are reported in medical journals or at meetings, identification of those taking part will be withheld. Medical records of patients will be maintained in strictest confidence,

according to current legal requirements. However, they will be made available for review, as required by the Food and Drug Administration (FDA) or other authorized users such as the National Cancer Institute (NCI), under the guidelines established by the Federal Privacy Act, or IDEC Pharmaceuticals Corporation.

#### 18.0 REFERENCES

- 1. Parker SL, Tong T, Bolden S, Wingo PA: Cancer Statistics, 1997 [published erratum appears in CA Cancer J Clin 1997 Mar-Apr;47(2):68]. CA.Cancer J.Clin. 47:5, 1997
- 2. Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CAJ, Miller TP: Comparison of a Standard Regimen (CHOP) with Three Intensive Chemotherapy Regimens for Advanced Non-Hodgkin's Lymphoma [see comments]. N.Engl.J.Med. 328:1002, 1993
- 3. Vose JM, Anderson JR, Kessinger A, Bierman PJ, Coccia P, Reed EC, Gordon B, Armitage JO: High-Dose Chemotherapy and Autologous Hematopoietic Stem-Cell Transplantation for Aggressive Non-Hodgkin's Lymphoma [see comments]. J.Clin.Oncol. 11:1846, 1993
- 4. Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL: Autologous Bone Marrow Transplantation as Compared with Salvage Chemotherapy in Relapses of Chemotherapy-Sensitive Non-Hodgkin's Lymphoma [see comments]. N.Engl.J.Med. 333:1540, 1995
- 5. Bierman PJ, Vose JM, Anderson JR, Bishop MR, Kessinger A, Armitage JO: High-Dose Therapy with Autologous Hematopoietic Rescue for Follicular Low-Grade Non-Hodgkin's Lymphoma. J.Clin.Oncol. 15:445, 1997
- 6. Nademanee A, Schmidt GM, O'Donnell MR, Snyder DS, Parker PM, Stein A, Smith E, Molina A, Wong KK, Stepan DE, Margolin KA, Somlo G, Raschko J, Sniecinski I, Lipsett JA, Dagis A, Niland JC, Forman SJ: Fractionated Total Body Irradiation (FTBI), High-Dose Etoposide (VP-16) and Cyclophosphamide (CY) Followed by Autologous Bone Marrow Transplantation (ABMT): The Results in 110 Patients with Non-Hodgkin's Lymphoma (NHL). Blood 82:143a (559), 1993 (abstr.)
- 7. Horning SJ, Negrin RS, Chao JC, Long GD, Hoppe RT, Blume KG: Fractionated Total-Body Irradiation, Etoposide, and Cyclophosphamide Plus Autografting in Hodgkin's Disease and Non-Hodgkin's Lymphoma. J.Clin.Oncol. 12:2552, 1994
- 8. Weaver CH, Petersen FB, Appelbaum FR, Bensinger WI, Press O, Martin P, Sandmaier B, Deeg HJ, Hansen JA, Brunvand M: High-Dose Fractionated Total-Body Irradiation, Etoposide, and Cyclophosphamide Followed by Autologous Stem-Cell Support in Patients with Malignant Lymphoma. J.Clin.Oncol. 12:2559, 1994
- 9. Maloney DG, Grillo-Lopez AJ, White CA, Bodkin D, Schilder RJ, Neidhart JA, Janakiraman N, Foon KA, Liles TM, Dallaire BK, Wey K, Royston I, Davis T, Levy R: IDEC-C2B8 (Rituximab) Anti-CD20 Monoclonal Antibody Therapy in Patients With Relapsed Low-Grade Non-Hodgkin's Lymphoma. Blood 90:2188, 1997
- McLaughlin P, Grillo-López AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK: Rituximab Chimeric Anti-CD20 Monoclonal Antibody Therapy for Relapsed Indolent Lymphoma: Half of Patients Respond to a Four-Dose Treatment Program. Journal of Clinical Oncology 16:2825, 1998
- 11. Czuczman M, Grillo-López AJ, White CA, Saleh M, Gordon L, LoBuglio AF, Jonas C, Dallaire B, Varns C: IDEC-C2B8/CHOP Chemoimmunotherapy in Patients With Low-

- Grade Lymphoma: Clinical and BCL-2 (PCR) Final Results. Blood 88:453a (1799), 1996 (abstr.)
- 12. Kaminski MS, Zasadny KR, Francis IR, Milik AW, Ross CW, Moon SD, Crawford SM, Burgess JM, Petry NA, Butchko GM: Radioimmunotherapy of B-Cell Lymphoma with [131][Anti-B1 (Anti-CD20) Antibody. N.Engl.J.Med. 329:459, 1993
- 13. Stagg R, Wahl RL, Estes J, Tidmarsh G, Kroll S, Shochat D, Zasadny K, Kaminski MS: Phase I/II Study of Iodine-131 Anti-B1 Antibody for Non-Hodgkin's Lymphoma (NHL): Final Results. Proceedings of ASCO 17:39a (150), 1998 (abstr.)
- 14. Vose J, Saleh M, Lister A, Rohatiner A, Knox S, Radford J, Zelenetz AD, Stagg R, Tidmarsh G, Wahl R, Kaminski MS: Iodine-131 Anti-B1 Antibody for Non-Hodgkin's Lymphoma (NHL): Overall Clinical Trial Experience. Proceedings of ASCO 17:10a (38), 1998 (abstr.)
- 15. Press OW, Eary JF, Appelbaum FR, Martin PJ, Badger CC, Nelp WB, Glenn S, Butchko G, Fisher D, Porter B: Radiolabeled-Antibody Therapy of B-Cell Lymphoma With Autologous Bone Marrow Support [see comments]. N.Engl.J.Med. 329:1219, 1993
- 16. Press O, Eary J, Liu S, Petersdorf S, Bush S, Durack L, Martin P, Maloney D, Matthews D, Fisher D, Gooley T, Appelbaum F, Bernstein I: A Phase I/II Trial of High Dose Iodine-131-Anti-B1 (Anti-CD20) Monoclonal Antibody, Etoposide, Cyclophosphamide, and Autologous Stem Cell Transplantation for Patients With Relapsed B Cell Lymphomas. Proceedings of ASCO 17:3a (9), 1998 (abstr.)
- 17. Knox SJ, Goris ML, Trisler K, Negrin R, Davis T, Liles TM, Grillo-Lopez A, Chinn P, Varns C, Ning S, Fowler S, Deb N, Becker M, Marquez C, Levy R: Yttrium-90-Labeled Anti-CD20 Monoclonal Antibody Therapy of Recurrent B-Cell Lymphoma. Clin.Cancer Res. 2:457, 1996
- 18. Witzig T, Wiseman G, White CA, Solinger A, Gordon L, Raubitschek A, Emmanoulides C, Royston I, Parker E, Chinn P, Grillo-López A: IDEC-Y2B8 <sup>90</sup>Yttrium Anti-CD20 Radioimmunotherapy of Relapsed Non-Hodgkin's Lymphoma (NHL): Interim Results of a Phase I/II Trial. Blood 90:586a (2606), 1997 (abstr.)
- 19. Wiseman GA, Solinger AM, Grillo-López A, Stabin M, Dunn WL, Witzig TE, Spies S, Gordon L, Raubitschek A, Margolin K, Karvelis K, Janakiraman N, Silverman DH, Emmanoulides C, Royston I, Chinn P, Parker E, Carter W, White CA: IDEC-Y2B8 (90 Y Conjugated Anti-CD20) Dosimetry Calculated From 111 In Anti-CD20 in Patients With Low and Intermediate Grade B-Cell Non-Hodgkin's Lymphoma (NHL) Emphasis on Bone Marrow (BM). Blood 90:510a (2273), 1997 (abstr.)
- Witzig TE, White CA, Wiseman GA, Gordon LI, Emmanoulides C, Raubitschek A, Janakiraman N, Gutheil J, Schilder RJ, Spies S, Silverman DH, Parker E, and Grillo-López A: Phase I/II Trial of Yttrium 90 Ibritumomab Tiuxetan (IDEC-Y2B8) Radioimmunotherapy for Treatment of Relapsed or Refractory CD20 Positive B-Cell Mon-Hodgkin's Lymphoma. Submitted 1999.

## Appendix I Common Toxicity Criteria (CTC)

## FINAL 1/30/98

CTC Version 2.0

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| ALLERGY/IMMUNOLOGY | | | | | |
| Allergic reaction/<br>hypersensitivity<br>(including drug<br>fever) | none | transient rash,<br>drug fever <<br>38°C (<100.4°F) | urticaria, drug<br>fever ≥ 38°C<br>(≥100.4°F),<br>and/or<br>asymptomatic<br>bronchospasm | symptomatic<br>bronchospasm,<br>requiring<br>parenteral<br>medication(s),<br>with or without<br>urticaria; allergy-<br>related<br>edema/angioede<br>ma | anaphylaxis |
| Note: Isolated urticaria DERMATOLOGY/SE | | of other manifestation | ns of an allergic or h | ypersensitivity reacti | on, is graded in the |
| Allergic rhinitis<br>(including sneezing,<br>nasal stuffiness,<br>postnasal drip) | none | mild, not<br>requiring<br>treatment | moderate,<br>requiring<br>treatment | - | - |
| Autoimmune reaction Also consider Hypothy | none yroidism, Colitis, | serologic or other evidence of autoimmune reaction but patient is asymptomatic (e.g., vitiligo), all organ function is normal and no treatment is required Hemoglobin, Hemoglobin, Hemoglobin, Hemoglobin, | evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism), requiring treatment other than immunosuppressi ve drugs | reversible autoimmune reaction involving function of a major organ or other toxicity (e.g., transient colitis or anemia), requiring short- term immunosuppressi ve treatment | autoimmune reaction causing major grade 4 organ dysfunction; progressive and irreversible reaction; long- term administration of high-dose immuno- suppressive therapy required |
| Serum sickness | none | - | - | present | - |
| Urticaria is graded in t<br>manifestations of aller | | | | olated symptom. If it | |
| Vasculitis | none | mild, not<br>requiring<br>treatment | symptomatic,<br>requiring<br>medication | requiring steroids | ischemic changes<br>or requiring<br>amputation |
| Allergy/Immunology -Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | | AUDITORY | //HEARING | | |
| Conductive hearing lo | | | the AUDITORY/HE | ARING category. | |
| Earache is graded in the External auditory canal Note: Changes associated as | normal | external otitis<br>with erythema or<br>dry desquamation | external otitis with moist desquamation nae) are graded unde | external otitis<br>with discharge,<br>mastoiditis<br>er Radiation dermatit | necrosis of the canal soft tissue or bone is in the |
| DERMATOLOGY/SE | | 1 . 1 | · · · · · | 4 | 11 4 1 |
| Inner ear/hearing | normal | hearing loss on<br>audiometry only | tinnitus or<br>hearing loss, not<br>requiring hearing<br>aid or treatment | tinnitus or hearing loss, correctable with hearing aid or treatment | or bilateral<br>hearing loss<br>(deafness), not<br>correctable |
| Middle ear/hearing | normal | serous otitis<br>without<br>subjective<br>decrease in<br>hearing | serous otitis or<br>infection<br>requiring medical<br>intervention;<br>subjective<br>decrease in<br>hearing; rupture<br>of tympanic<br>membrane with<br>discharge | otitis with<br>discharge,<br>mastoiditis or<br>conductive<br>hearing loss | necrosis of the<br>canal soft tissue<br>or bone |
| Auditory/Hearing-<br>Other<br>(Specify, | normal | mild | moderate | severe | life-threatening or<br>disabling |
| ) | | RLOOD/RON | NE MARROW | | |
| Bone marrow cellularity | normal for age | mildly<br>hypocellular or<br>25% reduction<br>from normal<br>cellularity for age | moderately hypocellular or >25 - \le 50\% reduction from normal cellularity for age or >2 but <4 weeks to recovery of normal bone marrow cellularity | severely hypocellular or >50 - ≤ 75% reduction in cellularity for age or 4 - 6 weeks to recovery of normal bone marrow cellularity | aplasia or >6<br>weeks to recovery<br>of normal bone<br>marrow<br>cellularity |
| Normal ranges:<br>children (≤ 18 years)<br>younger adults (19-<br>59)<br>older adults (≥ 60<br>years)<br>Note: Grade Bone man | 90% cellularity average 60-70% cellularity average 50% cellularity average | nly for changes relate | • | isease | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| CD4 count | WNL | < LLN -<br>500/mm <sup>3</sup> | $200 - < 500/\text{mm}^3$ | $\frac{3}{50 - < 200/\text{mm}^3}$ | < 50/mm <sup>3</sup> |
| Haptoglobin | normal | decreased | - | absent | - |
| Hemoglobin (Hgb) | WNL | < LLN - 10.0 g/dl | 8.0 - < 10.0 g/dl | 6.5 - < 8.0 g/dl | < 6.5 g/dl |
| | | < LLN - 100 g/L | 80 - 100 g/L | 65 - 80 g/L | < 65 g/L |
| | | < LLN - 6.2 | 4.9 - < 6.2 | 4.0 - < 4.9 | < 4.0 mmol/L |
| N | •. • | mmol/L | mmol/L | mmol/L | • |
| Note: The following criteria may be used for leukemia studies or bone marrow infiltrative/myelophthisic process if the | | | | | |
| protocol so specifies. | WAII | 10 <250/ | 25 <500/ | 50 <750/ | > 77.50/ 1 |
| For leukemia studies | WNL | 10 - <25% | 25 - <50% | 50 - <75% | ≥75% decrease |
| or bone marrow | | decrease from | decrease from | decrease from | from pretreatment |
| infiltrative/<br>myelophthisic | | pretreatment | pretreatment | pretreatment | |
| processes | | | | | |
| Hemolysis (e.g., | none | only laboratory | evidence of red | requiring | catastrophic |
| immune hemolytic | | evidence of | cell destruction | transfusion | consequences of |
| anemia, drug-related | | hemolysis [e.g., | and $\geq 2gm$ | and/or medical | hemolysis (e.g., |
| hemolysis, other) | | direct | decrease in | intervention (e.g., | renal failure, |
| • | | antiglobulin test | hemoglobin, no | steroids) | hypotension, |
| | | (DAT, Coombs') | transfusion | | bronchospasm, |
| | | schistocytes] | | | emergency |
| | | | | | splenectomy) |
| Also consider Haptogl | | .1111 20 109 | 20 20 109 | 10 20 109 | . 1 0 10 <sup>9</sup> /T |
| Leukocytes (total | WNL | < LLN - 3.0 x 10 <sup>9</sup><br>/L | $\geq 2.0 - < 3.0 \times 10^9$ /L | $\geq 1.0 - < 2.0 \times 10^9$ /L | $< 1.0 \times 10^9 / L$<br>$< 1000 / mm^3$ |
| WBC) | | /L<br>< LLN - | /L<br>≥2000 - < | | < 1000/mm |
| | | $\frac{2000}{\text{mm}^3}$ | $\frac{22000 - \sqrt{3000/mm^3}}{3000/mm^3}$ | $\geq 1000 - < 2000/\text{mm}^3$ | |
| For BMT studies: | WNL | $\geq 2.0 - < 3.0 \text{ X}$ | $\geq 1.0 - < 2.0 \times 10^9$ | $\geq 0.5 - < 1.0 \times 10^9$ | $< 0.5 \times 10^9 / L$ |
| TOT BIVIT Studies. | VI 12 | $\frac{22.0}{10^9/L}$ | /L≥1000 - | /L ≥500 - | <500/mm <sup>3</sup> |
| | | ≥2000 - | $< 2000/\text{mm}^3$ | $<1000/\text{mm}^3$ | |
| | | $<3000/\text{mm}^3$ | | | |
| Note: The following criteria using age, race and sex normal values may be used for pediatric studies if the protocol so | | | | | |
| specifies. | | | | | |
| | | ≥75 - <100%<br>LLN | ≥50 - <75% LLN | ≥25 - 50% LLN | <25% LLN |
| Lymphopenia | WNL | $<$ LLN - 1.0 x 10 $^{9}$ | $\geq 0.5 - < 1.0 \times 10^9$ | $<0.5 \times 10^9 / L$ | - |
| | | /L | /L | $< 500 / \text{mm}^3$ | |
| | | <lln -<="" td=""><td>≥500 -</td><td></td><td></td></lln> | ≥500 - | | |
| | | 1000/mm <sup>3</sup> | <1000/mm <sup>3</sup> | | |
| Note: The following criteria using age, race, and sex normal values may be used for pediatric studies if the protocol so specifies. | | | | | |
| , | | ≥75-<100%LLN | ≥50-<75%LLN | ≥25-<50%LLN | <25%LLN |
| Neutrophils/granuloc ytes | WNL | ≥1.5 - <2.0 x 10 <sup>9</sup><br>/L | ≥1.0 - <1.5 x 10 <sup>9</sup><br>/L | ≥0.5 - <1.0 x 10 <sup>9</sup><br>/L | $< 0.5 \times 10^9 / L$<br>$< 500 / mm^3$ |
| (ANC/AGC) | | ≥1500 - | ≥1000 - | ≥500 - | |
| , | | $< 2000 / \text{mm}^3$ | $<1500/\text{mm}^3$ | $<1000/\text{mm}^{3}$ | |
| For BMT: | WNL | $\geq 1.0 - < 1.5 \times 10^9$ | $\geq 0.5 - < 1.0 \times 10^9$ | $\geq 0.1 - < 0.5 \times 10^9$ | $<0.1 \times 10^{9} / L$ |
| | | /L | /L | /L | $<100/\text{mm}^{3}$ |
| | | ≥1000 - | ≥500 - | $\geq 100 - <500/\text{mm}^3$ | |
| | | <1500/mm <sup>3</sup> | $<1000/\text{mm}^3$ | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Note: The following criteria may be used for leukemia studies or bone marrow infiltrative/myelophthisic process if the protocol so specifies. | | | | | |
| For leukemia studies<br>or bone marrow<br>infiltrative/<br>myelophthisic<br>process | WNL | 10 - <25%<br>decrease from<br>baseline | 25 - <50%<br>decrease from<br>baseline | 50 - <75%<br>decrease from<br>baseline | ≥75% decrease from baseline |
| Platelets | WNL | < LLN - <75.0 x<br>10 <sup>9</sup> /L<br>< LLN -<br>75000/mm <sup>3</sup> | ≥50.0 - < 75.0 x<br>10 <sup>9</sup> /L<br>≥50000 - <<br>75000/mm <sup>3</sup> | $\geq 10.0 - < 50.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 10000 - <$<br>$50000 / \text{mm}^3$ | < 10.0 x 10 <sup>9</sup> /L<br>< 10000/mm <sup>3</sup> |
| For BMT: | WNL | $\geq 50.0 - <75.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 50000 - <75000 / \text{mm}^3$ | $\geq 20.0 - <50.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 20000 - <50000 / \text{mm}^3$ | $\geq 10.0 - <20.0 \text{ x}$<br>$10^9 / \text{L}$<br>$\geq 10000 - <20000 / \text{mm}^3$ | <10.0 x 10 <sup>9</sup> /L<br><10000/mm <sup>3</sup> |
| Note: The following cr<br>protocol so specifies. | riteria may be use | ed for leukemia studi | ies or bone marrow i | nfiltrative/myelophtl | nisic process if the |
| For leukemia studies or bone marrow infiltrative/ myelophthisic process | WNL | 10 - <25%<br>decrease from<br>baseline | 25 - <50%<br>decrease from<br>baseline | 50 - <75%<br>decrease from<br>baseline | ≥75% decrease from baseline |
| Transfusion:<br>Platelets | none | | | yes | platelet transfusions and other measures required to improve platelet increment; platelet transfusion refractoriness associated with life-threatening bleeding. (e.g., HLA or cross matched platelet transfusions) |

| Grade | | | | | | | |
|---|---|---|---|---|---|--|--|
| Toxicity | 0 | 1 | 2 | 3 | 4 | | |
| For BMT: | none | 1 platelet<br>transfusion in 24<br>hours | 2 platelet<br>transfusions in 24<br>hours | ≥3 platelet transfusions in 24 hours | platelet transfusions and other measures required to improve platelet increment; platelet transfusion refractoriness associated with life-threatening bleeding. (e.g., HLA or cross matched platelet transfusions) | | |
| Also consider Platelet | | | | | | | |
| Transfusion: pRBCs | none | - | - DDG ( 11 | Yes | - | | |
| For BMT: | none | ≤2 u pRBC<br>(≤15cc/kg) in 24<br>hours elective or<br>planned | 3 u pRBC (>15<br>≤30cc/kg) in 24<br>hours elective or<br>planned | $\geq$ 4 u pRBC ( $>30cc/kg$ ) in 24 hours | hemorrhage or<br>hemolysis<br>associated with<br>life-threatening<br>anemia; medical<br>intervention<br>required to<br>improve<br>hemoglobin | | |
| Also consider Hemog | lobin. | | | | | | |
| Blood/Bone<br>Marrow-Other<br>(Specify, | none | mild | moderate | severe | life-threatening or<br>disabling | | |
| | ( | CARDIOVASCULA | AR (ARRHYTHMIA | <b>A</b> ) | | | |
| Conduction<br>abnormality/<br>Atrioventricular<br>heart block | none | asymptomatic,<br>not requiring<br>treatment (e.g.,<br>Mobitz type I<br>second-degree<br>AV block,<br>Wenckebach) | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment (e.g., Mobitz type II second-degree AV block, third-degree AV block) | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | |
| Nodal/junctional<br>arrhythmia/dysrhyth<br>mia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | |
| Palpitations Note: Grade palpitation | none | present sence of a documente | -<br>ed arrhythmia | - | - | | |
| | Grade | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| Toxicity | 0 | 1 | 2 | 3 | 4 | | | | |
| Prolonged QTc<br>interval (QTc > 0.48<br>seconds) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | | | |
| Sinus bradycardia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | | | |
| Sinus tachycardia | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and<br>requiring<br>treatment of<br>underlying cause | - | | | | |
| Supraventricular<br>arrhythmias<br>(SVT/atrial<br>fibrillation/ flutter) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | | | |
| Syncope (fainting) is g | graded in the NEU | JROLOGY category | | | | | | | |
| Vasovagal episode | none | - | present without loss of consciousness | present with loss<br>of consciousness | - | | | | |
| Ventricular<br>arrhythmia<br>(PVCs/bigeminy/trig<br>eminy/<br>ventricular<br>tachycardia) | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic and requiring treatment | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | | | |
| Cardiovascular/ Arrhythmia-Other (Specify, | none | asymptomatic,<br>not requiring<br>treatment | symptomatic, but<br>not requiring<br>treatment | symptomatic, and<br>requiring<br>treatment of<br>underlying cause | life-threatening<br>(e.g., arrhythmia<br>associated with<br>CHF,<br>hypotension,<br>syncope, shock) | | | | |
| | | CARDIOVASCU | LAR (GENERAL) | | | | | | |
| Acute vascular leak syndrome | absent | - | symptomatic, but<br>not requiring<br>fluid support | respiratory<br>compromise or<br>requiring fluids | life-threatening;<br>requiring pressor<br>support and/or<br>ventilatory<br>support | | | | |
| Cardiac-<br>ischemia/infarction | none | non-specific T-<br>wave flattening<br>or changes | asymptomatic,<br>ST- and T- wave<br>changes<br>suggesting<br>ischemia | angina without<br>evidence of<br>infarction | acute myocardial infarction | | | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Cardiac left<br>ventricular function | normal | asymptomatic decline of resting ejection fraction of $\geq 10\%$ but $< 20\%$ of baseline value; shortening fraction $\geq 24\%$ but $< 30\%$ | asymptomatic but resting ejection fraction below LLN for laboratory or decline of resting ejection fraction ≥ 20% of baseline value; < 24% shortening fraction | CHF responsive to treatment | severe or<br>refractory CHF or<br>requiring<br>intubation |
| CNS cerebrovascular | ischemia is grade | ed in the NEUROLO | | | |
| Cardiac troponin I (cTnI) | normal | - | - | levels consistent<br>with unstable<br>angina as defined<br>by the<br>manufacturer | levels consistent<br>with myocardial<br>infarction as<br>defined by the<br>manufacturer |
| Cardiac troponin T (cTnT) | normal | $\geq 0.03 - < 0.05$ ng/ml | $\geq 0.05 - < 0.1$ ng/ml | $\geq 0.1 - < 0.2$ ng/ml | $\geq 0.2 \text{ ng/ml}$ |
| Edema | none | asymptomatic,<br>not requiring<br>therapy | symptomatic, requiring therapy | symptomatic<br>edema limiting<br>function and<br>unresponsive to<br>therapy or<br>requiring drug<br>discontinuation | anasarca (severe<br>generalized<br>edema) |
| Hypertension | none | asymptomatic,<br>transient increase<br>by >20 mmHg<br>(diastolic) or to ><br>150/100* if<br>previously WNL;<br>not requiring<br>treatment | recurrent or persistent or symptomatic increase by > 20 mmHg (diastolic) or to > 150/100* if previously WNL; not requiring treatment | requiring therapy<br>or more intensive<br>therapy than<br>previously | hypertensive<br>crisis |
| *Note: For pediatric | patients, use age | and sex appropriate | normal values > 95t | h percentile ULN. | |
| Hypotension | none | changes, but not<br>requiring therapy<br>(including<br>transient<br>orthostatic<br>hypotension) | requiring brief<br>fluid replacement<br>or other therapy<br>but not<br>hospitalization;<br>no physiologic<br>consequences | requiring therapy<br>and sustained<br>medical attention,<br>but resolves<br>without persisting<br>physiologic<br>consequences | shock (associated<br>with acidemia<br>and impairing<br>vital organ<br>function due to<br>tissue<br>hypoperfusion) |
| For pediatric patient. | I is graded as Car<br>s, systolic BP 65 i | | its up to 1 year old a | | |
| than 1 year of age, us<br>Myocarditis | none | or inree measuremen<br>- | | CHF responsive to treatment | severe or<br>refractory CHF |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Operative injury of vein/artery | none | primary suture<br>repair for injury,<br>but not requiring<br>transfusion | primary suture<br>repair for injury,<br>requiring<br>transfusion | vascular<br>occlusion<br>requiring surgery<br>or bypass for<br>injury | myocardial<br>infarction;<br>resection of organ<br>(e.g., bowel,<br>limb) |
| Pericardial effusion/<br>pericarditis | none | asymptomatic<br>effusion, not<br>requiring<br>treatment | pericarditis (rub,<br>ECG changes,<br>and/or chest pain) | physiologic<br>consequences<br>resulting from<br>symptoms | tamponade<br>(drainage or<br>pericardial<br>window required |
| Peripheral arterial ischemia | none | - | brief episode of ischemia managed non-surgically and without permanent deficit | requiring surgical intervention | life-threatening of<br>with permanent<br>functional deficit<br>(e.g., amputation |
| | | -<br>ed in the DERMATOI | | | - |
| | | in the CARDIOVASO | | ) category. | |
| Syncope (fainting) is g | | EUROLOGY category | | doon visin | ambalia at |
| Thrombosis/embolis m | none | - | deep vein<br>thrombosis, not<br>requiring<br>anticoagulant | deep vein<br>thrombosis,<br>requiring<br>anticoagulant<br>therapy | embolic event<br>including<br>pulmonary<br>embolism |
| Vein/artery operative is category. | injury is graded | as Operative injury of | f vein/artery in the CA | | (GENERAL) |
| Visceral arterial ischemia (non-myocardial) | none | - | brief episode of ischemia managed non-surgically and without permanent deficit | requiring surgical intervention | life-threatening of<br>with permanent<br>functional deficit<br>(e.g., resection of<br>ileum) |
| Cardiovascular/<br>General-Other<br>(Specify, | none | mild | moderate | severe | life-threatening of disabling |
| · | | | JLATION | | |
| Note: See the HEMOI | | ory for grading the se | verity of bleeding eve | | |
| DIC<br>(disseminated<br>intravascular<br>coagulation)<br>Also grade Platelets.<br>Note: Must have incre | absent | products or D-dimer | in order to grade as F | laboratory<br>findings present<br>with <u>no</u> bleeding | laboratory<br>findings <u>and</u><br>bleeding |
| Fibrinogen | WNL | ≥0.75 - <1.0 x<br>LLN | | ≥0.25 - <0.5 x<br>LLN | <0.25 x LLN |
| Note: The following c protocol so specifies. | riteria may be u | | | | isic process if the |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| For leukemia studies: | WNL | <20% decrease<br>from pretreatment<br>value or LLN | ≥20 - <40%<br>decrease from<br>pretreatment<br>value or LLN | ≥40 - <70%<br>decrease from<br>pretreatment<br>value or LLN | <50 mg% |
| Partial thromboplastin time (PTT) | WNL | > ULN - ≤ 1.5 x<br>ULN | $> 1.5 - \le 2 x$ ULN | >2 x ULN | - |
| Phelbitis is graded in the | | SCULAR (GENERA | | | |
| Prothrombin time (PT) | WNL | $>$ ULN - $\leq$ 1.5 x ULN | $> 1.5 - \le 2 x$<br>ULN | >2 x ULN | - |
| Thrombosis/embolism | | CARDIOVASCULA | R (GENERAL) cate | | |
| Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura/TTP or hemolytic uremic syndrome/HUS) | absent | - | - | laboratory<br>findings present<br>without clinical<br>consequences | laboratory findings and clinical consequences, (e.g., CNS hemorrhage/ bleeding or thrombosis/ embolism or renal failure) requiring therapeutic intervention |
| For BMT: | - | evidence of RBC<br>destruction<br>(schistocytosis)<br>without clinical<br>consequences | evidence of RBC<br>destruction with<br>elevated<br>creatinine (≤3 x<br>ULN) | evidence of RBC<br>destruction with<br>creatinine (>3 x<br>ULN) not<br>requiring dialysis | evidence of RBC<br>destruction with<br>renal failure<br>requiring dialysis<br>and/or<br>encephalopathy |
| Also consider Hemogle | | | | | |
| Note: Must have micro | | | | | |
| Coagulation-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| , | | CONSTITUTION | NAL SYMPTOMS | | |
| Fatigue (lethargy, malaise, asthenia) | none | increased fatigue<br>over baseline, but<br>not altering<br>normal activities | moderate (e.g., decrease in performance status by 1 ECOG level or 20% Karnofsky or <i>Lansky</i> ) or causing difficulty performing some activities | severe (e.g., decrease in performance status by ≥2 ECOG levels or 40% Karnofsky or <i>Lansky</i> ) or loss of ability to perform some activities | bedridden or<br>disabling |
| Note: See Appendix IV | (nttp://ctep.info | nın.gov/ctc3/ctc.htn | n) for performance st | tatus scales. | |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Fever (in the absence | none | 38.0 - 39.0°C | 39.1 - 40.0°C | > 40.0°C | > 40.0°C |
| of neutropenia, | | (100.4 - 102.2°F) | (102.3 - 104.0°F | $(>104.0^{\circ}F)$ for $<$ | $(>104.0^{\circ}F)$ for $>$ |
| where neutropenia is | | | ) | 24hrs | 24hrs |
| defined as AGC < | | | | | |
| $1.0 \times 10^9/L$ ) | | | | | |
| Also consider Allergic | | | | | |
| Note: The temperature | | | | | |
| Hot flashes/flushes are | | | | · | |
| Rigors, chills | none | mild, requiring | severe and/or | not responsive to | - |
| | | symptomatic | prolonged, | narcotic | |
| | | treatment (e.g., | requiring narcotic | medication | |
| | | blanket) or non- | medication | | |
| | | narcotic | | | |
| G 4: | 1 | medication | <u> </u> | | |
| Sweating | normal | mild and | frequent or | - | - |
| (diaphoresis) | < 5% | occasional<br>5 - <10% | drenching<br>10 - <20% | > 200/ | |
| Weight gain Also consider Ascites, | | | 10 - <20% | ≥ 20% | - |
| Weight gain - veno- | Edema, Fleurar | errusion. | | | |
| occlusive disease | | | | | |
| (VOD) | | | | | |
| Note: The following c | riteria is to be use | ed ONLY for weight | gain associated with | Veno-Occlusive Dis | sease |
| rote. The following e | <2% | >2 - <5% | ≥5 - <10% | $\geq 10\%$ or as | ≥10% or fluid |
| | _, · | =2 370 | _5 1070 | ascities | retention |
| | | | | | resulting in |
| | | | | | pulmonary failure |
| Weight loss | < 5% | 5 - <10% | 10 - <20% | ≥20% | - |
| Also consider Vomitin | ng, Dehydration, | Diarrhea. | | | |
| Constitutional | none | mild | moderate | severe | life-threatening or |
| Symptoms-Other | | | | | disabling |
| (Specify, | | | | | |
| ) | | | | | |
| | | | LOGY/SKIN | | |
| Alopecia | normal | mild hair loss | pronounced hair | - | - |
| _ | | | Îoss | | |
| Bruising | none | localized or in | generalized | - | - |
| (in absence of grade | | dependent area | | | |
| 3 or 4 | | | | | |
| thrombocytopenia) | | | | | |
| | | 3 or 4 thrombocytope | | | |
| Hemorrhage/bleeding | | thrombocytopenia in | n the HEMORRHAC | 3E category, <u>not</u> in th | ne |
| DERMATOLOGY/SI | CIN category | | | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Dermatitis, focal<br>(associated with<br>high-dose<br>chemotherapy and<br>bone marrow<br>transplant) | none | faint erythema or<br>dry desquamation | moderate to brisk<br>erythema or a<br>patchy moist<br>desquamation,<br>mostly confined<br>to skin folds and<br>creases; moderate<br>edema | confluent moist desquamation, ≥1.5 cm diameter, not confined to skin folds; pitting edema | skin necrosis or<br>ulceration of full<br>thickness dermis;<br>may include<br>spontaneous<br>bleeding not<br>induced by minor<br>trauma or<br>abrasion |
| Dry skin | normal | controlled with emollients | not controlled with emollients | - | - |
| Erythema multiforme<br>(e.g., Stevens-<br>Johnson syndrome,<br>toxic epidermal<br>necrolysis) | absent | - | scattered, but not<br>generalized<br>eruption | severe or<br>requiring IV<br>fluids (e.g.,<br>generalized rash<br>or painful<br>stomatitis) | life-threatening<br>(e.g., exfoliative<br>or ulcerating<br>dermatitis or<br>requiring enteral<br>or parenteral<br>nutritional<br>support) |
| Flushing | absent | present | - | | - |
| Hand-foot skin reaction | none | skin changes or<br>dermatitis<br>without pain<br>(e.g., erythema,<br>peeling) | skin changes with<br>pain, not<br>interfering with<br>function | skin changes with<br>pain, interfering<br>with function | - |
| Injection site reaction | none | pain or itching or<br>erythema | pain or swelling,<br>with<br>inflammation or<br>phlebitis | ulceration or<br>necrosis that is<br>severe or<br>prolonged, or<br>requiring surgery | - |
| Nail changes | normal | discoloration or<br>ridging<br>(koilonychia) or<br>pitting | partial or<br>complete loss of<br>nail(s) or pain in<br>nailbeds | - | - |
| Petechiae is graded in t | the HEMORRHA | | | | |
| Photosensitivity | none | painless erythema | painful erythema | erythema with desquamation | - |
| Pigmentation changes (e.g., vitiligo) | none | localized pigmentation changes | generalized<br>pigmentation<br>changes | - | - |
| Pruritus Purpura is graded in th | none | mild or localized, relieved spontaneously or by local measures | intense or<br>widespread,<br>relieved<br>spontaneously or<br>by systemic<br>measures | intense or<br>widespread and<br>poorly controlled<br>despite treatment | - |

| one | 1 | | | |
|---|---|---|---|---|
| one | 1 | 2 | 3 | 4 |
| | faint erythema or<br>dry desquamation | moderate to brisk<br>erythema or a<br>patchy moist<br>desquamation,<br>mostly confined<br>to skin folds and<br>creases; moderate<br>edema | confluent moist<br>desquamation,<br>≥1.5 cm<br>diameter, not<br>confined to skin<br>folds; pitting<br>edema | skin necrosis or<br>ulceration of full<br>thickness dermis;<br>may include<br>bleeding not<br>induced by minor<br>trauma or<br>abrasion |
| | dry desquamation | erythema or a<br>patchy moist<br>desquamation,<br>mostly confined<br>to skin folds and<br>creases; moderate<br>edema | desquamation,<br>≥1.5 cm<br>diameter, not<br>confined to skin<br>folds; pitting<br>edema | skin necrosis or<br>ulceration of full<br>thickness dermis;<br>may include<br>bleeding not<br>induced by minor<br>trauma or<br>abrasion |
| | papular eruption<br>or erythema<br>without<br>associated | macular or papular eruption or erythema with pruritis or other associated symptoms covering <50% of body surface or localized desquamation or other lesions covering <50% of body surface area | symptomatic generalized erythroderma or macular, papular or vesicular eruption or desquamation covering ≥50% of body surface area | generalized<br>exfoliative<br>dermatitis or<br>ulcerative<br>dermatitis |
| | papular eruption<br>or erythema<br>covering <25%<br>of body surface<br>area without<br>associated | macular or papular eruption or erythema with pruritis or other associated symptoms covering ≥25 - <50% of body surface or localized desquamation or other lesions covering ≥25 - <50% of body surface area | symptomatic generalized erythroderma or symptomatic macular, papular or vesicular eruption, with bullous formation, or desquamation covering ≥50% of body surface area | generalized<br>exfoliative<br>dermatitis or<br>ulcerative<br>dermatitis or<br>bullous formation |
| | one one action/hypersen | one faint erythema or dry desquamation macular or papular eruption or erythema without associated symptoms macular or papular eruption or erythema covering <25% of body surface area without associated symptoms metion/hypersensitivity. | to skin folds and creases; moderate edema n radiation dermatitis is graded separately in the PAIN of the patch of the pa | to skin folds and creases; moderate edema n radiation dermatitis is graded separately in the PAIN category as Pain due of the patch moist desquamation, mostly confined to skin folds and creases; moderate edema one macular or papular eruption or erythema without associated symptoms symptoms one macular or papular eruption or erythema without associated symptoms one macular or papular eruption or erythema without associated symptoms one macular or papular eruption or body surface or localized desquamation or or erythema covering <25% of body surface area without associated symptoms of body surface area without associated symptoms of body surface area without associated symptoms of body surface area without associated symptoms of body surface area without associated covering ≥25 - \$50% of body surface area one macular or papular eruption or erythema with pruritis or other associated symptoms of body surface area without associated covering ≥25 - \$50% of body surface area one macular or papular eruption or erythema with pruritis or other elsions covering ≥25 - \$50% of body surface area one macular or papular eruption or erythema with pruritis or other elsions covering ≥25 - \$50% of body surface area one macular or papular eruption or erythema with pruritis or other elsions covering ≥25 - \$50% of body surface area one macular or papular eruption or erythema with pruritis or other elsions covering ≥25 - \$50% of body surface area one macular or papular eruption or erythema with pruritis or other elsions covering ≥25 - \$50% of body surface area |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Urticaria<br>(hives, welts,<br>wheals) | none | requiring no<br>medication | requiring PO or<br>topical treatment<br>or IV medication<br>or steroids for<br><24 hours | requiring IV<br>medication or<br>steroids for ≥24<br>hours | - |
| Wound- infectious | none | cellulitis | superficial infection | infection<br>requiring IV<br>antibiotics | necrotizing fascitis |
| Wound- non-<br>infectious | none | incisional<br>separation | incisional hernia | fascial disruption without evisceration | fascial disruption with evisceration |
| Dermatology/Skin-<br>Other<br>(Specify, ) | none | mild | moderate | severe | life-threatening or disabling |
| | | ENDO | CRINE | | |
| Cushingoid appearance (e.g., moon face with or without buffalo hump, centripetal obesity, cutaneous striae) Also consider Hypergl | absent | - | present | - | - |
| Feminization of male | absent | - | _ | present | _ |
| Gynecomastia | none | mild | pronounced or<br>painful | pronounced or<br>painful and<br>requiring surgery | - |
| Hot flashes/flushes | none | mild or no more<br>than 1 per day | moderate and<br>greater than 1 per<br>day | - | - |
| Hypothyroidism | absent | asymptomatic,TS<br>H elevated, no<br>therapy given | symptomatic or<br>thyroid<br>replacement<br>treatment given | patient<br>hospitalized for<br>manifestations of<br>hypothyroidism | myxedema coma |
| Masculinization of female | absent | - | - | present | - |
| SIADH (syndrome<br>of inappropriate<br>antidiuretic<br>hormone) | absent | - | - | present | - |
| Endocrine-Other (Specify, | none | mild | moderate | severe | life-threatening or<br>disabling |
| | | GASTROIN | NTESTINAL | | |
| Amylase is graded in t | he METABOI | LIC/LABORATORY c | | | |
| Anorexia | none | loss of appetite | oral intake<br>significantly<br>decreased | requiring IV<br>fluids | requiring feeding<br>tube or parenteral<br>nutrition |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Ascites (non-malignant) | none | asymptomatic | symptomatic,<br>requiring<br>diuretics | symptomatic,<br>requiring<br>therapeutic<br>paracentesis | life-threatening<br>physiologic<br>consequences |
| Colitis | none | - | abdominal pain<br>with mucus<br>and/or blood in<br>stool | abdominal pain,<br>fever, change in<br>bowel habits with<br>ileus or peritoneal<br>signs, and<br>radiographic or<br>biopsy<br>documentation | perforation or<br>requiring surgery<br>or toxic<br>megacolon |
| | | g with grade 3 or 4 throm ding, Rectal bleeding/her | | | out grade 3 or 4 |
| Constipation | none | requiring stool<br>softener or<br>dietary<br>modification | requiring<br>laxatives | obstipation<br>requiring manual<br>evacuation or<br>enema | obstruction or toxic megacolon |
| Dehydration | none | dry mucous<br>membranes<br>and/or<br>diminished skin<br>turgor | requiring IV fluid<br>replacement<br>(brief) | requiring IV fluid<br>replacement<br>(sustained) | physiologic<br>consequences<br>requiring<br>intensive care;<br>hemodynamic<br>collapse |
| | ension, Diarrh | ea, Vomiting, Stomatitis/ | | ryngeal mucositis). | |
| Diarrhea<br>Patients without<br>colostomy: | none | increase of < 4<br>stools/day over<br>pre-treatment | increase of 4-6<br>stools/day, or<br>nocturnal stools | increase of ≥7<br>stools/day or<br>incontinence; or<br>need for<br>parenteral<br>support for<br>dehydration | physiologic<br>consequences<br>requiring<br>intensive care; or<br>hemodynamic<br>collapse |
| Patients with a colostomy: | none | mild increase in<br>loose, watery<br>colostomy output<br>compared with<br>pretreatment | moderate increase<br>in loose, watery<br>colostomy output<br>compared with<br>pretreatment, but<br>not interfering<br>with normal<br>activity | severe increase in<br>loose, watery<br>colostomy output<br>compared with<br>pretreatment,<br>interfering with<br>normal activity | physiologic<br>consequences,<br>requiring<br>intensive care; or<br>hemodynamic<br>collapse |
| For BMT | none | >500 - ≤1000ml<br>of diarrhea/day | >1000 - ≤1500ml<br>of diarrhea/day | >1500ml of diarrhea/day | severe abdominal<br>pain with or<br>without ileus |
| For Pediatric BMT: | | >5 - 10 ml/kg of diarrhea/day | of diarrhea/day | >15 ml/kg of<br>diarrhea/day | - |
| Also consider Hemor<br>thrombocytopenia, P | | g with grade 3 or 4 throm on, Hypotension. | nbocytopenia, Hemor | rhage/bleeding with | out grade 3 or 4 |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Duodenal ulcer<br>(requires<br>radiographic or<br>endoscopic<br>documentation) | none | - | requiring medical<br>management or<br>non-surgical<br>treatment | uncontrolled by outpatient medical management; requiring hospitalization | perforation or<br>bleeding,<br>requiring<br>emergency<br>surgery |
| Dyspepsia/heartburn | none | mild | moderate | severe | - |
| Dysphagia, esophagitis, odynophagia (painful swallowing) Note: If toxicity is rad pharyngeal related to response to the same and the s | adiation. | | | | |
| Dysphagia- esophageal related to radiation Also consider Pain due | | | dysphagia, requiring predominantly liquid, pureed or soft diet | dysphagia<br>requiring feeding<br>tube, IV<br>hydration or<br>hyperalimentatio<br>n | complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation |
| Note: Fistula is graded | | | 1 1 . | 1 1 . | 1 . |
| Dysphagia - pharyngeal related to radiation | none | mild dysphagia,<br>but can eat<br>regular diet | dysphagia,<br>requiring<br>predominantly<br>pureed, soft, or<br>liquid diet | dysphagia,<br>requiring feeding<br>tube, IV<br>hydration or<br>hyperalimentatio<br>n | complete obstruction (cannot swallow saliva); ulceration with bleeding not induced by minor trauma or abrasion or perforation |
| Also consider Pain due<br>Note: Fistula is graded | | | ion. | | |
| Fistula- esophageal | none | - | - | present | requiring surgery |
| Fistula- intestinal | none | | | present | requiring surgery |
| Fistula- pharyngeal | none | - | - | present | requiring surgery |
| Fistula- rectal/anal | none | - | - | present | requiring surgery |
| Flatulence | none | mild | moderate | - | - |

| | | G | rade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Gastric ulcer (requires radiographic or endoscopic documentation) | none | - | requiring medical<br>management or<br>non-surgical<br>treatment | bleeding without<br>perforation,<br>uncontrolled by<br>outpatient<br>medical<br>management;<br>requiring<br>hospitalization or | perforation or<br>bleeding,<br>requiring<br>emergency<br>surgery |
| Also consider Hemori<br>thrombocytopenia. | hage/bleeding w | rith grade 3 or 4 throi | mbocytopenia, Hemor | surgery<br>rhage/bleeding with | out grade 3 or 4 |
| Gastritis | none | - | requiring medical<br>management or<br>non-surgical<br>treatment | uncontrolled by<br>out-patient<br>medical<br>management;<br>requiring<br>hospitalization or<br>surgery | life-threatening<br>bleeding,<br>requiring<br>emergency<br>surgery |
| Also consider Hemori<br>thrombocytopenia.<br>Hematemesis is grade | | | nbocytopenia, Hemor | rhage/bleeding with | out grade 3 or 4 |
| Hematochezia is grade | | | s Rectal bleeding/her | natochezia. | |
| Ileus (or neuroconstipation) | none | - | intermittent, not requiring intervention | requiring non-<br>surgical<br>intervention | requiring surger |
| Mouth dryness | normal | mild | moderate | - | - |
| Mucositis Note: Mucositis not Esophagitis, Gastritis, RENAL/GENITOUR Radiation-related muc Mucositis due to radiation | Stomatitis/phary INARY category cositis is graded a none | yngitis (oral/pharynge<br>y for Vaginititis.<br>as Mucositis due to ra<br>erythema of the<br>mucosa | eal mucositis), and Ty | | necrosis or deep<br>ulceration; may<br>include bleeding<br>not induced by<br>minor trauma or<br>abrasion |
| Note: Grade radiation Dysphagia related to a pharyngeal related to | | graded as <u>either</u> Dysp | | ated to radiation <u>or</u> I | Dysphagia- |
| Nausea | none | able to eat | oral intake<br>significantly<br>decreased | no significant intake, requiring IV fluids | - |
| Pancreatitis | none | - | - | abdominal pain<br>with pancreatic<br>enzyme elevation | complicated by shock (acute circulatory |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Note: Asymptomatic a | | | | | |
| Pharyngitis is graded in the GASTROINTESTINAL category as Stomatitis/pharyngitis (oral/pharyngeal mucositis). | | | | | |
| Proctitis | none | increased stool<br>frequency,<br>occasional blood-<br>streaked stools, or<br>rectal discomfort<br>(including<br>hemorrhoids), not<br>requiring<br>medication | increased stool<br>frequency,<br>bleeding, mucus<br>discharge, or<br>rectal discomfort<br>requiring<br>medication; anal<br>fissure | increased stool<br>frequency/diarrhe<br>a, requiring<br>parenteral<br>support; rectal<br>bleeding,<br>requiring<br>transfusion; or<br>persistent mucus<br>discharge,<br>necessitating<br>pads | perforation,<br>bleeding or<br>necrosis or other<br>life-threatening<br>complication<br>requiring surgical<br>intervention (e.g.,<br>colostomy) |
| Also consider Hemorr<br>thrombocytopenia, and<br>Note: Fistula is grad<br>Proctitis occurring mo<br>Morbidity Scoring Sch | d Pain due to radied separately as I re than 90 days at | ation.<br>Fistula- rectal/anal.<br>fter the start of radiat<br>adix V, http://ctep.inf | ion therapy is grader<br>fo.nih.gov/ctc3/ctc.h | d in the RTOG/EOR' | TC Late Radiation |
| Salivary gland | none | slightly thickened | thick, ropy, sticky | - | acute salivary |
| changes | | saliva/may have<br>slightly altered<br>taste (e.g.,<br>metallic);<br>additional fluids<br>may be required | saliva; markedly<br>altered taste;<br>alteration in diet<br>required | | gland necrosis |
| Sense of smell | normal | slightly altered | markedly altered | - | - |
| Stomatitis/pharyngiti<br>s (oral/pharyngeal<br>mucositis) | none | painless ulcers,<br>erythema, or mild<br>soreness in the<br>absence of<br>lesions | painful erythema,<br>edema, or ulcers,<br>but can eat or<br>swallow | painful erythema,<br>edema, or ulcers<br>requiring IV<br>hydration | severe ulceration<br>or requires<br>parenteral or<br>enteral nutritional<br>support or<br>prophylatic<br>intubation |
| For BMT: | none | painless ulcers,<br>erythema, or mild<br>soreness in the<br>absence of<br>lesions | painful erythema,<br>edema or ulcers<br>but can swallow | painful erythema,<br>edema, or ulcers<br>preventing<br>swallowing or<br>requiring<br>hydration or<br>parenteral (or<br>enteral)<br>nutritional<br>support | severe ulceration<br>requiring<br>prophylactic<br>intubation or<br>resulting in<br>documented<br>aspiration<br>pneumonia |
| Note: Radiation-relate | d mucositis is gra | ded as Mucositis due | e to radiation. | , , | |
| Taste disturbance (dysgeusia) | normal | slightly altered | markedly altered | - | _ |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Typhlitis (inflammation of the cecum) | none | - | - | abdominal pain,<br>diarrhea, fever, or<br>radiographic<br>documentation | perforation,<br>bleeding or<br>necrosis or other<br>life-threatening<br>complication<br>requiring surgical<br>intervention (e.g.,<br>colostomy) |
| Also consider Hemorri<br>thrombocytopenia, Hy | | | nbocytopenia, Hemor | rhage/bleeding with | |
| Vomiting | none | 1 episode in 24<br>hours over<br>pretreatment | 2-5 episodes in<br>24 hours over<br>pretreatment | ≥6 episodes in 24 hours over pretreatment; or need for IV fluids | Requiring parenteral nutrition; or physiologic consequences requiring intensive care; hemodynamic collapse |
| Also consider Dehydra Weight gain is graded | | HITIONIAI CVMDT | OMS antagory | | |
| Weight loss is graded | | | | | |
| Gastrointestinal-<br>Other<br>(Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | НЕМОБ | RRHAGE | | |

Note: Transfusion in this section refers to pRBC infusion.

For <u>any</u> bleeding with grade 3 or 4 platelets (< 50,000), <u>always</u> grade Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia. Also consider platelets, transfusion-pRBCS, and transfusion-platelets in addition to the grade that incorporates the site or type of bleeding.

If the site or type of hemorrhage/bleeding is listed, also use the grading that incorporates the site of bleeding: CNS hemorrhage/bleeding, Hematuria, Hematemesis, Hemoptysis, Hemorrhage/bleeding with surgery, Melena/lower GI bleeding, Petechiae/purpura (Hemorrhage/bleeding into skin), Rectal bleeding/hematochezia, Vaginal bleeding. If the platelet count is  $\geq 50,000$  and the site or type of bleeding is listed, grade the specific site. If the site or type is not listed and the platelet count is  $\geq 50,000$ , grade Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia and specify the site or type in the OTHER category.

| Hemorrhage/ble none mild without requiring catastrophic eding with transfusion transfusion bleeding, grade 3 or 4 requiring thrombocytopen ia elective intervention | | | | |
|---|---|---|---|---|
| | eding with grade 3 or 4 thrombocytopen | none | 1 0 | bleeding,<br>requiring<br>major non-<br>elective |

Also consider Platelets, Hemoglobin, Transfusion-platelet, Transfusion-pRBCs.

Note: This toxicity must be graded for any bleeding with grade 3 or 4 thrombocytopenia. Also grade the site or type of hemorrhage/bleeding. If the site is not listed, grade as Other in the HEMORRHAGE category.

| | | Grad | e | | |
|---|---|---|---|---|---|
| Toxicity | 0 1 | 2 | 3 | 4 | |
| Hemorrhage/ble eding without grade 3 or 4 thrombocytopen ia Also consider Platelets, Note: Bleeding in th | e absence of grade 3 | or 4 thrombocytope | sfusion-pRBCs.<br>enia is graded here or<br>ategory. Also grade a | | |
| CNS<br>hemorrhage/ble<br>eding | none | - | - | bleeding<br>noted on CT<br>or other scan<br>with no<br>clinical<br>consequence<br>s | hemorrhagic<br>stroke or<br>hemorrhagic<br>vascular<br>event<br>(CVA) with<br>neurologic<br>signs and<br>symptoms |
| Epistaxis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hematemesis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hematuria<br>(in the absence<br>of vaginal<br>bleeding) | none | microscopic<br>only | intermittent<br>gross<br>bleeding, no<br>clots | persistent gross bleeding or clots; may require catheterizati on or instrumentat ion, or transfusion | open surgery<br>or necrosis<br>or deep<br>bladder<br>ulceration |
| Hemoptysis | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |

| | | Grad | de | | |
|---|---|---|---|---|---|
| oxicity | 0 | 1 | 2 | 3 | 4 |
| Hemorrhage/ble eding associated with surgery | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Melena/GI | none none | e of surgery is not grant mild without | raded as a toxicity. | requiring | catastrophic |
| bleeding | none | transfusion | | transfusion | bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Petechiae/purpu | none | rare | petechiae or | generalized | - |
| ra<br>(hemorrhage/bl<br>eeding into skin<br>or mucosa) | | petechiae of<br>skin | purpura in<br>dependent<br>areas of skin | petechiae or<br>purpura of<br>skin or<br>petechiae of<br>any mucosal<br>site | |
| Rectal bleeding/<br>hematochezia | none | mild without<br>transfusion<br>or<br>medication | persistent, requiring medication (e.g., steroid suppositorie s) and/or break from radiation treatment | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Vaginal<br>bleeding | none | spotting,<br>requiring <<br>2 pads per<br>day | requiring ≥ 2 pads per day, but not requiring transfusion | requiring<br>transfusion | catastrophi<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| Hemorrhage-Other (Specify site, | none | mild without<br>transfusion | - | requiring<br>transfusion | catastrophic<br>bleeding,<br>requiring<br>major non-<br>elective<br>intervention |
| | | HEPA | TIC | | |
| Alkaline<br>phosphatase | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5.0 x<br>ULN | > 5.0 - 20.0<br>x ULN | > 20.0 x<br>ULN |
| Bilirubin | WNL | > ULN - 1.5<br>x ULN | > 1.5 - 3.0 x<br>ULN | > 3.0 - 10.0<br>x ULN | > 10.0 x<br>ULN |
| | ersus host disease ( | | | | |
| Note: The follow | | | | versus host disease. | . 1.5 |
| | normal | $\ge 2 - < 3$ mg/100 ml | $\geq 3 - < 6$ mg/100 ml | $\geq 6 - <15$ mg/100 ml | ≥15 mg/10<br>ml |

| | | Grad | le | | |
|---|---|---|---|---|---|
| Toxicity | <b>0</b> 1 | 1 2 | 2 3 | 3 | 4 |
| GGT | WNL | > ULN - 2.5 | > 2.5 - 5.0 x | > 5.0 - 20.0 | > 20.0 x |
| (γ - Glutamyl | | x ULN | ULN | x ULN | ULN |
| transpeptidase) | | | | | |
| Hepatic | absent | - | - | present | - |
| enlargement | atia anlargament an | ly for abangas relata | d to VOD or other tr | antmant related toxic | siter |
| Hypoalbumine | WNL | LLN - 3 | $\frac{d \text{ to VOD or other tr}}{\geq 2 - \langle 3 \text{ g/dl}}$ | <2 g/dl | ity. |
| mia | WINL | g/dl | ≥2 - \3 g/u1 | \2 g/u1 | _ |
| Liver | normal | - | - | asterixis | encephalopa |
| dysfunction/fail | | | | | thy or coma |
| ure (clinical) | | | | | J |
| | ed viral hepatitis is g | graded in the INFEC | TION category. | | |
| Portal vein flow | normal | - | decreased | reversal/retr | - |
| | | | portal vein | ograde | |
| | | | flow | portal vein | |
| CCOT (ACT) | WNL | > ULN - 2.5 | > 2.5 - 5.0 x | flow > 5.0 - 20.0 | > 20.0 |
| SGOT (AST)<br>(serum glutamic | WINL | > ULN - 2.5<br>x ULN | > 2.5 - 5.0 x<br>ULN | > 5.0 - 20.0<br>x ULN | > 20.0 x<br>ULN |
| oxaloacetic | | A OLIV | OLIV | A OLIV | OLIV |
| transaminase) | | | | | |
| SGPT (ALT) | WNL | > ULN - 2.5 | > 2.5 - 5.0 x | > 5.0 - 20.0 | > 20.0 x |
| (serum glutamic | | x ULN | ULN | x ULN | ULN |
| pyruvic | | | | | |
| transaminase) | | | | | |
| Hepatic-Other | none | mild | moderate | severe | life- |
| (Specify, | | | | | threatening |
| ) | | | | | or disabling |
| | INF | | E NEUTROPENIA | | |
| Catheter-related | none | mild, no | moderate, | severe, | life- |
| infection | | active | localized | systemic | threatening |
| | | treatment | infection, | infection, | sepsis (e.g., |
| | | | requiring<br>local or oral | requiring IV<br>antibiotic or | septic<br>shock) |
| | | | treatment | antifungal | SHOCK) |
| | | | treatment | treatment or | |
| | | | | hospitalizati | |
| | | | | on | |
| Febrile | none | - | - | Present | Life- |
| neutropenia | | | | | threatening |
| (fever of | | | | | sepsis (e.g., |
| unknown origin | | | | | septic |
| without<br>clinically or | | | | | shock) |
| microbiological | | | | | |
| ly documented | | | | | |
| infection) | | | | | |
| (ANC < 1.0 x) | | | | | |
| 10 <sup>9</sup> /L, fever | | | | | |
| ≥38.5°C) | | | | | |
| Note: Hypotherm | nia instead of fever i | nay be associated wi | th neutropenia and is | s graded here. | |

| | | Grad | le | | |
|---|---|---|---|---|---|
| Гохісіty | 0 | 1 2 | 2 3 | 3 | |
| Infection (documented clinically or microbiological ly) with grade 3 or 4 neutropenia (ANC < 1.0 x | none | - | - | present | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| | | may be associated with i | | | sence of |
| | | e 3 or 4 neutropenia, grad | le as Febrile neutrope | | 1: 0 |
| Infection with unknown ANC | none | - | - | present | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| | ty criterion is u | sed in the rare case when | | | |
| Infection<br>without<br>neutropenia | none | mild, no<br>active<br>treatment | moderate,<br>localized<br>infection,<br>requiring<br>local or oral<br>treatment | severe, systemic infection, requiring IV antibiotic or antifungal treatment, or hospitalizati on | life-<br>threatening<br>sepsis (e.g.,<br>septic<br>shock) |
| Infection/Febril e Neutropenia- Other (Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| Wound-infectious | s is graded in th | ne DERMATOLOGY/SK | IN category. | | |
| | | LYMPHA | ATICS | | |
| Lymphatics | normal | mild<br>lymphedema | moderate<br>lymphedema<br>requiring<br>compression<br>; lymphocyst | severe lymphedema limiting function; lymphocyst requiring surgery | severe lymphedema limiting function with ulceration |
| Lymphatics-<br>Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | METABOLIC/LA | BORATORY | | |

| | | Gra | de | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Acidosis<br>(metabolic or<br>respiratory) | normal | pH < normal, but ≥7.3 | - | pH < 7.3 | pH < 7.3<br>with life-<br>threatening<br>physiologic<br>consequence<br>s |
| Alkalosis<br>(metabolic or<br>respiratory) | normal | pH ><br>normal, but<br>≤7.5 | - | pH > 7.5 | pH > 7.5<br>with life-<br>threatening<br>physiologic<br>consequence<br>s |
| Amylase | WNL | > ULN - 1.5<br>x ULN | > 1.5 - 2.0 x<br>ULN | > 2.0 - 5.0 x<br>ULN | >5.0 x ULN |
| Bicarbonate | WNL | < LLN - 16<br>mEq/dl | 11 - 15<br>mEq/dl | 8 - 10<br>mEq/dl | < 8 mEq/dl |
| CPK (creatine phosphokinase) | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5 x<br>ULN | > 5 - 10 x<br>ULN | > 10 x ULN |
| Hypercalcemia | WNL | > ULN -<br>11.5 mg/dl<br>> ULN - 2.9<br>mmol/L | >11.5 - 12.5<br>mg/dl<br>> 2.9 - 3.1<br>mmol/L | >12.5 - 13.5<br>mg/dl<br>> 3.1 - 3.4<br>mmol/L | > 13.5 mg/dl<br>> 3.4<br>mmol/L |
| Hypercholester<br>olemia | WNL | > ULN -<br>300 mg/dl<br>> ULN -<br>7.75<br>mmol/L | > 300 - 400<br>mg/dl<br>> 7.75 -<br>10.34<br>mmol/L | > 400 - 500<br>mg/dl<br>>10.34 -<br>12.92<br>mmol/L | > 500 mg/dl<br>> 12.92<br>mmol/L |
| Hyperglycemia | WNL | > ULN -<br>160 mg/dl<br>> ULN - 8.9<br>mmol/L | > 160 - 250<br>mg/dl<br>> 8.9 - 13.9<br>mmol/L | > 250 - 500<br>mg/dl<br>> 13.9 -<br>27.8<br>mmol/L | > 500 mg/dl<br>> 27.8<br>mmol/L or<br>ketoacidosis |
| Hyperkalemia | WNL | > ULN - 5.5<br>mmol/L | > 5.5 - 6.0<br>mmol/L | > 6.0 - 7.0<br>mmol/L | > 7.0<br>mmol/L |
| Hypermagnese<br>mia | WNL | > ULN - 3.0<br>mg/dl<br>> ULN -<br>1.23<br>mmol/L | - | > 3.0 - 8.0<br>mg/dl<br>> 1.23 -<br>3.30<br>mmol/L | > 8.0 mg/dl<br>> 3.30<br>mmol/L |
| Hypernatremia | WNL | > ULN -<br>150 mmol/L | >150 - 155<br>mmol/L | >155 - 160<br>mmol/L | >160<br>mmol/L |
| Hypertriglyceri demia | WNL | > ULN - 2.5<br>x ULN | > 2.5 - 5.0 x<br>ULN | > 5.0 - 10 x<br>ULN | > 10 x ULN |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hyperuricemia | WNL | > ULN - \le 10 mg/dl \le 0.59 mmol/L without physiologic consequence s | - | > ULN - \le 10 mg/dl \le 0.59 mmol/L with physiologic consequence s | > 10 mg/dl<br>> 0.59<br>mmol/L |
| Also consider Tu | umor lysis syndror | ne, Renal failure, Cr | eatinine, Potassium. | 5 | |
| Hypocalcemia | WNL | <lln -="" 8.0<br="">mg/dl<br/><lln -="" 2.0<br="">mmol/L</lln></lln> | 7.0 - < 8.0<br>mg/dl<br>1.75 - < 2.0 | 6.0 - < 7.0<br>mg/dl<br>1.5 - < 1.75 | <6.0 mg/dl<br>< 1.5<br>mmol/L |
| Hypoglycemia | WNL | <pre>mmol/L</pre> | mmol/L<br>40 - < 55<br>mg/dl<br>2.2 - < 3.0<br>mmol/L | mmol/L<br>30 - < 40<br>mg/dl<br>1.7 - < 2.2<br>mmol/L | < 30 mg/dl<br>< 1.7<br>mmol/L |
| Hypokalemia | WNL | <lln -="" 3.0<br="">mmol/L</lln> | - | 2.5 - <3.0<br>mmol/L | <2.5<br>mmol/L |
| Hypomagnesem ia | WNL | <lln -="" 1.2<br="">mg/dl<br/><lln -="" 0.5<br="">mmol/L</lln></lln> | 0.9 - <1.2<br>mg/dl<br>0.4 - < 0.5<br>mmol/L | 0.7 - < 0.9<br>mg/dl<br>0.3 - < 0.4<br>mmol/L | < 0.7 mg/dl<br>< 0.3<br>mmol/L |
| Hyponatremia | WNL | <lln -="" 130<br="">mmol/L</lln> | - | 120 - <130<br>mmol/L | <120<br>mmol/L |
| Hypophosphate<br>mia | WNL | <lln -2.5<br="">mg/dl<br/><lln -="" 0.8<br="">mmol/L</lln></lln> | ≥2.0 - <2.5<br>mg/dl<br>≥0.6 - <0.8<br>mmol/L | ≥1.0 - <2.0<br>mg/dl<br>≥0.3 - <0.6<br>mmol/L | < 1.0 mg/dl<br><0.3<br>mmol/L |
| | | NDOCRINE categor | | | |
| Lipase | WNL | > ULN - 1.5<br>x ULN | > 1.5 - 2.0 x<br>ULN | > 2.0 - 5.0 x<br>ULN | > 5.0 x ULN |
| Metabolic/Labo<br>ratory-Other<br>(Specify, | none | mild | moderate | severe | life-<br>threatening<br>or disabling |
| | | MUSCULO | SKELETAL | | |
| | ded in the PAIN c | | ~ | | |
| Arthritis | none | mild pain with<br>inflammation,<br>erythema or joint<br>swelling but not<br>interfering with<br>function | moderate pain with inflammation, erythema, or joint swelling interfering with function, but not interfering with activities of daily living | severe pain with<br>inflammation,<br>erythema, or joint<br>swelling and<br>interfering with<br>activities of daily<br>living | disabling |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Muscle weakness<br>(not due to<br>neuropathy) | normal | asymptomatic<br>with weakness on<br>physical exam | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | bedridden or<br>disabling |
| Myalgia is graded in the | | | | | |
| Myositis<br>(inflammation/dama<br>ge of muscle) | none | mild pain, not interfering with function | pain interfering<br>with function, but<br>not interfering<br>with activities of<br>daily living | pain interfering<br>with function and<br>interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| Also consider CPK. | | - (;1 | | | |
| Note: Myositis implies Osteonecrosis (avascular necrosis) | s muscle damag<br>none | asymptomatic<br>and detected by<br>imaging only | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | symptomatic; or disabling |
| Musculoskeletal-<br>Other<br>(Specify, | none | mild | moderate | severe | life-threatening or<br>disabling |
| , | | NEURO | OLOGY | | |
| Aphasia, receptive and | /or expressive, | is graded under Speec | h impairment in the | NEUROLOGY cates | gory. |
| Arachnoiditis/menin gismus/radiculitis | absent | mild pain not interfering with function | moderate pain<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain<br>interfering with<br>activities of daily<br>living | unable to<br>function or<br>perform activities<br>of daily living;<br>bedridden;<br>paraplegia |
| Also consider Headach | | | | 1 | 1 1 1.1 |
| Ataxia (incoordination) | normal | asymptomatic but<br>abnormal on<br>physical exam,<br>and not<br>interfering with<br>function | mild symptoms<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | moderate<br>symptoms<br>interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| CNS cerebrovascular ischemia | none | <u>-</u> | - | transient<br>ischemic event or<br>attack (TIA) | permanent event<br>(e.g., cerebral<br>vascular<br>accident) |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Cognitive<br>disturbance/<br>learning problems | none | cognitive disability; not interfering with work/school performance; preservation of intelligence | cognitive disability; interfering with work/school performance; decline of 1 SD (Standard Deviation) or loss of developmental milestones | cognitive disability; resulting in significant impairment of work/school performance; cognitive decline > 2 SD | inability to<br>work/frank<br>mental<br>retardation |
| Confusion | normal | confusion or<br>disorientation or<br>attention deficit<br>of brief duration;<br>resolves<br>spontaneously<br>with no sequelae | confusion or<br>disorientation or<br>attention deficit<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | confusion or<br>delirium<br>interfering with<br>activities of daily<br>living | harmful to others<br>or self; requiring<br>hospitalization |
| Cranial neuropathy is | | EUROLOGY categor | y as Neuropathy-crar | nial. | |
| Delusions | normal | - | - | present | toxic psychosis |
| Depressed level of consciousness | normal | somnolence or<br>sedation not<br>interfering with<br>function | somnolence or<br>sedation<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | obtundation or<br>stupor; difficult<br>to arouse;<br>interfering with<br>activities of daily<br>living | coma |
| Note: Syncope (faintir | ng) is graded in t | he NEUROLOGY ca | itegory. | | |
| Dizziness/lightheade dness | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| Dysphasia, receptive a | nd/or expressive | e, is graded under Spe | | ne NEUROLOGY ca | tegory. |
| Extrapyramidal/<br>involuntary<br>movement/<br>restlessness | none | mild involuntary<br>movements not<br>interfering with<br>function | moderate involuntary movements interfering with function, but not interfering with activities of daily living | severe<br>involuntary<br>movements or<br>torticollis<br>interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| | normal | | - | present | toxic psychosis |
| Hallucinations | поннач | - | <del>-</del> | DIESEIII | 101210 11500 1101212 |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Insomnia Note: This toxicity is g | normal graded when inso | occasional difficulty sleeping not interfering with function mnia is related to tree | difficulty sleeping interfering with function, but not interfering with activities of daily living atment. If pain or oth | frequent difficulty sleeping, interfering with activities of daily living er symptoms interfer | re with sleep do |
| NOT grade as insomni | | | | | |
| Irrit ability (children <3 years of age) | normal | mild; easily<br>consolable | moderate;<br>requiring<br>increased<br>attention | severe;<br>inconsolable | - |
| Leukoencephalopath<br>y associated<br>radiological findings | none | mild increase in SAS (subarachnoid space) and/or mild ventriculomegaly; and/or small (+/- multiple) focal T2 hyperintensities, involving periventricular white matter or < 1/3 of susceptible areas of cerebrum | moderate increase in SAS; and/or moderate ventriculomegaly ; and/or focal T2 hyperintensities extending into centrum ovale; or involving 1/3 to 2/3 of susceptible areas of cerebrum | severe increase in SAS; severe ventriculomegaly; near total white matter T2 hyperintensities or diffuse low attenuation (CT); focal white matter necrosis (cystic) | severe increase in SAS; severe ventriculomegaly; diffuse low attenuation with calcification (CT); diffuse white matter necrosis (MRI) |
| Memory loss | normal | memory loss not interfering with function | memory loss<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | memory loss<br>interfering with<br>activities of daily<br>living | amnesia |
| Mood alteration-<br>anxiety agitation | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | suicidal ideation<br>or danger to self |
| Mood alteration-<br>depression | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | suicidal ideation<br>or danger to self |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Mood alteration-<br>euphoria | normal | mild mood<br>alteration not<br>interfering with<br>function | moderate mood<br>alteration<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe mood<br>alteration<br>interfering with<br>activities of daily<br>living | danger to self |
| Neuropathic pain is gr | | N category. | | | life threatening |
| Neuropathy- cranial | absent | - | present, not<br>interfering with<br>activities of daily<br>living | present,<br>interfering with<br>activities of daily<br>living | life-threatening,<br>disabling |
| Neuropathy- motor | normal | subjective<br>weakness but no<br>objective findings | mild objective<br>weakness<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | objective<br>weakness<br>interfering with<br>activities of daily<br>living | paralysis |
| Neuropathy-sensory | normal | loss of deep<br>tendon reflexes or<br>paresthesia<br>(including<br>tingling) but not<br>interfering with<br>function | objective sensory<br>loss or<br>paresthesia<br>(including<br>tingling),<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | sensory loss or<br>paresthesia<br>interfering with<br>activities of daily<br>living | permanent<br>sensory loss that<br>interferes with<br>function |
| Nystagmus<br>Also consider Vision- | absent<br>double vision. | present | - | - | - |
| Personality/behavior<br>al | normal | change, but not<br>disruptive to<br>patient or family | disruptive to patient or family | disruptive to<br>patient and<br>family; requiring<br>mental health<br>intervention | harmful to others<br>or self; requiring<br>hospitalization |
| Pyramidal tract<br>dysfunction (e.g., ↑<br>tone, hyperreflexia,<br>positive Babinski, ↓<br>fine motor<br>coordination) | normal | asymptomatic<br>with abnormality<br>on physical<br>examination | symptomatic or<br>interfering with<br>function but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden or<br>disabling;<br>paralysis |
| Seizure(s) | none | - | seizure(s) self-<br>limited and<br>consciousness is<br>preserved | seizure(s) in<br>which<br>consciousness is<br>altered | seizures of any<br>type which are<br>prolonged,<br>repetitive, or<br>difficult to<br>control (e.g.,<br>status epilepticus,<br>intractable<br>epilepsy) |

| | | Gı | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Speech impairment<br>(e.g., dysphasia or<br>aphasia) | normal | - | awareness of<br>receptive or<br>expressive<br>dysphasia, not<br>impairing ability<br>to communicate | receptive or<br>expressive<br>dysphasia,<br>impairing ability<br>to communicate | inability to communicate |
| Syncope (fainting) | absent | - | - | present | -<br>1 · |
| Also consider CARD | none | mild and brief or<br>intermittent but<br>not interfering<br>with function | moderate tremor interfering with function, but not interfering with activities of daily living | severe tremor<br>interfering with<br>activities of daily<br>living | - |
| Vertigo | none | not interfering with function | interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | bedridden or<br>disabling |
| Neurology-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | OCULAI | R/VISUAL | | |
| Cataract | none | asymptomatic | symptomatic,<br>partial visual loss | symptomatic, visual loss requiring treatment or interfering with function | - |
| Conjunctivitis | none | abnormal ophthalmologic changes, but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Dry eye | normal | mild, not<br>requiring<br>treatment | moderate or requiring artificial tears | - | - |
| Glaucoma | none | increase in<br>intraocular<br>pressure but no<br>visual loss | increase in intraocular pressure with retinal changes | visual<br>impairment | unilateral or<br>bilateral loss of<br>vision (blindness) |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Keratitis<br>(corneal<br>inflammation/<br>corneal ulceration) | none | abnormal ophthalmologic changes but asymptomatic or symptomatic without visual impairment (i.e., pain and irritation) | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | unilateral or<br>bilateral loss of<br>vision (blindness) |
| Tearing (watery eyes) | none | mild: not<br>interfering with<br>function | moderate:<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | interfering with<br>activities of daily<br>living | - |
| Vision- blurred vision | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- double<br>vision (diplopia) | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- flashing<br>lights/floaters | normal | mild, not<br>interfering with<br>function | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- night<br>blindness<br>(nyctalopia) | normal | abnormal electro-<br>retinography but<br>asymptomatic | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Vision- photophobia | normal | - | symptomatic and interfering with function, but not interfering with activities of daily living | symptomatic and interfering with activities of daily living | - |
| Ocular/Visual-Other (Specify, | normal | mild | moderate | severe | unilateral or<br>bilateral loss of<br>vision (blindness) |

| | | G | rade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Abdominal pain or cramping | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Arthralgia<br>(joint pain) | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Arthritis (joint pain w | ith clinical sig | ns of inflammation) is g | graded in the MUSCU | JLOSKELETAL cat | egory. |
| Bone pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Chest pain<br>(non-cardiac and<br>non-pleuritic) | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Dysmenorrhea | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Dyspareunia | none | mild pain not interfering with function | moderate pain interfering with sexual activity | severe pain<br>preventing sexual<br>activity | - |
| | he RENAL/GI | ENITOURINARY cate | | | |
| Earache (otalgia) | none | mild pain not interfering with function | moderate pain:<br>pain or analgesics<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Headache | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Hepatic pain | none | mild pain not interfering with function | moderate pain:<br>pain or analgesics<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Myalgia<br>(muscle pain) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Neuropathic pain<br>(e.g., jaw pain,<br>neurologic pain,<br>phantom limb pain,<br>post-infectious<br>neuralgia, or painful<br>neuropathies) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pain due to radiation | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pelvic pain | none | mild pain not interfering with function | moderate pain:<br>pain or analgesics<br>interfering with<br>function, but not<br>interfering with<br>activities of daily<br>living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Pleuritic pain | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |

| | | Gı | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Rectal or perirectal pain (proctalgia) | none | mild pain not<br>interfering with<br>function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Tumor pain (onset or exacerbation of tumor pain due to treatment) | none | mild pain not interfering with function | moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living | severe pain: pain<br>or analgesics<br>severely<br>interfering with<br>activities of daily<br>living | disabling |
| Tumor flair is graded: Pain-Other | | mild | moderate | severe | disabling |
| (Specify, | none | IIIIQ | moderate | severe | disabiling |
| | | PULM | ONARY | | |
| Adult Respiratory<br>Distress Syndrome<br>(ARDS) | absent | - | - | - | present |
| Apnea | none | - | - | present | requiring intubation |
| Carbon monoxide diffusion capacity (DL <sub>CO</sub> ) | ≥ 90% of pretreatment or normal value | ≥75 - <90% of pretreatment or normal value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of pretreatment or normal value | < 25% of<br>pretreatment or<br>normal value |
| Cough | absent | mild, relieved by<br>non-prescription<br>medication | requiring narcotic antitussive | severe cough or<br>coughing spasms,<br>poorly controlled<br>or unresponsive<br>to treatment | - |
| Dyspnea (shortness of breath) | normal | - | dyspnea on exertion | dyspnea at<br>normal level of<br>activity | dyspnea at rest or<br>requiring<br>ventilator support |
| FEV <sub>1</sub> | ≥ 90% of pretreatment or normal value | ≥75 - <90% of pretreatment or normal value | ≥50 - <75% of pretreatment or normal value | ≥25 - <50% of pretreatment or normal value | < 25% of<br>pretreatment or<br>normal value |
| Hiccoughs (hiccups, singultus) | none | mild, not<br>requiring<br>treatment | moderate,<br>requiring<br>treatment | severe,<br>prolonged, and<br>refractory to<br>treatment | - |

| | Grade | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Hypoxia | normal | - | decreased O <sub>2</sub> saturation with exercise | decreased O <sub>2</sub> saturation at rest, requiring supplemental oxygen | decreased O <sub>2</sub> saturation, requiring pressure support (CPAP) or assisted ventilation |
| Pleural effusion<br>(non-malignant) | none | asymptomatic<br>and not requiring<br>treatment | symptomatic,<br>requiring<br>diuretics | symptomatic, requiring O <sub>2</sub> or therapeutic | life-threatening<br>(e.g., requiring<br>intubation) |
| Dlauritia nain ia arada | d in the DAIN est | 20071 | | thoracentesis | |
| Pleuritic pain is graded<br>Pneumonitis/pulmon<br>ary infiltrates | none | radiographic changes but asymptomatic or symptoms not requiring steroids | radiographic<br>changes and<br>requiring steroids<br>or diuretics | radiographic<br>changes and<br>requiring oxygen | radiographic<br>changes and<br>requiring assisted<br>ventilation |
| Pneumothorax | none | no intervention | chest tube | sclerosis or | life-threatening |
| | | required | required | surgery required | |
| Pulmonary embolism | | | | | category. |
| Pulmonary fibrosis | none | radiographic<br>changes, but<br>asymptomatic or<br>symptoms not<br>requiring steroids | requiring steroids<br>or diuretics | requiring oxygen | requiring assisted ventilation |
| Note: Radiation-relate | d pulmonary fibro | | RTOG/EORTC Late | Radiation Morbidity | Scoring Scheme- |
| Lung. (See Appendix | | | | | s coming s chieffing |
| Voice changes/stridor/laryn x (e.g., hoarseness, loss of voice, laryngitis) | normal | mild or<br>intermittent<br>hoarseness | persistent<br>hoarseness, but<br>able to vocalize;<br>may have mild to<br>moderate edema | whispered<br>speech, not able<br>to vocalize; may<br>have marked<br>edema | marked<br>dyspnea/stridor<br>requiring<br>tracheostomy or<br>intubation |
| Radiation-related | hemoptysis from TINAL category. | Radiation-related h | raded as Grade 4 Mu | y.<br>acositis due to radiati<br>horacic cavity is grad | |
| Pulmonary-Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| , | | RENAL/CENI | ITOURINARY | | |
| Bladder spasms | absent | mild symptoms,<br>not requiring<br>intervention | symptoms<br>requiring<br>antispasmotic | severe symptoms requiring narcotic | - |
| Creatinine Note: Adjust to age-ap | WNL | > ULN - 1.5 x<br>ULN | > 1.5 - 3.0 x<br>ULN | > 3.0 - 6.0 x<br>ULN | > 6.0 x ULN |
| Dysuria | none | mild symptoms | symptoms | symptoms not | |
| (painful urination) | 110110 | requiring no intervention | relieved with<br>therapy | relieved despite<br>therapy | |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Fistula or GU fistula (e.g., vaginal, vesicovaginal) | none | - | - | requiring intervention | requiring surgery |
| Hemoglobinuria | - | present | - | - | - |
| Hematuria (in the abse | ence of vaginal b | | the HEMORRHAG | | |
| Incontinence | none | with coughing, sneezing, etc. | spontaneous,<br>some control | no control (in the absence of fistula) | - |
| Operative injury to bladder and/or ureter | none | - | injury of bladder<br>with primary<br>repair | sepsis, fistula, or<br>obstruction<br>requiring<br>secondary<br>surgery; loss of<br>one kidney;<br>injury requiring<br>anastomosis or<br>re-implantation | septic obstruction<br>of both kidneys<br>or vesicovaginal<br>fistula requiring<br>diversion |
| Proteinuria | normal or < 0.15 g/24 hours | 1+ or 0.15 - 1.0<br>g/24 hours | 2+ to 3+ or 1.0 -<br>3.5 g/24 hours | 4+ or > 3.5 g/24 hours | nephrotic<br>syndrome |
| Note: If there is an inc | | een absolute value an | d uristix reading, use | e the absolute value f | or grading. |
| Renal failure | none | - | - | requiring dialysis,<br>but reversible | requiring dialysis and irreversible |
| Ureteral obstruction | none | unilateral, not requiring surgery | - | bilateral, not<br>requiring surgery | stent,<br>nephrostomy<br>tube, or surgery |
| Urinary electrolyte<br>wasting (e.g.,<br>Fanconi's syndrome,<br>renal tubular<br>acidosis) | none | asymptomatic,<br>not requiring<br>treatment | mild, reversible<br>and manageable<br>with oral<br>replacement | reversible but requiring IV replacement | irreversible,<br>requiring<br>continued<br>replacement |
| Also consider Acidosi | | | | 1 1 | |
| Urinary<br>frequency/urgency | normal | increase in frequency or nocturia up to 2 x normal | increase > 2 x<br>normal but <<br>hourly | hourly or more<br>with urgency, or<br>requiring catheter | - |
| Urinary retention | normal | hesitancy or<br>dribbling, but no<br>significant<br>residual urine;<br>retention<br>occurring during<br>the immediate<br>postoperative<br>period | hesitancy requiring medication or occasional in/out catheterization (<4 x per week), or operative bladder atony requiring indwelling catheter beyond immediate postoperative period but for < 6 weeks | requiring frequent in/out catheterization (≥ 4 x per week) or urological intervention (e.g., TURP, suprapubic tube, urethrotomy) | bladder rupture |

| | | Gr | ade | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Urine color change<br>(not related to other<br>dietary or<br>physiologic cause<br>e.g., bilirubin,<br>concentrated urine,<br>hematuria) | normal | asymptomatic,<br>change in urine<br>color | - | - | - |
| Vaginal bleeding is gra | aded in the HEM | ORRHAGE categor | V. | | |
| Vaginitis<br>(not due to infection) | none | mild, not<br>requiring<br>treatment | moderate,<br>relieved with<br>treatment | severe, not<br>relieved with<br>treatment, or<br>ulceration not<br>requiring surgery | ulceration<br>requiring surgery |
| Renal/Genitourinary-<br>Other (Specify, | none | mild | moderate | severe | life-threatening or disabling |
| | | SECONDARY | MALIGNANCY | | |
| Secondary Malignancy-Other (Specify type,) excludes metastastic tumors | none | - | - | - | present |
| | <b>C</b> 1 | EVITAT /DEPDANI | UCTIVE FUNCTIO | N | |
| Dyspareunia is graded | | | JCIIVE FUNCTIO | 71 | |
| Dysmenorrhea is grade | ed in the PAIN ca | ategory. | | | |
| Erectile impotence | normal | mild (erections<br>impaired but<br>satisfactory) | moderate<br>(erections<br>impaired,<br>unsatisfactory for<br>intercourse) | no erections | - |
| Female sterility | normal | - | - | sterile | - |
| Femininization of male | | | | | |
| Irregular menses<br>(change from<br>baseline) | normal | occasionally irregular or lengthened interval, but continuing menstrual cycles | very irregular, but<br>continuing<br>menstrual cycles | persistent<br>amenorrhea | - |
| Libido | normal | decrease in interest | severe loss of interest | - | - |
| Male infertility | - | - | Oligospermia<br>(low sperm<br>count) | Azoospermia<br>(no sperm) | - |
| Masculinization of fen | nale is graded in | the ENDOCRINE ca | tegory. | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Vaginal dryness | normal | mild | requiring | - | - |
| | | | treatment and/or | | |
| | | | interfering with | | |
| | | | sexual function, | | |
| C 1/D 1 .: | | '1 1 | dyspareunia | | 1: 11: |
| Sexual/Reproductive | none | mild | moderate | severe | disabling |
| Function-Other (Specify, | | | | | |
| (specify, | | | | | |
| , | | | | | |
| | | | ded in previous cate | | |
| Acute vascular leak sy | | | | | |
| ARDS (Adult Respira | | | | | |
| Autoimmune reactions | | | | | |
| DIC (disseminated int | | | | | |
| Fanconi's syndrome is | | | | | |
| Renal tubular acidosis Stevens-Johnson synd | | | | | |
| SIADH (syndrome of | | | | | у. |
| Thrombotic microangi | | | | | gymdrom/HIIC) ig |
| graded in the COAGU | | | openie purpura/111 ( | of hemorytic dreinic | syndrom/1103) is |
| Tumor flare | none | mild pain not | moderate pain; | severe pain; pain | Disabling |
| | | interfering with | pain or analgesics | or analgesics | |
| | | function | interfering with | interfering with | |
| | | | function, but not | function and | |
| | | | interfering with | interfering with | |
| | | | activities of daily | activities of daily | |
| A1: 1 II | .1 | | living | living | |
| Also consider Hyperca<br>Note: Tumor flare is | | o constallation of a | mantona and sice sie | direct relation to ini | itiation of the areas |
| | | | mptoms and signs in ). The symptoms/sign | | |
| visible tumor, hy | | | ther electrolyte distu | | n, mnammadon of |
| Tumor lysis | absent | - | - | present | - |
| syndrome | | | | | |
| Also consider Hyperka | alemia, Creatinin | e | . 1 1 | 1 1 1 2 | |
| Urinary electrolyte wa RENAL/GENITOUR | | | tubular acidosis) is a | graded under the | |
| Syndromes-Other | | | 1 4 . | | 1:0 4 |
| 25 | none | mild | moderate | severe | life-threatening or |
| (Specify, | none | mild | moderate | severe | life-threatening or disabling |

## Appendix II Toxicity Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| Toxicity: | Date of Treatment | : | Course Number: |
|---|---|---|---|
| Date of onset: | | | Grade at onset: |
| Date of first change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Date of next change in grade: | | | Grade: |
| Did toxicity resolve? | Yes | No | |
| If so, date of resolution of toxicity: | | | |
| Date of last observation (if prior to | | | |
| recovery): | | | |
| Reason(s) observations stopped (if | | | |
| prior to recovery): | | | |
| Was patient retreated? | Yes | No | |
| If yes, was treatment delayed for | Yes | No | |
| recovery? | | | |
| Date of next treatment? | | | |
| Dose reduced for next treatment? | Yes | No | |
| Additional Comments: | | | |
| If module is being activated for new | toxicity, not currer | ntly in CTC, please | e provide definitions for |
| toxicity grading: | • • | , 1 | |
| Grade 0 = | | | |
| Grade 1 = | | | |
| Grade 2 = | | | |
| Grade 3 = | | | |
| Grade 4 = | | | |

## Appendix III Infection Module

To be implemented at the request of the study sponsor or principal investigator in the protocol or by protocol amendment when more detailed information is considered pertinent.

| | | • | definitions to grade the following (CHOOSE O | • | ection. |
|---|---|---|---|---|---|
| | BACTERIAL | <b>FUNGAL</b> | PROTOZOAL | VIRAL | UNKNOWN |
| 3. | Specify site of infe<br>BLOOD CULTUR<br>BONE INFECTIO<br>CATHETER (intra<br>CATHETER (intra<br>CENTRAL NERV<br>EAR INFECTION<br>EYE INFECTION<br>GASTROINTEST<br>ORAL INFECTIO<br>PNEUMONIA<br>SKIN INFECTION<br>UPPER RESPIRA<br>URINARY TRAC<br>VAGINAL INFEC | RE POSITIVE N avenous) avenous), tunnel OUS SYSTEM INAL INFECTION TORY INFECT | INFECTION<br>ON | LL THAT APPLY): | |
| | INFECTION, not of | otherwise specifi | ed (Specify site, | ) | |
| 4.<br>5. | Specify organism, if known: Prophylactic antibiotic, antifungal, or antiviral therapy administration Yes No If prophylaxis was given prior to infection, please specify below: Antibiotic prophylaxis | | | | |
| | Antifungal prophylaxis | | | | |
| | Antiviral prophylaxis | | | | |
| | Other prophylaxis | | | | |

## Appendix IV Performance Status Scales/Scores

| ECOG or Zubrod Scale | | Karnofsky Score |
|---|---|---|
| 0 | Asymptomatic and fully active | 100% |
| 1 | Symptomatic; fully ambulatory; restricted in physically strenuous activity | 80-90% |
| 2 | Symptomatic; ambulatory; capable of self-care; more than 50% of waking hours are spent out of bed | 60-70% |
| 3 | Symptomatic; limited self-care; spends more than 50% of time in bed, but not bedridden | 40-50% |
| 4 | Completely disabled; no self-care; bedridden | 20-30% |

Appendix V
RTOG/EORTC Late Radiation Morbidity Scoring Scheme
Use for toxicities occurring greater than 90 days after radiation therapy.

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Bladder-<br>Late RT Morbidity<br>Scoring | No change<br>from baseline | Slight epithelial<br>atrophy/minor<br>telangiectasia<br>(microscopic<br>hematuria) | Moderate<br>frequency/<br>generalized<br>telangiectasia/<br>intermittent<br>macroscopic<br>hematuria | Severe frequency and dysuria/severe generalized telangiectasia (often with petechiae); frequent hematuria; reduction in bladder capacity (< 150 cc) | Necrosis/contract<br>ed bladder<br>(capacity < 100<br>cc)/severe<br>hemorrhagic<br>cystitis |
| Bone-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic;<br>no growth<br>retardation;<br>reduced bone<br>density | Moderate pain or<br>tenderness;<br>growth<br>retardation;<br>irregular bone<br>sclerosis | Severe pain or<br>tenderness;<br>complete arrest of<br>bone growth;<br>dense bone<br>sclerosis | Necrosis/<br>spontaneous<br>fracture |
| Brain-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild headache;<br>slight lethargy | Moderate<br>headache; great<br>lethargy | Severe<br>headaches; severe<br>CNS dysfunction<br>(partial loss of<br>power or<br>dyskinesia) | Seizures or paralysis; coma |
| Esophagus-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild fibrosis;<br>slight difficulty in<br>swallowing<br>solids; no pain on<br>swallowing | Unable to take<br>solid food<br>normally;<br>swallowing semi-<br>solid food;<br>dilatation may be<br>indicated | Severe fibrosis;<br>able to swallow<br>only liquids; may<br>have pain on<br>swallowing;<br>dilation required | Necrosis/<br>perforation;<br>fistula |
| Heart-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic or<br>mild symptoms;<br>transient T wave<br>inversion and ST<br>changes; sinus<br>tachycardia > 110<br>(at rest) | Moderate angina<br>on effort; mild<br>pericarditis;<br>normal heart size;<br>persistent<br>abnormal T wave<br>and ST changes;<br>low QRS | Severe angina; pericardial effusion; constrictive pericarditis; moderate heart failure; cardiac enlargement; EKG abnormalities | Tamponade/sever<br>e heart<br>failure/severe<br>constrictive<br>pericarditis |
| Joint-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild joint<br>stiffness; slight<br>limitation of<br>movement | Moderate<br>stiffness;<br>intermittent or<br>moderate joint<br>pain; moderate | Severe joint<br>stiffness; pain<br>with severe<br>limitation of<br>movement | Necrosis/complet<br>e fixation |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| | | | limitation of movement | | |
| Kidney-<br>Late RT Morbidity<br>Scoring | No change from baseline | Transient albuminuria; no hypertension; mild impairment of renal function; urea 25 - 35 mg%; creatinine 1.5 - 2.0 mg%; creatinine clearance > 75% | Persistent moderate albuminuria (2+); mild hypertension; no related anemia; moderate impairment of renal function; urea > 36 - 60 mg%; creatinine clearance > 50 - 74% | Severe albuminuria; severe hypertension; persistent anemia (< 10 g%); severe renal failure; urea > 60 mg%; creatinine > 4 mg%; creatinine clearance < 50% | Malignant hypertension; uremic coma/urea > 100% |
| Larynx-<br>Late RT Morbidity<br>Scoring | No change from baseline | Hoarseness;<br>slight arytenoid<br>edema | Moderate arytenoid edema; chondritis | Severe edema;<br>severe chondritis | Necrosis |
| Liver-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild lassitude;<br>nausea;<br>dyspepsia;<br>slightly abnormal<br>liver function | Moderate<br>symptoms; some<br>abnormal liver<br>function tests;<br>serum albumin<br>normal | Disabling hepatic insufficiency; liver function tests grossly abnormal; low albumin; edema or ascites | Necrosis/hepatic<br>coma or<br>encephalopathy |
| Lung-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic or<br>mild symptoms<br>(dry cough);<br>slight<br>radiographic<br>appearances | Moderate<br>symptomatic<br>fibrosis or<br>pneumonitis<br>(severe cough);<br>low grade fever;<br>patchy<br>radiographic<br>appearances | Severe<br>symptomatic<br>fibrosis or<br>pneumonitis;<br>dense<br>radiographic<br>changes | Severe<br>respiratory<br>insufficiency/<br>continuous<br>O2/assisted<br>ventilation |
| Mucous membrane-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight atrophy<br>and dryness | Moderate atrophy and telangiectasia; little mucus | Marked atrophy<br>with complete<br>dryness; severe<br>telangiectasia | Ulceration |
| Salivary glands-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight dryness of<br>mouth; good<br>response on<br>stimulation | Moderate dryness<br>of mouth; poor<br>response on<br>stimulation | Complete dryness<br>of mouth; no<br>response on<br>stimulation | Fibrosis |
| Skin-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight atrophy;<br>pigmentation<br>change; some<br>hair loss | Patchy atrophy;<br>moderate<br>telangiectasia;<br>total hair loss | Marked atrophy;<br>gross<br>telangiectasia | Ulceration |
| Small/Large<br>intestine-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild diarrhea;<br>mild cramping;<br>bowel movement<br>5 x daily slight<br>rectal discharge | Moderate diarrhea and colic; bowel movement > 5 x daily; excessive | Obstruction or bleeding, requiring surgery | Necrosis/<br>perforation fistula |

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | oxicity 0 | | 1 2 | | 4 |
| | | or bleeding | rectal mucus or intermittent bleeding | | |
| Spinal cord-<br>Late RT Morbidity<br>Scoring | No change from baseline | Mild Lhermitte's syndrome | Severe<br>Lhermitte's<br>syndrome | Objective<br>neurological<br>findings at or<br>below cord level<br>treatment | Mono-, para-,<br>quadriplegia |
| Subcutaneous tissue-<br>Late RT Morbidity<br>Scoring | No change from baseline | Slight induration<br>(fibrosis) and loss<br>of subcutaneous<br>fat | Moderate fibrosis<br>but<br>asymptomatic;<br>slight field<br>contracture; <<br>10% linear<br>reduction | Severe induration<br>and loss of<br>subcutaneous<br>tissue; field<br>contracture ><br>10% linear<br>measurement | Necrosis |
| Eye-<br>Late RT Morbidity<br>Scoring | No change from baseline | Asymptomatic cataract; minor corneal ulceration or keratitis | Symptomatic cataract; moderate corneal ulceration; minor retinopathy or glaucoma | Severe keratitis;<br>severe<br>retinopathy or<br>detachment;<br>severe glaucoma | Panophthalmitis;<br>blindness |
| Radiation-Other (Specify, | None | Mild | Moderate | Severe | Life-threatening or disabling |

| A Phase I/II Trial of Escalating Dose of Yttrium-90-labeled Anti-CD20 Monoclonal Antibody in |
|---|
| Combination with High-Dose Etoposide and Cyclophosphamide followed by Autologous Stem |
| Cell Transplantation for Patients with Relapsed B-Cell Non-Hodgkin's Lymphoma |

NCT00562978

Document Date 03/28/2014

## Appendix VI BMT Complex/Multi-Component Events

| Grade | | | | | |
|---|---|---|---|---|---|
| Toxicity | 0 | 1 | 2 | 3 | 4 |
| Note: The grading of Complex/Multi-Component Events in bone marrow transplant will be defined in the protocol. | | | | | |
| The grading so | ale must use the | CTC criteria for | r grading the specific con | nponent events (to | oxicities). |
| Failure to engraft | absent | mild | moderate | severe | life-threatening |
| Also consider Hemo | oglobin (Hgb), N | Veutrophils/gran | ulocytes (ANC/AGC), Pla | atelets | |
| Graft versus host | absent | mild | moderate | severe | life-threatening |
| disease | | | | | |
| Also consider Fatig | Also consider Fatigue, Rash/desquamation, Diarrhea, Bilirubin-GVHD | | | | |
| Stem cell infusion | absent | mild | moderate | severe | life-threatening |
| complications | | | | | |
| | Also consider Allergic reaction/hypersensitivity, Arrhythmia, Hypertension, Hypotension, Fever, Rigors/chills, | | | | |
| Sweating, Rash/desquamation, Urticaria, Diarrhea, Nausea, Vomiting, Hemorrhage/bleeding with grade 3 or 4 | | | | | |
| thrombocytopenia, Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia, Hemoptysis, Alkaline phosphatase, | | | | | |
| Bilirubin, GGT, SGOT, SGPT, Infection, Hyperkalemia, Hypernatremia, Hypokalemia, Depressed level of | | | | | |
| consciousness, Seizures, Abdominal pain, Headache, Creatinine, Hemoglobinuria | | | | | |
| Veno-Occlusive | absent | mild | moderate | severe | life-threatening |
| Disease (VOD) | | | | | |
| Also consider Weight gain-VOD, Bilirubin, Depressed level of consciousness, Hepatic pain, Renal failure, Hepatic | | | | | |
| enlargement. | | | | | |